## **Statistical Analysis Plan**

**Study ID:** 212496

**Official Title of Study:** A phase 3, randomized, open-label, multi-country study to evaluate the immunogenicity, safety, reactogenicity and persistence of a single dose of the RSVPreF3 OA investigational vaccine and different revaccination schedules in adults aged 60 years and above.

NCT number: NCT04732871

**EudraCT number:** 2019-004680-51

**Date of Document:** 27-MAR-2023

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 3

| Statistical Analysis Plan | |
|---|---|
| Title: | A phase 3, randomized, open-label, multi-country study to evaluate the immunogenicity, safety, reactogenicity and persistence of a single dose of the RSVPreF3 OA investigational vaccine and different revaccination schedules in adults aged 60 years and above. |
| eTrack study number and<br>Abbreviated Title | 212496 (RSV OA=ADJ-004) |
| Scope: All data pertaining to the above study except the Safety Review Team analyses for the first 50 participants aged 80 years and above | |
| Date of Statistical Analysis Amendment 3 Final: 27 Mar 2023 Plan | |

APP 9000058193 Statistical Analysis Plan Template V5 (Effective date: 1July2020)

27 Mar 2023 Page 1 of 38

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 3

## **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| LIS | ST OF | ABBREV | IATIONS | 6 |
| 1. | DOC | JMENT H | HISTORY | 7 |
| 2. | OBJE | ECTIVES/ | /ENDPOINTS | 8 |
| 3. | STUE | OY DESIG | 3N | q |
| <b>J</b> . | 3.1. | | design | |
| 4. | ANAL | | TS | |
| | 4.1. | | on | |
| | 4.2. | | for eliminating data from Analysis Sets | |
| | | | Elimination from ES | |
| | | 4.2.2. | | |
| | | | 4.2.2.1. Excluded participants | 12 |
| 5. | STAT | ISTICAL | ANALYSES | 17 |
| | 5.1. | Genera | I considerations | |
| | | 5.1.1. | Demography | |
| | | | Immunogenicity | |
| | | 5.1.3. | | 19 |
| | 5.2. | | s of demography and baseline characteristics | |
| | | 5.2.1. | | |
| | <b>-</b> 0 | 5.2.2. | | |
| | 5.3. | • | rendpoint(s) | |
| | | 5.3.1. | | 20 |
| | | | 5.3.1.1. Humoral immune response – up to Month 12 | 20 |
| | 5.4. | Second | ary endpoint(s) | |
| | 5.4. | 5.4.1. | | |
| | | 5.4.2. | | |
| | | 5.4.3. | Additional considerations | |
| | | 011101 | 5.4.3.1. Mixed effects model | |
| | | | 5.4.3.2. Cell-mediated immune response | |
| | | | 5.4.3.3. Assessment of long-term persistence of the | |
| | | | immune response at Months 18, 24 and 36 | |
| | | | after dose 1 | 25 |
| | | | 5.4.3.4. Sensitivity analyses | 27 |
| | | 5.4.4. | Safety analysis | |
| | | 5.4.5. | Additional considerations | |
| | | | 5.4.5.1. Concomitant Medication | |
| | | 5.4.6. | Sensitivity Analyses | 30 |
| 6 | ANAI | YSIS IN | TERPRETATION | 30 |

| | | | | 212496 (RSV OA=A<br>Statistical Analysis Plan Amen | |
|---|---|---|---|---|---|
| 7. | INTERIM | / ANAL | YSES | ······································ | |
| | | | | ses | |
| | | | | rations for interim analyses | |
| 8. | CHANGI | ES TO | THE PRO | TOCOL DEFINED STATISTICAL | |
| | | | | | 31 |
| 9. | NON-ST | ANDAI | RD DATA | DERIVATION RULES AND STATISTICAL | |
| | | | | | 32 |
| | 9.1. H | andling | of missin | g data | 32 |
| 10. | ANNEXE | S | | | 33 |
| | 10.1. B | usines | s rules for | standard data derivations and statistical | |
| | | ethods | | | |
| | 10 | | | g events to vaccine doses | |
| | 10 | 0.1.2. | | of missing data | |
| | | | 10.1.2.1. | Dates | 33 |
| | | | 10.1.2.2. | Laboratory data | 33 |
| | | | 10.1.2.3. | Daily recording of solicited events | 33 |
| | | | | 10.1.2.3.1. Studies with paper diaries | |
| | | | 10.1.2.4. | Unsolicited adverse events | |
| | 10 | 0.1.3. | | /ation | |
| | | | | Age at first dose in years | |
| | | | 10.1.3.1. | Temperature | 35 |
| | | | 10.1.3.2. | Numerical serology results | 3F |
| | | | 10.1.3.4. | Geometric mean titers (GMTs) and | 25 |
| | | | 40 4 0 5 | concentrations (GMCs) | |
| | | | | Onset day | |
| | | | | Duration of events | 36 |
| | | | 10.1.3.7. | Counting rules for combining solicited and | |
| | | | | unsolicited AEs | 36 |
| | | | 10.1.3.8. | Counting rules for occurrences of solicited | |
| | | | | events | 36 |
| | 10 | 0.1.4. | Display of | decimals | 36 |
| | | | 10.1.4.1. | Percentages | 36 |
| | | | | Demographic/baseline characteristics | |
| | | | | statistics | 37 |
| | | | 10 1 4 3 | Serological summary statistics | |
| | 10 | 0.1.5. | | methodology | |
| | - 10 | J. 1.J. | | Exact confidence intervals around | 31 |
| | | | 10.1.5.1. | | 27 |
| | | | | proportions | 31 |
| 1 1 | ADDITIO | ) | NIAI VOEG | S DUE TO THE COVID-19 PANDEMIC | 27 |
| 11. | | ハソベレ ゲ | いったこうごう | J DUL TU THE GUVID-13 FANDEIVIU | o <i>I</i> |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 3

# **LIST OF TABLES**

| PAGE | |
|------|-----------------------------------------------------------------------|
| y10 | Table 1 Study groups, intervention and blinding foreseen in the study |
| 10 | Table 2 Group names and definition for footnote in the TFLs |
| 11 | Table 3 Pooled group names and definition for footnote in the TFLs |
| 11 | Table 4 Sub-group names and definitions for footnote in the TFLs |
| 12 | Table 5 Populations for analyses |
| 13 | Table 6 List of elimination codes |
| 29 | Table 7 Intensity grading scale for solicited events |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 3

# **LIST OF FIGURES**

| | | PAGE |
|----------|-----------------------|------|
| Figure 1 | Study design overview | 9 |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 3

## LIST OF ABBREVIATIONS

**AE** Adverse event

**AESI** Adverse Events of Special Interest

ANCOVA Analysis of Covariance
CD Community Dwelling

CI Confidence Interval

**COVID-19** Coronavirus Disease 2019

**CRF** Case Report Form

CTRS Clinical Trial Registry Summary

Eli Type Internal database code for type of elimination code

**ELISA** Enzyme-linked immunosorbent assay

**ES** Exposed Set

**EU/mL** ELISA unit per milliliter

**GMC** Geometric mean antibody concentration

**GMT** Geometric mean antibody titer

**GSK** GlaxoSmithKline

IU/mL International units per milliliter

LL Lower Limit of the confidence interval

**MedDRA** Medical Dictionary for Regulatory Activities

NA Not Applicable

PD Protocol Deviation
PPS Per-Protocol Set

SAE Serious adverse event
SAP Statistical Analysis Plan

SBIR GSK Biologicals Internet Randomization System

**SD** Standard Deviation

**SDTM** Study Data Tabulation Model

UL Upper Limit of the confidence interval

# 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|---|---|---|
| 15 February 2021 | First version | Final: 28 October 2020 |
| 04 March 2022 | Amendment 1: | Final: 28 October 2020 |
| 20 June 2022 | <ul> <li>Amendment 2:</li> <li>The study design (Figure 1) was updated with the addition of a revaccination dose at Month 24 and a new follow-up visit at Month 25 for the RSV_flexible revaccination group. (Section 3.1).</li> <li>Table 1 was updated with the addition of a revaccination dose at Month 24 for the RSV_flexible revaccination group (Section 3.1).</li> <li>Table 6 was updated with the addition of RSV_flexible revaccination group at Months 24 and 25 to the list of elimination codes</li> <li>SAEs/pIMDs within 30 days following</li> </ul> | |
| each vaccination (Section 5.4.5) Amendment 3: The elimination code 2100 has been split into 2100h and 2100c (Section 4.2.2). Table 6 has been updated to include these 2 codes. This change will impact the participant disposition tables from ES to PPS for humoral immunogenicity and PPS for CMI. Also the table that shows summary of important protocol deviations leading to elimination from any analyses will be impacted | | Amendment 1: 01 April 2022 |

# 2. OBJECTIVES/ENDPOINTS

| Objectives | Endpoints |
|---|---|
| To evaluate the humoral immune response following a 1-dose primary schedule of RSVPreF3 OA investigational vaccine up to 12 months post-Dose 1. | Humoral immune response at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), and at 6 and 12 months post-Dose 1 (Months 6 and 12), in a subset of participants: Neutralizing antibody titers against RSV-A Neutralizing antibody titers against RSV-B. |
| Sec | ondary |
| To further evaluate the humoral immune response following a 1-dose primary schedule of RSVPreF3 OA investigational vaccine up to 12 months post-Dose 1. | Humoral immune response at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), and at 6 and 12 months post-Dose 1 (Months 6 and 12), in a subset of participants: RSVPreF3-specific Immunoglobulin G (IgG) antibody concentrations. |
| To evaluate the humoral immune response following 1 dose of the RSVPreF3 OA investigational vaccine and following revaccination doses, up to study end. | Humoral immune response at Months 18, 24, 30 and 36 post-Dose 1, and at 1 month after each revaccination dose (Months 13 and 25), in a subset of participants: Neutralizing antibody titers against RSV-A and RSV-B RSVPreF3-specific IgG antibody concentrations. |
| To evaluate the cell-mediated immune (CMI) response following 1 dose of the RSVPreF3 OA investigational vaccine and following revaccination doses up to study end. | <ul> <li>CMI response at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), at Months 6, 12, 18, 24, 30 and 36 post-Dose 1, and at 1 month after each revaccination dose (Months 13 and 25), in a subset of participants:</li> <li>Frequency of RSVPreF3-specific CD4+ and/or CD8+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 4-1BB, IL-2, TNF-α, IFN-γ, IL-13, IL-17.</li> </ul> |
| To evaluate the safety and reactogenicity of each vaccination schedule of the RSVPreF3 OA investigational vaccine in all participants. | <ul> <li>Occurrence of each solicited administration-site and systemic event during a 4-day follow-up period (i.e., on the day of vaccination and 3 subsequent days) after each vaccination.</li> <li>Occurrence of any unsolicited AE during a 30-day follow up period (i.e., on the day of vaccination and 29 subsequent days) after each vaccination.</li> <li>Occurrence of all SAEs and pIMDs up to 6 months after each vaccination.</li> <li>Occurrence of fatal SAEs, related SAEs and related pIMDs from first vaccination (Day 1) up to study end (Month 36).</li> </ul> |
| | rtiary |
| To further characterize immune responses to the RSVPreF3 OA investigational vaccine. | <ul> <li>Any further exploratory immunology in a subset of participants, such as, but not limited to: <ul> <li>Antibodies against specific protein F epitopes.</li> <li>Potential new immunological markers for protection.</li> </ul> </li> <li>Frequency of RSVPreF3-specific CD4+ and/or CD8+ T cells expressing one or any combination of immune marker(s)</li> </ul> |

CMI = cell-mediated immunity, AE = adverse event, SAE = serious adverse event, pIMD = potential immune-mediated disease.

## STUDY DESIGN

## 3.1. Overall design

#### Figure 1 Study design overview



N = number of participants; D = day; M = month; AE = adverse event; HI = humoral immunity; CMI = cell-mediated immunity; pIMD = potential immune-mediated disease; SAE = serious adverse event.

= blood sample for humoral immune responses (only applicable for ~ 345 participants of the RSV\_annual group; and for all participants of the RSV\_flexible revaccination and RSV\_1dose groups)

= blood sample for CMI (only applicable for ~345 participants of the RSV\_annual group, and for ~115 participants each from the RSV\_flexible revaccination and RSV\_1dose groups).

Note: For group RSV\_annual: Revaccination Year 1 = Month 12; Revaccination Year 2 = Month 24; for group RSV\_flexible revaccination: Revaccination Year 2 = Month 24.

- \*Visit and follow-up of solicited events, unsolicited AEs, SAEs and pIMDs are only applicable for RSV\_annual group.

  \*\*Visit and follow-up of solicited events, unsolicited AEs, SAEs and pIMDs are only applicable for RSV\_annual and RSV\_flexible revaccination groups.
- \*\*\*For the RSV\_annual group, the same ~345 participants will be part of both the HI and CMI subsets. The remaining ~645 participants will have no blood draws and will only be followed up for safety and reactogenicity.
- \*\*\*\*\*For those participants in the RSV\_annual group without blood sample collections, visits at Months 6, 18, 30 and 36 may be held through a contact. However, contact should be attempted only if site visit is not possible at Months 6, 18, 30 and 36.
- Type of study: self-contained.
- Experimental design: Phase 3, randomized, open-label, multi-country study with 3 parallel groups (see Figure 1).
- **Duration of the study**: ~ 36 months for each participant.
- **Primary completion date**: Month 12.

- Control: none.
- **Blinding**: open-label. Refer to the protocol for details.
- **Data collection**: standardized electronic Case Report Form (eCRF). Solicited events and unsolicited adverse events (AEs) will be collected using a participant Diary card (paper Diary card).
- Safety monitoring: the study will be conducted with oversight by the project Safety Review Team (SRT). Please refer to protocol for the description of review of safety data by the SRT.
- Study groups: refer to Figure 1 and Table 1 for an overview of the study groups

Table 1 Study groups, intervention and blinding foreseen in the study

| | | | Intervention | | | Blinding |
|---|---|---|---|---|---|---|
| Study Groups | Number of participants | Age | Primary vaccination | Revaccination<br>Year 1 (Month<br>12) | Revaccination<br>Year 2 (Month<br>24) | Open |
| RSV_annual* | ~990 | ≥60 years | RSVPreF3 OA investigational vaccine | RSVPreF3 OA investigational vaccine | RSVPreF3 OA investigational vaccine | Х |
| RSV_flexible revaccination | ~330 | ≥60 years | RSVPreF3 OA investigational vaccine | (none) | RSVPreF3 OA investigational vaccine | Х |
| RSV_1dose | ~330 | ≥60 years | RSVPreF3 OA investigational vaccine | (none) | (none) | Х |

<sup>\*</sup> RSV\_annual group will be split in 3 technical groups in SBIR in order to have a randomization ratio of 1:1:1:1:1: for treatment allocation and avoid predictability.

• **Groups and sub-groups definition for analysis:** Refer to the tables below for a description of the groups and subgroups labels that will be used in the Tables Figures and Listings (TFLs).

The analyses pertaining to timepoints up to Month 12 will be performed for each group and for the 3 groups pooled. From Month 13 up to study end, the analyses will be performed by group.

The following group names will be used in the TFLs:

Table 2 Group names and definition for footnote in the TFLs

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | RSV_annual | Participants receiving the first dose (Dose 1) of RSVPreF3 OA investigational vaccine at Day 1, followed by a revaccination dose at 12 months post-Dose 1 and at 24 months post-Dose 1 |
| 2 | RSV_flexible revaccination | Participants receiving the first dose (Dose 1) of RSVPreF3 OA investigational vaccine at Day 1 and a revaccination dose at 24 months post-Dose 1 |
| 3 | RSV_1dose | Participants receiving a single dose (Dose 1) of RSVPreF3 OA investigational vaccine at Day 1 |

Table 3 Pooled group names and definition for footnote in the TFLs

| Pooled Group label in tables | Groups to be pooled | Pooled definition for footnote | Comment |
|---|---|---|---|
| Total | RSV_annual,<br>RSV_flexible<br>revaccination and<br>RSV_1dose | Participants receiving one dose of RSVPreF3 OA investigational vaccine at Day 1 in all the three groups | Applicable on data reported up to Month 12 |
| Flexible+1dose | RSV_flexible<br>revaccination, and<br>RSV_1dose | Participants receiving one dose of RSVPreF3 OA investigational vaccine at Day 1 in the RSV_flexible revaccination, and RSV_1dose groups | Applicable on data reported at Month 13, Month 18 and Month 24 |

Table 4 Sub-group names and definitions for footnote in the TFLs

| Sub-analysis | Subgroup order in tables | Subgroup label in tables | Subgroup definition for footnote |
|---|---|---|---|
| By age | 1 | ≥65YOA | ≥65 years old participants |
| | 2 | ≥70YOA | ≥70 years old participants |
| | 3 | ≥80YOA | ≥80 years old participants |
| | 4 | 60-69YOA | 60-69 years old participants |
| | 5 | 70-79YOA | 70-79 years old participants |
| By sex | 1 | Female | Female |
| | 2 | Male | Male |
| By region | 1 | North America | Participants from North America (United States of America) |
| | 2 | Europe | Participants from Europe (Finland, Germany) |
| | 3 | Asia | Participants from Asia (Japan, Taiwan) |

YOA = Years of age

#### Allocation of participants to assay subsets

Allocation of participants to assay subsets will be performed using SBIR. The subsets are detailed below.

| | RSV_annual | RSV_flexible revaccination | RSV_1dose |
|---|---|---|---|
| HI subset | ~345* | All participants (~330) | All participants (~330) |
| CMI subset | ~345* | ~115 | ~115 |

<sup>\*</sup>For the RSV\_annual group, the same ~345 participants will be part of both the HI and CMI subsets. The remaining ~645 participants will have no blood draws, and will only be followed up for safety and reactogenicity.

- **HI subset:** ~345 participants from the RSV\_annual group, and all participants from the RSV\_flexible revaccination and RSV\_1dose groups. These participants will have blood samples collected for testing of humoral immunity at each visit applicable for their study group.
- **CMI subset**: ~345 participants from the RSV\_annual group, and ~115 participants each from the RSV\_flexible revaccination and RSV\_1dose groups. These participants will have additional blood samples collected for CMI testing at each visit applicable for their study group.

## 4. ANALYSIS SETS

### 4.1. Definition

Table 5 Populations for analyses

| Analysis set | Description |
|---|---|
| Enrolled set | Participants who agreed to participate in a clinical study after completion of the informed consent process. |
| Exposed set (ES) | All participants who received at least 1 dose of the study intervention. The allocation in a group is done in function of the administered intervention. |
| Per Protocol set (PPS) | All participants who received at least 1 dose of the study intervention to which they are randomized and have post-vaccination data, minus participants with protocol deviations that lead to exclusion. |

The primary analysis for immunogenicity will be performed on the Per Protocol set (PPS). If the percentage of vaccinated participants with serological results excluded from the PPS for immunogenicity is at least 5% for at least 1 visit and at least 1 group, a second analysis will be performed on the Exposed Set (ES). The immunogenicity analysis will be performed overall, by sex, by age category (age at Dose  $1: \ge 65$  YOA,  $\ge 70$  YOA,  $\ge 80$  YOA, 60-69 YOA and 70-79 YOA, and by region (North America, Europe, Asia).

## 4.2. Criteria for eliminating data from Analysis Sets

#### 4.2.1. Elimination from ES

Code 1030 (Study intervention not administered at all), 800 (Fraudulent data) and code 900 (Invalid informed consent) will be used for identifying participants eliminated from the ES.

## 4.2.2. Elimination from Per-protocol analysis Set (PPS)

## 4.2.2.1. Excluded participants

A participant will be excluded from the populations of analysis under the following conditions

- For codes 800, 900, 1030 and 1050: participants will be eliminated for all visits.
- For codes 1040, 1070, 1080, 1090, 2010, 2040, 2050, 2080: participants will be eliminated from a specific visit (at which the condition is met) onwards.
- For codes 2090, 2100h, 2100c, 2120: participants will be eliminated at the specific visit at which the condition is met.

# Table 6 List of elimination codes

| Code | Condition under which the code is used | Visit (timepoints) where the code is checked | Applicable for analysis set |
|---|---|---|---|
| 800 | Fraudulent data | All | ES and PPS |
| 900 | Invalid informed consent | All | ES and PPS |
| 1030 | Study intervention not administered at all | All | ES and PPS |
| 1040 | Administration of concomitant vaccine(s) forbidden in the protocol | All | PPS |
| | • Any investigational or non-registered vaccine other than the study vaccine used during the study period beginning 30 days before the first dose of study vaccine, or planned use during the study period. | | |
| | • Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before each dose and ending 30 days after each dose of study vaccine administration, with the exception of inactivated, split virion and subunit influenza vaccines which can be administered up to 14 days before or from 14 days after each study vaccination. | | |
| | Previous vaccination with an RSV vaccine | | |
| 1050 | Randomization failure | Day 1 | PPS |
| 1070 | Vaccine administration not according to protocol Incomplete vaccination course | Vaccination visits at Day 1, Month 12, and 24 | PPS |
| | Participant was vaccinated with the correct vaccine but containing a lower volume | Months 12 and 24 are applicable to the RSV_annual group and Month 24 applies | |
| | Participant was re-vaccinated while it was not planned | to the RSV_flexible revaccination group | |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 3

| <u> </u> | Statistical Analysis Plan Amendmen | | |
|---|---|---|---|
| Code | Condition under which the code is used | Visit (timepoints) where the code is checked | Applicable for analysis set |
| | Route of the study intervention is not intramuscular | | |
| | Wrong reconstitution of<br>administered vaccine | | |
| 1080 | Vaccine administration after a Temperature deviation | Day 1, Month 12, and 24 | PPS |
| | Vaccine administered despite<br>a Good Manufacturing<br>Practices (GMP) no-go<br>temperature deviation | Months 12 and 24 are applicable to the RSV_annual group and Month 24 applies to RSV_flexible revaccination group | |
| 1090 | Vaccine administration after expiration | Day 1, Month 12, and 24 Months 12 and 24 are applicable to the RSV_annual group and Month 24 belongs to the RSV_flexible revaccination group | PPS |
| 2010 | Protocol deviation linked to inclusion/exclusion criteria | All | PPS |
| 2040 | Administration of any medication forbidden by the protocol | All | PPS |
| | Any investigational or non-<br>registered medication used<br>during the study period | | |
| | Administration of long-acting immune-modifying drugs at any time during the study period (e.g. infliximab) | | |
| | Immunoglobulins and/or any<br>blood products administered<br>during the study period | | |
| | Chronic administration (defined as more than 14 consecutive days in total) of immunosuppressants or other immune-modifying drugs during the period starting | | |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 3

| <b>C</b> 1 | Statistical Analysis Plan Amendment | | |
|---|---|---|---|
| Code | Condition under which the code is used | Visit (timepoints) where the code is checked | Applicable for analysis set |
| | 90 days prior to the study vaccine administration or planned administration during the study period. For corticosteroids, this will mean prednisone ≥20 mg/day, or equivalent. | | |
| 2050 | Intercurrent medical condition | All | PPS |
| | • Participants may be eliminated from the PPS for immunogenicity if, during the study, they incur a condition that has the capability of altering their immune response (intercurrent medical condition) or are confirmed to have an alteration of their initial immune status. | | |
| 2080 | Participants did not comply with dosing schedule | Month 12 and 24 | PPS |
| | • RSV_annual: number of days between dose 1 and revaccination dose at Month 12 is outside [350-380 days] | | |
| | • RSV_annual and RSV_flexible revaccination: number of days between dose 1 and revaccination dose at Month 24 is outside [715-745 days] | | |
| 2090 | Participants did not comply with blood sample schedule | Day 31, Month 6, 12, 13, 18, 24, 25, 30, 36 | PPS |
| | • Number of days between dose 1 and Day 31 blood sample is outside [30-42 days] | | |
| | • Number of days between dose 1 and Month 6 blood sample is outside [180-210 days] | | |
| | • Number of days between dose 1 and Month 12 blood sample is outside [350-380 days] | | |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 3

| | Statistical Analysis Plan Amendment | | |
|---|---|---|---|
| Code | Condition under which the code is used | Visit (timepoints) where the code is checked | Applicable for analysis set |
| | Number of days between Month 12 and Month 18 blood sample is outside [180-210 days] | | |
| | • Number of days between dose 1 and Month 24 blood sample is outside [715-745 days] | | |
| | Number of days between Month 24 and Month 30 blood sample is outside [180-210 days] | | |
| | Number of days between dose<br>1 and Month 36 blood sample<br>is outside [1080-1110 days] | | |
| | For RSV_annual group only: | | |
| | • Number of days between revaccination at Month 12 and Month 13 blood sample is outside [30-42 days] | | |
| | For RSV_annual and RSV_flexible groups: | | |
| | • Number of days between revaccination at Month 24 and Month 25 blood sample is outside [30-42 days] | | |
| 2600* | Participants not included in the humoral immunogenicity subset | Day 1, 31, Month 6, 12, 13, 18, 24, 25, 30, 36 | PPS |
| 2700* | Participants not included in the cell-mediated immune response subset | Day 1, 31, Month 6, 12, 13, 18, 24, 25, 30, 36 | PPS |
| 2100h | For participants in the humoral immunogenicity subset. No immunological result at visit x for all the following tests: RSV A/B Neutralizing antibody titer and RSV PreF3-specific IgG antibody concentration | Day 1, Day 31, Month 6, 12, 13, 18, 24, 25, 30, 36 Month 13 and 25 are applicable to the RSV_annual and only Month 25 is applicable to the RSV_flexible revaccination group | PPS |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 3

| Code | Condition under which the code is used | Visit (timepoints)<br>where the code is<br>checked | Applicable for analysis set |
|---|---|---|---|
| 2100c | <ul> <li>For participants in the CMI subset</li> <li>No immunological result at visit x for all the following tests: Frequency of RSVPreF3-specific CD4+ and CD8+ T cells</li> </ul> | Day 1, Day 31, Month 6, 12, 13, 18, 24, 25, 30, 36 Month 13 and 25 are applicable to the RSV_annual and only Month 25 is applicable to the RSV_flexible revaccination group | PPS |
| 2120 | Obvious incoherence or abnormality or error in laboratory data • Unreliable released data as a result of confirmed sample mismatch or confirmed inappropriate sample handling at laboratory | Day 1, 31, Month 6, 12, 13, 18, 24, 25, 30, 36 | PPS |

<sup>\*</sup> codes 2600 and 2700 are not considered as protocol deviations, but those codes will be used to identify participants that are not part of the immunogenicity subsets.

## 5. STATISTICAL ANALYSES

Standard data derivation rules and stat methods are described in Section 10.1 while the study specific data derivation rules and stat methods are described in Section 9.

For the sake of analysis, data up to Month 12 will be analyzed by group (RSV\_annual, RSV\_flexible revaccination and RSV\_1dose), and also the 3 groups will be pooled. For Month 13, Month 18 and Month 24, the analyses will be tabulated for RSV\_annual group versus the pooled RSV\_flexible revaccination and RSV\_1dose groups. From Month 25 up to study end, the analyses will be performed by group

If more than 5% of participants in the RSV\_annual and RSV\_flexible revaccination groups receive different number of doses, an analysis by subgroup according to the number of dose(s) administered might be performed. The goal of this analysis is to describe the characteristics of participants in the RSV\_annual and RSV\_flexible revaccination groups who ultimately receive different numbers of revaccination doses in order to rule out the possibility of systematic differences between these subgroups.

#### 5.1. General considerations

## 5.1.1. Demography

For a given participant and a given demographic variable, missing measurements will not be replaced.

## 5.1.2. Immunogenicity

- Any missing or non-evaluable immunogenicity measurement will not be replaced. The descriptive analysis performed for each assay at each timepoint will exclude participants with a missing or non-evaluable measurement. This is applicable to the standard way of computing geometric mean titers/concentrations (GMTs/GMCs).
- During the computation of GMTs/GMCs from the mixed effects model (Section 5.4.3.1). Multiple imputation (MI) technique will not be applied for any missing immunogenicity measurement. This is because the mixed effects model inherently accounts for the missingness, under the assumption that the missing data are missing at random (MAR). Thus considering that missing data are MAR is a reasonable assumption for this descriptive clinical trial, then it is not necessary to perform MI [Rubin et al., 1995]
- The GMTs/GMCs will be computed by taking the anti-logarithm of the arithmetic mean of the log<sub>10</sub> transformed titers/concentrations.
- A seronegative participant will be defined as a participant whose antibody titer/concentration is below the technical cut-off value of the assay. A seropositive participant is a participant whose antibody titer/concentration is greater than or equal to the technical cut-off value of the assay.
- Antibody titers/concentrations below the technical assay cut-off will be given an arbitrary value of half the technical assay cut-off for the purpose of GMT/GMC calculation.
- Antibody titers/concentrations above the Upper Limit of Quantification (ULOQ) value will be given the ULOQ value for the purpose of GMT/GMC calculation.
- The mean geometric increase (MGI) is calculated by the geometric mean of ratios of antibody titers/concentrations of each post vaccination time point over pre vaccination (Day 1).

## 5.1.3. Reactogenicity/Safety

- For a given participant and the analysis of solicited events within 4 days post-vaccination, missing or non-evaluable measurements will not be replaced. Therefore, the analysis of solicited events will include only vaccinated participants with documented solicited safety data (i.e., paper diary completed).
- For analysis of unsolicited AEs, serious adverse events (SAEs), potential immunemediated diseases (pIMDs) and concomitant medications, all vaccinated participants will be considered. Participants who did not report an event or concomitant medication will be considered as participants without the event or the concomitant medication, respectively.

## 5.2. Analysis of demography and baseline characteristics

## 5.2.1. Analysis planned in the protocol

Descriptive summaries will be performed for each group (RSV\_annual, RSV\_flexible revaccination and RSV\_1dose) and overall. The same will be performed in each subset (humoral immune subset and CMI subset).

Demographic/baseline characteristics (age at vaccination in years, sex, race, ethnicity, type of residence (CD/LTCF) and smoking status) will be summarized using descriptive statistics:

- Frequency tables will be generated for categorical variables such as race.
- Mean, median, standard deviation and range will be provided for continuous data such as age.

The distribution of participants will be tabulated as a whole and per group, for each age category, and for each subset.

The number of doses of the study intervention administered will be tabulated by group and by visit.

Withdrawal status will be summarized by group using descriptive statistics:

- The number of participants enrolled into the study as well as the number of participants excluded from Per Protocol (PP) analyses will be tabulated.
- The numbers of participants withdrawn from the study will be tabulated according to the reason for withdrawal.

Participant disposition in the ES and PPS will be reported as a whole and per group

The number and percentage of participants using concomitant medication (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) during the 4-day follow-up period (i.e., on the day of vaccination and 3 subsequent days) and during the 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) will be summarized by group after each vaccine dose and after the revaccination.

#### 5.2.2. Additional considerations

- The analysis of demographic characteristics by group will be performed on the ES and on the PPS.
- Demography and baseline characteristics will also be summarized by sex and region.
- A summary of important protocol deviations leading to elimination from any analyses will be provided by group, based on the Enrolled Set.
- Medical history will be tabulated by System Organ Class (SOC), High Level Term (HLT) and Preferred Term (PT).

## 5.3. Primary endpoint(s)

## 5.3.1. Analysis planned in the protocol

The primary analysis for immunogenicity will be performed on the PPS. If the percentage of vaccinated participants with serological results excluded from the PPS for immunogenicity is at least 5% for at least 1 visit and at least 1 group, a second analysis will be performed on the ES.

### 5.3.1.1. Humoral immune response – up to Month 12

The analysis of the primary vaccination timepoints up to Month 12 will be performed for each group and for the 3 groups pooled. For each timepoint with blood sample collection for humoral immune response up to Month 12 and for each assay (RSV-A/-B neutralization assays), unless otherwise specified, the following analyses will be performed:

#### Within groups evaluation:

- Percentage of participants with antibody titers/concentrations above or equal to the technical assay cut-off and their exact 95% confidence interval (CI) will be tabulated.
- GMTs/GMCs and their 95% CI will be tabulated and represented graphically. Furthermore, to account for all the timepoints at which the blood samples are collected, a mixed effects model (see Section 5.4.3.1) will be fitted, from which the GMTs/GMCs will be computed.
- Antibody titers/concentrations will be displayed using reverse cumulative curves.
- The MGI i.e. geometric mean of ratios of antibody titer/concentrations will be tabulated with 95% CI.

## 5.4. Secondary endpoint(s)

## 5.4.1. Humoral immune response

The same analyses as described above for the primary endpoint will be performed for RSVPreF3-specific IgG ELISA up to Month 12 and for each timepoint with blood sample collection for humoral immune response **from study Month 13 up to study end** and for each assay (RSVpreF3-specific IgG **ELISA and RSV-A/-B neutralization assays**). For Month 13, Month 18, and Month 24, the analyses will be tabulated for RSV\_annual group versus the pooled RSV\_flexible revaccination and RSV\_1dose groups. From Month 25 up to study end, the analyses will be performed by group.

Only the analyses requiring further clarification of the exact timepoints analyzed are summarized below:

## Within groups evaluation:

- The MGI i.e. geometric mean of ratios of antibody titer/concentrations will be tabulated with 95% CI:
  - For each post-primary vaccination time point (at Months 18, 24, 30 and 36 when applicable) over pre-primary vaccination (Day 1),
  - For each post-revaccination time point over corresponding pre-revaccination (Months 12 and 24) in the RSV annual group,
  - For each post-revaccination timepoint over corresponding pre-revaccination (Month 24) in the RSV flexible revaccination group,
  - For 1 month post-revaccination at Month 12 (Month 13) over 1 month post-Dose 1 vaccination (Day 31) in RSV annual group.
  - For 1 month post-revaccination at Month 24 (Month 25) over 1 month post-revaccination at Month 12 (Month 13) in RSV\_annual group
  - For 1 month post-revaccination at Month 24 (Month 25) over 1 month post-Dose 1 vaccination (Day 31) in RSV flexible revaccination group.

In addition, the following evaluation will be performed:

• The kinetics of GMTs/GMCs will be plotted as a function of time for participants with results available at all post vaccination timepoints.

The immunogenicity analysis will be performed overall, by sex, age category (age at Dose  $1: \ge 65 \text{ YOA}, \ge 70 \text{ YOA}, \ge 80 \text{ YOA}, 60-69 \text{ YOA}$  and 70-79 YOA), and region (North America, Europe, Asia).

## 5.4.2. Cell-mediated immune response

### Within groups evaluation:

The following parameters will be summarized by group at each timepoint for which blood samples are collected, for the 3 groups pooled for time points up to study Month 12, for Month 13, Month 18 and Month 24, the analyses will be tabulated for RSV\_annual group versus the pooled RSV\_flexible revaccination and RSV\_1dose groups. From Month 25 up to study end, the analyses will be performed by group using descriptive statistics (N, geometric mean, min, Q1, median, Q3, max) in the CMI subset:

- Frequency of RSVPreF3-specific CD4+ and/or CD8+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13, IL-17, measured by intracellular cytokine staining (ICS) using peripheral blood mononuclear cells PBMCs.
- The kinetics of RSVPreF3-specific CD4+ T cells frequencies will be plotted as a function of time for participants with results available at all timepoints.
- Fold increase of the frequency of RSVPreF3-specific CD4+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13, IL-17, measured by ICS at each post-primary vaccination timepoint over pre-vaccination (Day 1) by group, at each post-revaccination over the corresponding pre-revaccination (Month 12/Month 24 in the RSV\_annual group and Month 24 in the RSV\_flexible revaccination group), at one month post-revaccination over 1 month post-previous dose in the RSV\_annual group [one month post-revaccination at Month 12 (Month 13) over one month post-Dose 1 vaccination (Day 31) and one month post-revaccination at Month 24 (Month 25) over one month post-revaccination at Month 12 (Month 13)] and in the RSV\_flexible revaccination group [one month post-revaccination at Month 24 (Month 25) over one month post-Dose 1 vaccination (Day 31)].

The immunogenicity analysis will be performed overall, by sex, age category (age at Dose  $1: \ge 65 \text{ YOA}, \ge 70 \text{ YOA}, \ge 80 \text{ YOA}, 60-69 \text{ YOA}$  and 70-79 YOA, and region (North America, Europe, Asia).

#### 5.4.3. Additional considerations

#### 5.4.3.1. Mixed effects model

For the GMTs/GMCs calculation based on the mixed effects model mentioned in Section 5.3.1.1, repeated measures analysis of covariance (ANCOVA) model will be fitted including age category (60-69 YOA, 70-79 YOA and ≥80 YOA,), study group (RSV\_annual, RSV\_flexible revaccination and RSV\_1dose), sex (male and female), visit (Day 31, Months 6, 12, 13, 18, 24, 25, 30, 36), as fixed effects, pre-vaccination log10-transformed titers/concentrations as a covariate and the response variable is the post-vaccination log10-transformed titers/concentrations. The PROC MIXED procedure in SAS® will be used to carry out the ANCOVA.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 3

The following SAS codes will be used:

For the analysis by study group, study group and visit will be included as the fixed effects in the model

```
Analysis by group
PROC MIXED DATA=SERO method=reml empirical;
CLASS subjid group visit;
MODEL post-vac=pre-vacc group visit visit*group/ noint s cl;
RANDOM intercept/ subject=usubjid g v vcorr type = un;
REPEATED visit/type=unsubject=subjid;
LSMEANS visit*group/ E cl;
ODS OUTPUT LSMEANS=LS;
RUN;
```

For the analysis by age category, age category and visit will be included as the fixed effects in the model. However, this is only applicable at timepoints where the 3 study groups will be pooled. Otherwise for the timepoints where pooling of the 3 groups is not possible, the fixed effects will include study group, age category and visit.

#### Analysis by age-category

```
PROC MIXED DATA=SERO method=reml empirical;
CLASS subjid visit agecat;
MODEL post-vac=pre-vacc agecat visit visit* agecat /noint s cl;
RANDOM intercept/ subject=usubjid g v vcorr type = un;
REPEATED visit/type=un subject=subjid;
LSMEANS visit*agecat/ E cl;
ODS OUTPUT LSMEANS=LS;
RUN;
```

For the analysis by sex, sex and visit will be included as the fixed effects in the model. However, this is only applicable at timepoints where the 3 study groups will be pooled. Otherwise for the timepoints where pooling of the 3 groups is not possible, the fixed effects will include study group, sex and visit.

#### Analysis by sex

```
PROC MIXED DATA=SERO method=reml empirical;
CLASS subjid visit agecat;
MODEL post-vac=pre-vacc sex visit visit* sex / noint s cl;
RANDOM intercept/ subject=usubjid g v vcorr type = un;
REPEATED visit/type=un subject=subjid;
LSMEANS visit*sex/ E cl;
ODS OUTPUT LSMEANS=LS;
RUN;
```

For the analysis by region, region and visit will be included as the fixed effects in the model. However this is only applicable at timepoints where the 3 study groups will be pooled. Otherwise for the timepoints where pooling of the 3 groups is not possible, the fixed effects will include study group, region and visit.

#### Analysis by region

```
PROC MIXED DATA=SERO method=reml empirical;
CLASS subjid visitregion;
MODEL post-vac=pre-vacc region visit visit* region / noint scl;
RANDOM intercept/ subject=usubjid g v vcorr type = un;
REPEATED visit/type=un subject=subjid;
LSMEANS visit*region/ E cl;
ODS OUTPUT LSMEANS=LS;
RUN;
```

The GMTs/GMCs, lower and upper confidence limits are obtained from the following data step:

```
DATA LS;
   SET LS;
   gm=10**estimate;
   11=10**lower;
   u1=10**upper;
RIIN:
```

The above SAS codes may be adapted in case of convergence issues.

#### 5.4.3.2. Cell-mediated immune response

#### Within groups evaluation

- The frequency of RSVPreF3 specific-CD4+ T cells will be displayed graphically using boxplots (min, Q1, median, Q3, max), by group and timepoint.
- The RSVPreF3-specific CD4+/ CD8+ T cell frequencies will be obtained by subtracting the background value to the antigen-induced value, and by setting to 1 all values less than or equal to zero for geomean calculation and graphical representation. Frequencies will be expressed as the number of cells per million of CD4+ T cells.
- More specifically, the frequencies of RSVPreF3-specific CD4+/ CD8+ T cells expressing at least 2 activation markers including at least one cytokine [Freq<sup>2+</sup>] will be computed as follows:

$$Freq_{Background}^{2+} = \frac{n_{background}^{2+}}{N_{Background}^{CD4}}$$
 and  $Freq_{Induction}^{2+} = \frac{n_{Induction}^{2+}}{N_{Induction}^{CD4}}$ 

And

$$Freq_{Specific}^{2+} = Freq_{Induction}^{2+} - Freq_{Background}^{2+}$$

where

 $n_{Background}^{2+}$  = number of CD4+ T cells expressing at least 2 activation markers including at least one cytokine after stimulation with medium only (background),

 $n_{Induction}^{2+}$  = number of CD4+ T cells expressing at least 2 activation markers including at least one cytokine after stimulation with a pool of peptides covering RSVPreF3 (induction),

 $N_{\it Back/Ind}^{\it CD4}$  = Total number of CD4 T cells involved in the assay (background or induction).

For the computation of the fold increase (post- over pre-vaccination) of the frequency of RSVPreF3-specific CD4+ T-cells identified as expressing **at least 2 activation marker(s) including at least one cytokine\*** among CD40L, 4-1BB, IL-2, TNF-α, IFN-γ, IL-13, IL-17.the results **below the LLOQ** of the assay will be replaced by the value of the LLOQ.

# 5.4.3.3. Assessment of long-term persistence of the immune response at Months 18, 24 and 36 after dose 1

The exploratory analysis for modelling the long-term persistence of immune response (humoral and cellular) post dose 1 vaccination will constitute of the following;

- A piece-wise linear mixed model, power law model and modified power law model [David et al, 2009] for repeated measurements (all data available from Day 31, Month 6, 12, 18, 24, 30, 36 post-Dose 1 vaccination, will be used to model over time
  - the frequency of RSVPreF3-specific CD4+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 4-1BB, IL-2, TNF-α, IFN-γ, IL-13, IL-17.
  - the neutralizing antibody titers against RSV-A, RSV-B and RSVPreF3-specific IgG antibody concentrations.

The *piece-wise linear mixed model* is expressed as follows

The piece-wise model fits the data on non-overlapping time intervals. This corresponds to the observed decay of humoral and cellular antibodies. Each piece of the model uses a linear function. Break points will be selected on the basis of Akaike's Information Criterion (AIC) [Pan, 2001].

$$(ft) = \beta_0 + \beta_1 t \qquad \text{if } x \le t < xx \text{ months}$$

$$(ft) = \beta_0 + \beta_1 t + \beta_2 (t - xx) \quad \text{if } xx \le t < xxx \text{ months}.$$

$$(ft) = \beta_0 + \beta_1 t + \beta_2 (t - xx) + \beta_3 (t - xxx) \quad \text{if } t \ge xxx \text{ months}$$

where f(t) is the log-10 transformed antibody titer/concentration/ RSVPreF3-specific CD4+ T cells at time t post-vaccination,  $\beta_0$  is the intercept and  $\beta_1(i=1,2,3...)$  are the

<sup>\*</sup> cytokines are IL-2, TNF-α, IFN-γ, IL-13, and IL-17

parameters corresponding to the time intervals, respectively. All the model effects will be fitted using the SAS PROC MIXED standard code for linear regression methodology for repeated data.

```
ODS OUTPUT FitStatistics= stat;
ODS OUTPUT ConvergenceStatus= conv;
PROC MIXED DATA=kin&i.&j. EMPIRICAL COVTEST NOCLPRINT IC;
CLASS pid;
MODEL log val = int m int m pw m&i.*m&i. int m pw m&j.*m&j./s cl
covb outp=pred outpm=predm;
RANDOM intercept/SUBJECT=pid;
MAKE "solutionF" out=est;
RUN:
```

The *power-law model* is expressed as follows:

$$f(t) = k - a \log(c + t)$$

where f(t) is the log-10 transformed antibody titer/concentration/ RSVPreF3-specific CD4+ T cells at time t post-vaccination, k is the peak log level, a is the decay rate, and c is an arbitrary small constant (set to zero in this case). The estimated maximum likelihood (ML) values for the model parameters will be obtained using the PROC NLMIXED SAS procedure.

```
PROC NLMIXED DATA=kineticm;
PARMS se=&se a0 =&a k0 = k sk=&sk sa=&sa ska=&ska;
q = (1/\&time)**a;
lg=\&log(q);
mean = k + lq;
MODEL log val ~ NORMAL(mean, se*se);
RANDOM k a ~ NORMAL([k0,a0], [sk*sk, ska, sa*sa]) SUBJECT=pid out=indiv;
RUN;
```

The *modified power-law model* is expressed as follows:

It is an extension of the power law model, and it is expressed as follows.

$$f(t) = k + \log[(1 - \pi)(c + t)^{a} + \pi]$$

The quantity  $\pi$  (between 0 and 1) represents the proportion of antibodies that are produced in the long term. When the value of  $\pi$  is positive, this implies long-term antibody persistence, as noted by [Fraser et al, 2007]. If  $\pi = 0$ , then the modified powerlaw model reduces to the standard power-law model. The estimated maximum likelihood (ML) values for the model parameters will be obtained using the PROC NLMIXED SAS procedure.

```
PROC NLMIXED DATA=kineticm ;
PARMS pi=&pi se=&se a0 =&a k0 =&k sk=&sk sa=&sa ska=&ska;
q = (1-pi)*(1/\&time)**a;
lg=&log(q+pi);
mean = k + lq;
MODEL log val ~ NORMAL(mean, se*se);
RANDOM k a ~ NORMAL([k0,a0], [sk*sk, ska, sa*sa]) SUBJECT=pid out =indiv
RUN;
```

- The three models based on data up to Month 36 will be presented graphically. Models based on data up to Month 18 vs. Month 24, Month 24 vs. Month 30 and Month 30 vs. Month 36 will be presented side by side.
- The above models and SAS codes may be adapted in case of convergence issues.

#### 5.4.3.4. Sensitivity analyses

- In case the COVID-19 pandemic is still ongoing during the study conduct, the following sensitivity analyses might be considered.
  - During the assessment of long-term persistence of the immune response, the models described in Section 5.4.3.3 might be fitted taking into account participants who received the first dose of study vaccine and with full follow-up (attending all study visits).
  - Similarly, a mixed model might be fitted for the evaluation of GMT/GMC based on participants with full follow-up (attending all study visits).

The goal of this sensitivity analysis is to determine the extent to which results might be impacted by considering the different scenarios.

## 5.4.4. Safety analysis

## Primary vaccination and revaccination dose:

The safety analysis will be performed on the ES. A descriptive analysis by group, for the 3 groups pooled up to Month 12, for the RSV\_flexible revaccination and RSV\_1dose groups pooled vs RSV\_annual group for Month 13, Month 18 and Month 24, and by group from Month 25 up to study end, will present a summary of:

- The number and percentage of participants with at least one administration site event (solicited and unsolicited), with at least one systemic event (solicited and unsolicited) and with any AE during the 4-day or 30-day follow-up period will be tabulated with exact 95% CI after each dose. The same computations will be done for Grade 3 AEs, and for Grade 3 non-serious AEs and for AEs resulting in medically attended visit.
- The number and percentage of participants reporting each individual solicited administration site event (any grade, Grade 3 and resulting in medically attended visit) and solicited systemic event (any grade, Grade 3 and resulting in medically attended visit) during the 4-day follow-up period (i.e., on the day of vaccination and 3 subsequent days) will be tabulated for each group after each dose.
- For fever, the number and percentage of participants reporting fever by half degree (°C) cumulative increments during the 4-day follow-up period (i.e., on the day of vaccination and 3 subsequent days) will be tabulated for each group after each dose.
- The incidence of each solicited administration site event and solicited systemic event (any grade and grade 3) will be represented graphically after each dose.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 3

- The number and percentage of participants with any unsolicited AEs during the 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) with its exact 95% CI will be tabulated for each dose by group and by Medical Dictionary for Regulatory Activities (MedDRA) Primary System Organ Class (SOC), High Level Term (HLT) and preferred term (PT). Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs, for Grade 3 causally related unsolicited AEs and for unsolicited AEs resulting in a medically attended visit. The verbatim reports of unsolicited AEs will be reviewed by a qualified person and the signs and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. Every verbatim term will be matched with the appropriate Preferred Term.
- The number and percentage of participants with at least one report of SAE classified by the MedDRA Primary SOC, HLT and PTs and reported from Dose 1 up to 6 months post-Dose 1 and from revaccination dose up to 6 months post-revaccination will be tabulated with exact 95% CI. The same tabulation will be presented for causally related SAEs and fatal SAEs,.
- The number and percentage of participants with at least one report of causally related SAEs classified by the MedDRA Primary SOC, HLT and PTs will be reported after each dose and from Day 1 up to study end with exact 95% CI. The same tabulation will be presented for fatal SAEs.
- All SAEs will also be described in detail in a tabular listing.
- All AEs/SAEs leading to study/intervention discontinuation from dose 1 up to study end will be tabulated.
- The number and percentage of participants with at least one report of pIMD classified by the MedDRA Primary SOC, HLT and PTs and reported from Dose 1 up to 6 months post-Dose 1 and from revaccination dose up to 6 months post-revaccination will be tabulated with exact 95% CI. The same tabulation will be presented for causally related pIMDs
- The number and percentage of participants with at least one causally related pIMD classified by the MedDRA Primary SOC, HLT and PTs will be reported after each dose and from Day 1 up to study end with exact 95% CI.
- All pIMDs will also be described in detail in a tabular listing.
- The analyses of unsolicited AEs will include SAEs (unless otherwise specified).

The analysis of safety will also be performed by age category (age at Dose  $1: \ge 65$  YOA,  $\ge 70$  YOA,  $\ge 80$  YOA, 60-69 YOA and 70-79 YOA) and region (North America, Europe, Asia).

#### 5.4.5. Additional considerations

- Compliance in completing solicited events information will be tabulated after each dose.
- The number and percentage of participants with at least one administration site event (solicited only), with at least one systemic event (solicited only) and with any solicited event during the 4-day follow-up period after each dose will be tabulated with exact 95% CI. The same computations will be done for Grade 3 AEs and for AEs resulting in a medically attended visit.
- The number of days with solicited events reported during the 4-day follow-up period will be tabulated for each solicited event, after each dose using descriptive statistics (mean, min, Q1, median, Q3, maximum).
- The number of each solicited events (any and Grade 3) that are ongoing beyond the 4-day follow-up period will be reported with the duration in days (mean, min, Q1, median, Q3, maximum).
- The list of solicited administration site and systemic events, and definition of intensity are described in Section 10.3.3 and 10.3.9.1 of the protocol.
- The number and percentage of participants with at least one report of SAE classified by the MedDRA Primary SOC, HLT and PTs and reported within 30 days following each vaccination will be tabulated with the exact 95% CI. The same tabulation will be presented for pIMDs.

The measurement of erythema/swelling (in mm) and fever (in °C/F) will be categorized as follows:

Table 7 Intensity grading scale for solicited events

| Grading | Erythema/swelling | Fever |
|---------|-------------------|---------------------------------------|
| 0: | ≤ 20 mm | < 38.0°C (100.4°F) |
| 1: | > 20 - ≤ 50 mm | ≥ 38.0°C(100.4°F) - ≤ 38.5°C(101.3°F) |
| 2: | > 50 - ≤ 100 mm | > 38.5°C(101.3°F) - ≤ 39.0°C(102.2°F) |
| 3: | > 100 mm | > 39.0°C(102.2°F) |

#### Combined Solicited events and Unsolicited AEs

For clinicaltrials.gov and EudraCT posting purposes, a summary of combined solicited and unsolicited non-serious adverse events will be produced by System Organ Class and preferred terms and according to occurrence of each event.

Solicited events will be coded by MedDRA as per the following codes:

| Solicited event | Lower level term code | Corresponding Lower level term decode |
|---|---|---|
| Pain | 10022086 | Injection site pain |
| Erythema | 10022061 | Injection site erythema |
| Swelling | 10053425 | Injection site swelling |
| Fever | 10016558 | Fever |
| Headache | 10019211 | Headache |
| Fatigue | 10016256 | Fatigue |
| Myalgia | 10028411 | Myalgia |
| Arthralgia | 10003239 | Arthralgia |

#### 5.4.5.1. Concomitant Medication

Medications will be coded using the GSKDRUG dictionary.

#### 5.4.6. **Sensitivity Analyses**

If more than 10% of participants miss the revaccination dose or don't have safety data reported after revaccination, the safety analysis described in section 5.4.4 will also be conducted on participants with full follow-up (attending all study visits).

The goal of this sensitivity analysis is to determine the extent to which results might be impacted by considering the different scenarios.

#### 6. ANALYSIS INTERPRETATION

All analyses are descriptive.

#### 7. INTERIM ANALYSES

#### 7.1. Sequence of analyses

Analyses to evaluate objectives and endpoints will be performed stepwise:

- **Month 6:** A first analysis will be performed on all reactogenicity, safety and immunogenicity data available and as clean as possible, when data for at least primary and secondary endpoints up to Month 6 are available for all participants. This analysis will be considered as final for those endpoints. \*
- Month 13: A second analysis will be performed on all reactogenicity, safety and immunogenicity data available and as clean as possible, when data for at least primary and secondary endpoints up to Month 12 are available for all participants, as well as data up to 1 month after the first revaccination (Month 13) in the RSV annual group. This analysis will be considered as final for those endpoints \*.

- Month 18: A third analysis will be performed on all safety and/or immunogenicity data available and as clean as possible, when data for secondary endpoints up to Month 18 are available for all participants. This analysis will be considered as final for those endpoints \*. Safety and immunogenicity analysis may be performed at different time depending on data availability.
- Month 25: A fourth analysis will be performed on all safety, reactogenicity and immunogenicity data available and as clean as possible, when data for at least primary and secondary endpoints up to Month 24 are available for all participants, as well as data up to 1 month after the second revaccination (Month 25) in the RSV\_annual group and up to 1 month after the first revaccination (Month 25) in the RSV\_flexible revaccination group. This analysis will be considered as final for those endpoints \*.
- The final **End of Study** analysis will be performed when all reactogenicity, safety and immunogenicity data for at least primary and secondary endpoints up to study conclusion are available for all participants (Month 36).
- If the data for tertiary endpoints become available at a later stage, (an) additional analysis/analyses will be performed.
- \*Each analysis can be considered as final, as it is based on data that is as clean as possible. However, the consecutive analysis of the same time point might slightly differ at the next analysis e.g when M6 data are re-analyzed at the time of M13 analysis. If major changes are identified, they will be described in the clinical study report.

| Description | Analysis | Disclosure Purpose |
|---|---|---|
| | ID | (CTRS=public posting, SR=study report, internal) |
| End of study analysis | E1_01 | CTRS, SR |
| Analysis up to Month 6 | E1_02 | SR |
| Analysis up to Month 13 | E1_03 | CTRS, SR |
| Analysis up to Month 18 | E1_04 | Internal |
| Analysis up to Month 25 | E1_05 | Internal |

# 7.2. Statistical considerations for interim analyses

All analyses will be conducted on final data (as clean as possible) and therefore no statistical adjustment for interim analyses is required.

# 8. CHANGES TO THE PROTOCOL DEFINED STATISTICAL ANALYSIS

This statistical analysis plan complements the analyses described in the protocol.

The changes compared to the planned statistical analysis specified in the Protocol amendment 1 (Dated: 01 April 2022) are described below:

• The number and percentage of participants with at least one administration site event (solicited only), with at least one systemic event (solicited only) and with any solicited event during the 4-day follow-up period after vaccination

- Related SAEs/pIMDs and Fatal SAEs will be tabulated after each dose.
- SAEs/pIMDs within 30 days following each vaccination.

# 9. NON-STANDARD DATA DERIVATION RULES AND STATISTICAL METHODS

The following sections describe additional derivation rules and statistical methods which are not presented in Section 10.1 (Business rules for standard data derivations and statistical methods).

## 9.1. Handling of missing data

#### 9.1.1. Dates

When partially completed dates (i.e. with missing day or month) are used in calculations, the following rules will be applied:

- AE start dates with missing day:
  - If the month is not the same as the vaccine dose, then the imputed start date will be the 1<sup>st</sup> of the month
  - If the event starts in the same month as the vaccine dose, the flag indicating if the event occurred before or after vaccination (AE.AESTRTPT) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the vaccine dose given during that month. If 'before vaccination' is selected, the imputed date will be one day before the vaccine dose given during that month.
- AE start dates with missing day and month:
  - If the year is not the same as the vaccine dose, then the imputed start date will be the 1<sup>st</sup> of January.
  - If the event starts in the same year as the vaccine dose, the flag indicating if the event occurred before or after vaccination (AE.AESTRTPT) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first vaccine dose given during that year. If 'before vaccination' is selected, the imputed date will be one day before the first vaccine dose given during that year.
- AE end dates with missing day: the imputed end date will be the last day of the month (30 or 31) or the study conclusion date whichever comes first.
- AE end dates with missing day and month: the imputed end date will be the last day of the year (31st of December) or the study conclusion date whichever comes first.

All incomplete concomitant medication/vaccination start/end date will follow the rules above.

### 10. ANNEXES

# 10.1. Business rules for standard data derivations and statistical methods

This section contains standard rules for data display and derivation for clinical and epidemiological studies.

## 10.1.1. Attributing events to vaccine doses

The dose relative to an event is the most recent study dose given to a participant prior to the start of a given event. For example, if the start date of an AE is between Dose 1 and Dose 2, the relative dose will be Dose 1.

If an event starts on the same day as a study dose, the relative dose will be derived from the additional information provided in the case report form (CRF) using the contents of the flag indicating if the event occurred before or after study dose. If 'after vaccination is selected, the relative dose for the event will be the one administered on the start day of the event. If 'before vaccination is selected, the relative dose for the event will be the dose prior to this one.

## 10.1.2. Handling of missing data

#### 10.1.2.1. Dates

When partially completed dates (i.e. dates missing a day and/or month) are used in calculations, the following standard rules will be applied:

- A missing day will be replaced by 15<sup>th</sup>
- A missing day and month will be replaced by June 30<sup>th</sup>.

See also exceptions in Section 9.1.

#### 10.1.2.2. Laboratory data

Refer to Section 5.1.2 for more details.

#### 10.1.2.3. Daily recording of solicited events

#### 10.1.2.3.1. Studies with paper diaries

For studies using paper diaries which have questions in the CRF indicating the presence or absence of solicited events, the following rules are applicable:

• Denominators for the summary of administration site (or systemic) solicited events will be calculated using the number of participants who respond "Yes" or "No" to the question concerning the occurrence of administration site (or systemic) events.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 3

- When a specific solicited event is marked as having not occurred following a specific study dose (i.e. SDTM CE.CEOCCUR=N for the specified post-dose period for the event in question), all daily measurements will be imputed as Grade 0.
- When a specific solicited event is marked as having occurred following a specific study dose (i.e. SDTM CE.CEOCCUR=Y for the specified post-dose period for the event in question), any missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the solicited event summary tables.
- When the occurrence of a specific solicited event is not present (i.e. SDTM CE.CEOCCUR is neither Y nor N for the specified post-dose period for the event in question) but the group of solicited events (administration site or systemic) is marked as having occurred (i.e. SDTM CE.CEOCCUR=Y), all missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the solicited event summary tables.

The following table shows how participants contribute to each category for a specific solicited event over the Day X to Day Y post-dose period:

| Solicited event category | Participants included in the calculation of the numerator |
|---|---|
| Any | All participants with at least one occurrence of the adverse event at grade 1, grade 2, or grade 3 between Day X and Day Y or with the adverse event marked as present and at least one missing daily recording between Day X and Day Y |
| At least grade 1 | All participants with at least one occurrence of the adverse event at grade 1, grade 2, or grade 3 between Day X and Day Y |
| At least grade 2 | All participants with at least one occurrence of the adverse event at grade 2 or grade 3 between Day X and Day Y |
| At least grade 3 | All participants with at least one occurrence of the adverse event at grade 3 between Day X and Day Y |

#### 10.1.2.4. **Unsolicited adverse events**

Unsolicited AE summaries are including SAEs unless specified otherwise.

Missing severity, relationship with study vaccine, and outcome of unsolicited AEs will not be replaced and will appear as 'UNKNOWN' when displayed in a statistical output.

#### 10.1.3. **Data derivation**

#### 10.1.3.1. Age at first dose in years

When age at first dose is to be displayed in years, it will be calculated as the number of complete calendar years between the date of birth and the date of first dose. For example:

DOB = 10SEP1983, Date of first dose = 09SEP2018 -> Age = 34 years

DOB = 10SEP1983, Date of first dose = 10SEP2018 -> Age = 35 years

In this study, we will collect only the year of birth. The rules for handling missing day and/or month in the DOB are given in Section 10.1.2.1.

Since only the year of birth will be collected in the eCRF, there might be some discrepancies between the age computed using standard derivation rules and the age category used in SBIR for the minimization.

Therefore, for the analysis by age, the age categories defined in Table 4 will be determined according to the information entered in SBIR (variable AGEGRP in SDTM SUPPDM), except for " $\geq$ 65 YOA" category which will be obtained using the derived age because this category is not used in SBIR for minimization

## 10.1.3.2. Temperature

Temperatures will be presented in degrees Celsius (°C). Temperatures reported in degrees Fahrenheit (°F) will be converted as follows:

Temperature (Celsius) =  $((Temperature (Fahrenheit) - 32) \times 5)/9$ 

## 10.1.3.3. Numerical serology results

Numerical serology results will be derived from the content of IS.ISORRES in the SDTM dataset. For humoral assays with a specific cut-off, the following derivation rules apply:

| IS.ISORRES | Derived value |
|-----------------------------------------------------|---------------|
| "NEG", "-", or "(-)" | cut-off/2 |
| "POS", "+", or "(+)" | cut-off |
| "< value" and value is <= assay cut-off | cut-off/2 |
| "< value" and value is > assay cut-off | Value |
| "> value" and value is < assay cut-off | cut-off/2 |
| "> value" and value is >= assay cut-off | Value |
| "value" and value is < cut-off | cut-off/2 |
| "value" and value is >= cut-off and value is <=ULOQ | value |
| "value" and value is > ULOQ | ULOQ* |
| All other cases | Missing |

<sup>\*</sup>This rule will be used to compute descriptive statistics (GMTs, fold increase etc).

#### 10.1.3.4. Geometric mean titers (GMTs) and concentrations (GMCs)

GMT or GMC calculations are performed by taking the inverse logarithm of the mean of the log titer or concentration transformations. Non quantifiable antibody titers or concentrations will be converted as described in Section 10.1.3.3 for the purpose of GMT/GMC calculation. Cut-off values are defined by the laboratory before the analysis.
#### 10.1.3.5. Onset day

The onset day for an event (e.g. AE, concomitant medication/vaccination) is the number of days between the last study dose and the start date of the event. This is 1 for an event occurring on the same day as a study dose (and reported as starting after study dose).

#### 10.1.3.6. Duration of events

The duration of an event with a start and end date will be the difference between the start and end date plus one day, i.e. an event that starts on 3 March 2018 and ends on 12 March 2018 has a duration of 10 days.

The duration of solicited events will be calculated as the sum of the individual days with the event reported at grade 1 or higher or reported as missing ("NOT DONE"), during the solicited event period. The duration of solicited events ongoing beyond the solicited period will be calculated as end date – start date + 1. The goal of this change was to align this text with the standard programs.

#### 10.1.3.7. Counting rules for combining solicited and unsolicited AEs

For output combining solicited and unsolicited AEs, all SAEs will be considered systemic events since the administration site flag is not included in the Expedited Adverse Event CRF pages. Unsolicited AEs with missing administration site flag will also be considered systemic.

Multiple events with the same PT which start on the same day are counted as only one occurrence.

In case a solicited event is worsening to Grade 3 after the solicited period, it should be reported only in the following table.

Summary of grade 3 AEs (solicited and unsolicited) within 30 days following each dose and overall

#### 10.1.3.8. Counting rules for occurrences of solicited events

When the occurrences of solicited events are summarized, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurs. Also, in the case of co-administered study interventions, an administration site event recorded for a participant following multiple study interventions will be counted as only one occurrence.

#### 10.1.4. Display of decimals

#### 10.1.4.1. Percentages

Percentages and their corresponding confidence limits will be displayed with one decimal except for 100% in which case no decimal will be displayed.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 3

#### 10.1.4.2. Demographic/baseline characteristics statistics

The mean, median, and SD for continuous baseline characteristics will be presented with one decimal.

The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values.

The maximum and minimum of transformed body temperatures will be displayed with one decimal.

## 10.1.4.3. Serological summary statistics

For each assay, GMT or GMC and their confidence limits will be presented with one decimal, as well as GMT/GMC fold increase from pre-dose.

The mean, median, SD and quartile values for frequency of RSVPreF3-specific-CD4+ and CD8+ T cells and for the fold increase (post- over pre-vaccination) will be presented with one decimal. The minimum and maximum values will be presented with no decimal.

# 10.1.5. Statistical methodology

#### 10.1.5.1. Exact confidence intervals around proportions

The exact confidence intervals around within-group proportions are derived using the method of Clopper and Pearson [Clopper, 1934].

# 11. ADDITIONAL ANALYSES DUE TO THE COVID-19 PANDEMIC

Depending on how the COVID-19 situation evolves, the SAP might be amended to reflect the analysis corresponding to COVID-19.

## 12. REFERENCES

Clopper CJ, Pearson E. The Use of Confidence or Fiducial Limits Illustrated in the case of the Binomial. *Biometrika*. 1934;26:404-13.

David M-P, Van Herck K, Hardt K, Tibaldi F, Dubin G, Descamps D, et al. Long-term persistence of anti-HPV-16 and-18 antibodies induced by vaccination with the AS04-adjuvanted cervical cancer vaccine: modeling of sustained antibody responses. GYNECOLOGIC ONCOLOGY. 2009;115(3):S1–6.

Fraser C, Tomassini JE, Xi L, Golm G, Watson M, Giuliano AR, et al. Modeling the long-term antibody response of a human papillomavirus (HPV) virus-like particle (VLP) type 16 prophylactic vaccine. Vaccine 2007 May 22;25(21):4324-33

Pan W Akaike's information criterion in generalized estimating equations Biometrics, 57 (1) (2001), pp. 120-125

Rubin, D. B., Stern, H. S. AND Vehovar, V. Handling "don't know" survey responses: the case of the Slovenian plebiscite. Journal of the American Statistical Association 90, 1995, 822–828

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 2

| | Statistical Analysis Plan Amendment 2 |
|---|---|
| gsk | Statistical Analysis Plan |
| Title: | A phase 3, randomized, open-label, multi-country study to evaluate the immunogenicity, safety, reactogenicity and persistence of a single dose of the RSVPreF3 OA investigational vaccine and different revaccination schedules in adults aged 60 years and above. |
| eTrack study number and<br>Abbreviated Title | 212496 (RSV OA=ADJ-004) |
| Scope: | All data pertaining to the above study except the Safety Review Team analyses for the first 50 participants aged 80 years and above |
| Date of Statistical Analysis<br>Plan | Amendment 2 Final: 20 Jun 2022 |

APP 9000058193 Statistical Analysis Plan Template V5 (Effective date: 1July2020)

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 2

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| LIS | ST OF A | ABBREV | IATIONS | 6 |
| 1. | DOCU | JMENT H | HISTORY | 7 |
| 2. | OBJE | CTIVES | ENDPOINTS | 8 |
| 3. | STUD<br>3.1. | | GNdesign | |
| 4. | ANAL<br>4.1.<br>4.2. | Definition | frs | 12<br>12<br>12 |
| 5. | STAT<br>5.1. | | Immunogenicity | 17<br>17 |
| | 5.2. | Analysis 5.2.1. 5.2.2. | s of demography and baseline characteristics | 19<br>19 |
| | 5.3. | Primary<br>5.3.1. | endpoint(s) Analysis planned in the protocol 5.3.1.1. Humoral immune response – up to Month 12 | 20<br>20 |
| | 5.4. | Second 5.4.1. 5.4.2. 5.4.3. | <ul> <li>5.4.3.1. Mixed effects model</li></ul> | 20<br>21<br>22<br>22 |
| | | 5.4.4.<br>5.4.5.<br>5.4.6. | after dose 1 | 27<br>29<br>30 |
| 6 | ΔΝΔΙ | YSIS IN | TERPRETATION | 30 |

| | | | | Otatistical Allarysis i lali Allicha | IIICIIL 2 |
|---|---|---|---|---|---|
| 7. | INTER | RIM ANA | LYSES | · | |
| | 7.1. | Sequen | ce of analy | /ses | 30 |
| | 7.2. | | | rations for interim analyses | |
| 0 | CHAN | ICES TO | THE DDC | DIOCOL DEFINED STATISTICAL | |
| 8. | ANIAI | VOIC | I I I PRO | OTOCOL DEFINED STATISTICAL | 21 |
| | ANAL | .1313 | | | ا د |
| 9. | NON- | STANDA | ARD DATA | DERIVATION RULES AND STATISTICAL | |
| | METH | HODS | | | 32 |
| | 9.1. | | | ıg data | |
| | | 9.1.1. | Dates | | 32 |
| 10 | ANNE | XES | | | 33 |
| | 10.1. | | | standard data derivations and statistical | |
| | | method | S | | 33 |
| | | | | g events to vaccine doses | |
| | | 10.1.2. | Handling | of missing data | 33 |
| | | | | Dates | |
| | | | 10.1.2.2. | Laboratory data | 33 |
| | | | 10.1.2.3. | Daily recording of solicited events | 33 |
| | | | | 10.1.2.3.1. Studies with paper diaries | 33 |
| | | | 10.1.2.4. | Unsolicited adverse events | |
| | | 10.1.3. | | vation | |
| | | | 10.1.3.1. | Age at first dose in years | 34 |
| | | | | Temperature | |
| | | | | Numerical serology results | |
| | | | | Geometric mean titers (GMTs) and | |
| | | | | concentrations (GMCs) | 35 |
| | | | 10.1.3.5. | Onset day | |
| | | | 10.1.3.6. | Duration of events | 36 |
| | | | | Counting rules for combining solicited and | |
| | | | | unsolicited AEs | 36 |
| | | | 10.1.3.8. | Counting rules for occurrences of solicited | |
| | | | | events | |
| | | 10.1.4. | Display o | f decimals | |
| | | | | Percentages | |
| | | | | Demographic/baseline characteristics | |
| | | | | statistics | 36 |
| | | | 10 1 4 3 | Serological summary statistics | |
| | | 10.1.5. | Statistica | I methodology | 37 |
| | | | 10 1 5 1 | Exact confidence intervals around | |
| | | | | proportions | 37 |
| | | | | FF 3. 40. | |
| 11. | ADDI <sup>*</sup> | TIONAL | ANALYSE | S DUE TO THE COVID-19 PANDEMIC | 37 |
| | | | | - | |
| 12. | REFE | RENCES | S | | 38 |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 2

# **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | Study groups, intervention and blinding foreseen in the study | 10 |
| Table 2 | Group names and definition for footnote in the TFLs | 10 |
| Table 3 | Pooled group names and definition for footnote in the TFLs | 11 |
| Table 4 | Sub-group names and definitions for footnote in the TFLs | 11 |
| Table 5 | Populations for analyses | 12 |
| Table 6 | List of elimination codes | 13 |
| Table 7 | Intensity grading scale for solicited events | 29 |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 2

# **LIST OF FIGURES**

| | | PAGE |
|----------|-----------------------|------|
| Figure 1 | Study design overview | 9 |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 2

# LIST OF ABBREVIATIONS

**AE** Adverse event

**AESI** Adverse Events of Special Interest

**ANCOVA** Analysis of Covariance

**CD** Community Dwelling

CI Confidence Interval

**COVID-19** Coronavirus Disease 2019

**CRF** Case Report Form

CTRS Clinical Trial Registry Summary

Eli Type Internal database code for type of elimination code

**ELISA** Enzyme-linked immunosorbent assay

EU/mL ELISA unit per milliliter

**ES** Exposed Set

**GMC** Geometric mean antibody concentration

**GMT** Geometric mean antibody titer

**GSK** GlaxoSmithKline

IU/mL International units per milliliter

LL Lower Limit of the confidence interval

**MedDRA** Medical Dictionary for Regulatory Activities

NA Not Applicable

**PD** Protocol Deviation

**PPS** Per-Protocol Set

**SAE** Serious adverse event

**SAP** Statistical Analysis Plan

SBIR GSK Biologicals Internet Randomization System

**SD** Standard Deviation

**SDTM** Study Data Tabulation Model

UL Upper Limit of the confidence interval

# 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|---|---|---|
| Date Description First version Amendment 1: Amendment 2: The study design (Figure 1) was updated with the addition of a revaccination dose at Month 24 and a new follow-up visit at Month 25 for the RSV_flexible revaccination group. (Section 3.1). Table 1 was updated with the addition of a revaccination dose at Month 24 for the RSV_flexible revaccination group (Section 3.1). | | Protocol Version Final: 28 October 2020 Final: 28 October 2020Final Amendment 1: 01 April 2022 |
| | <ul> <li>(Section 3.1).</li> <li>Table 6 was updated with the addition of RSV_flexible revaccination group at Months 24 and 25 to the list of elimination codes</li> <li>SAEs/pIMDs within 30 days following each vaccination (Section 5.4.5)</li> </ul> | |

# 2. OBJECTIVES/ENDPOINTS

| Objectives | Endpoints |
|---|---|
| Prim | |
| To evaluate the humoral immune response following a 1-dose primary schedule of RSVPreF3 OA investigational vaccine up to 12 months post-Dose 1. | Humoral immune response at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), and at 6 and 12 months post-Dose 1 (Months 6 and 12), in a subset of participants: Neutralizing antibody titers against RSV-A Neutralizing antibody titers against RSV-B. |
| Seco | ondary |
| To further evaluate the humoral immune response following a 1-dose primary schedule of RSVPreF3 OA investigational vaccine up to 12 months post-Dose 1. | Humoral immune response at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), and at 6 and 12 months post-Dose 1 (Months 6 and 12), in a subset of participants: RSVPreF3-specific Immunoglobulin G (IgG) antibody concentrations. |
| To evaluate the humoral immune response following 1 dose of the RSVPreF3 OA investigational vaccine and following revaccination doses, up to study end. | Humoral immune response at Months 18, 24, 30 and 36 post-Dose 1, and at 1 month after each revaccination dose (Months 13 and 25), in a subset of participants: Neutralizing antibody titers against RSV-A and RSV-B RSVPreF3-specific IgG antibody concentrations. |
| To evaluate the cell-mediated immune (CMI) response following 1 dose of the RSVPreF3 OA investigational vaccine and following revaccination doses up to study end. | <ul> <li>CMI response at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), at Months 6, 12, 18, 24, 30 and 36 post-Dose 1, and at 1 month after each revaccination dose (Months 13 and 25), in a subset of participants:</li> <li>Frequency of RSVPreF3-specific CD4+ and/or CD8+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 4-1BB, IL-2, TNF-α, IFN-γ, IL-13, IL-17.</li> </ul> |
| To evaluate the safety and reactogenicity of each vaccination schedule of the RSVPreF3 OA investigational vaccine in all participants. | <ul> <li>Occurrence of each solicited administration-site and systemic event during a 4-day follow-up period (i.e., on the day of vaccination and 3 subsequent days) after each vaccination.</li> <li>Occurrence of any unsolicited AE during a 30-day follow up period (i.e., on the day of vaccination and 29 subsequent days) after each vaccination.</li> <li>Occurrence of all SAEs and pIMDs up to 6 months after each vaccination.</li> <li>Occurrence of fatal SAEs, related SAEs and related pIMDs from first vaccination (Day 1) up to study end (Month 36).</li> </ul> |
| Tertiary | |
| To further characterize immune responses to the RSVPreF3 OA investigational vaccine. | Any further exploratory immunology in a subset of participants, such as, but not limited to: Antibodies against specific protein F epitopes. Potential new immunological markers for protection. Frequency of RSVPreF3-specific CD4+ and/or CD8+ T cells expressing one or any combination of immune marker(s) **SAF = periods adverse event in IMD = petential immune mediated.** |

CMI = cell-mediated immunity, AE = adverse event, SAE = serious adverse event, pIMD = potential immune-mediated disease.

#### 3. STUDY DESIGN

# 3.1. Overall design

Figure 1 Study design overview



N = number of participants; D = day; M = month; AE = adverse event; HI = humoral immunity; CMI = cell-mediated immunity; pIMD = potential immune-mediated disease; SAE = serious adverse event.

= blood sample for humoral immune responses (only applicable for ~ 345 participants of the RSV\_annual group; and for all participants of the RSV flexible revaccination and RSV 1dose groups)

= blood sample for CMI (only applicable for ~345 participants of the RSV\_annual group, and for ~115 participants each from the RSV flexible revaccination and RSV 1dose groups).

Note: For group RSV\_annual: Revaccination Year 1 = Month 12; Revaccination Year 2 = Month 24; for group RSV\_flexible revaccination: Revaccination Year 2 = Month 24.

\*Visit and follow-up of solicited events, unsolicited AEs, SAEs and pIMDs are only applicable for RSV\_annual group.

\*\*Visit and follow-up of solicited events, unsolicited AEs, SAEs and pIMDs are only applicable for RSV\_annual and RSV flexible revaccination groups.

\*\*\*For the RSV\_annual group, the same ~345 participants will be part of both the HI and CMI subsets. The remaining ~645 participants will have no blood draws and will only be followed up for safety and reactogenicity.

\*\*\*\*\*For those participants in the RSV\_annual group without blood sample collections, visits at Months 6, 18, 30 and 36 may be held through a contact. However, contact should be attempted only if site visit is not possible at Months 6, 18, 30 and 36.

- Type of study: self-contained.
- Experimental design: Phase 3, randomized, open-label, multi-country study with 3 parallel groups (see Figure 1).
- **Duration of the study**: ~ 36 months for each participant.
- **Primary completion date**: Month 12.
- Control: none.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 2

- **Blinding**: open-label. Refer to the protocol for details.
- **Data collection**: standardized electronic Case Report Form (eCRF). Solicited events and unsolicited adverse events (AEs) will be collected using a participant Diary card (paper Diary card).
- Safety monitoring: the study will be conducted with oversight by the project Safety Review Team (SRT). Please refer to protocol for the description of review of safety data by the SRT.
- Study groups: refer to Figure 1 and Table 1 for an overview of the study groups

Table 1 Study groups, intervention and blinding foreseen in the study

| | Study Groups Number of participants Age | | Intervention | | | Blinding |
|---|---|---|---|---|---|---|
| Study Groups | | | Primary vaccination | Revaccination<br>Year 1 (Month<br>12) | Revaccination<br>Year 2 (Month<br>24) | Open |
| RSV_annual* | ~990 | ≥60 years | RSVPreF3 OA investigational vaccine | RSVPreF3 OA investigational vaccine | RSVPreF3 OA investigational vaccine | Х |
| RSV_flexible revaccination | ~330 | ≥60 years | RSVPreF3 OA investigational vaccine | (none) | RSVPreF3 OA investigational vaccine | Х |
| RSV_1dose | ~330 | ≥60 years | RSVPreF3 OA investigational vaccine | (none) | (none) | Х |

<sup>\*</sup> RSV\_annual group will be split in 3 technical groups in SBIR in order to have a randomization ratio of 1:1:1:1: for treatment allocation and avoid predictability.

• **Groups and sub-groups definition for analysis:** Refer to the tables below for a description of the groups and subgroups labels that will be used in the Tables Figures and Listings (TFLs).

The analyses pertaining to timepoints up to Month 12 will be performed for each group and for the 3 groups pooled. From Month 13 up to study end, the analyses will be performed by group.

The following group names will be used in the TFLs:

Table 2 Group names and definition for footnote in the TFLs

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | RSV_annual | Participants receiving the first dose (Dose 1) of RSVPreF3 OA investigational vaccine at Day 1, followed by a revaccination dose at 12 months post-Dose 1 and at 24 months post-Dose 1 |
| 2 | RSV_flexible revaccination | Participants receiving the first dose (Dose 1) of RSVPreF3 OA investigational vaccine at Day 1 and a revaccination dose at 24 months post-Dose 1 |
| 3 | RSV_1dose | Participants receiving a single dose (Dose 1) of RSVPreF3 OA investigational vaccine at Day 1 |

Table 3 Pooled group names and definition for footnote in the TFLs

| Pooled Group label in tables | Groups to be pooled | Pooled definition for footnote | Comment |
|---|---|---|---|
| Total | RSV_annual,<br>RSV_flexible<br>revaccination and<br>RSV_1dose | Participants receiving one dose of RSVPreF3 OA investigational vaccine at Day 1 in all the three groups | Applicable on data reported up to Month 12 |
| Flexible+1dose | RSV_flexible<br>revaccination, and<br>RSV_1dose | Participants receiving one dose of RSVPreF3 OA investigational vaccine at Day 1 in the RSV_flexible revaccination, and RSV_1dose groups | Applicable on data reported at Month 13, Month 18 and Month 24 |

Table 4 Sub-group names and definitions for footnote in the TFLs

| Sub-analysis | Subgroup order in tables | Subgroup label in tables | Subgroup definition for footnote |
|---|---|---|---|
| By age | 1 | ≥65YOA | ≥65 years old participants |
| | 2 | ≥70YOA | ≥70 years old participants |
| | 3 | ≥80YOA | ≥80 years old participants |
| | 4 | 60-69YOA | 60-69 years old participants |
| | 5 | 70-79YOA | 70-79 years old participants |
| By sex | 1 | Female | Female |
| | 2 | Male | Male |
| By region | 1 | North America | Participants from North America (United States of America) |
| | 2 | Europe | Participants from Europe (Finland, Germany) |
| | 3 | Asia | Participants from Asia (Japan, Taiwan) |

YOA = Years of age

## • Allocation of participants to assay subsets

Allocation of participants to assay subsets will be performed using SBIR. The subsets are detailed below.

| | RSV_annual | RSV_flexible revaccination | RSV_1dose |
|---|---|---|---|
| HI subset | ~345* | All participants (~330) | All participants (~330) |
| CMI subset | ~345* | ~115 | ~115 |

<sup>\*</sup>For the RSV\_annual group, the same ~345 participants will be part of both the HI and CMI subsets. The remaining ~645 participants will have no blood draws, and will only be followed up for safety and reactogenicity.

- HI subset: ~345 participants from the RSV\_annual group, and all participants from the RSV\_flexible revaccination and RSV\_1dose groups. These participants will have blood samples collected for testing of humoral immunity at each visit applicable for their study group.
- **CMI subset**: ~345 participants from the RSV\_annual group, and ~115 participants each from the RSV\_flexible revaccination and RSV\_1dose groups. These participants will have additional blood samples collected for CMI testing at each visit applicable for their study group.

#### 4. ANALYSIS SETS

#### 4.1. Definition

Table 5 Populations for analyses

| Analysis set | Description |
|---|---|
| Enrolled set | Participants who agreed to participate in a clinical study after completion of the |
| | informed consent process. |
| Exposed set (ES) | All participants who received at least 1 dose of the study intervention. The |
| , , | allocation in a group is done in function of the administered intervention. |
| Per Protocol set (PPS) | All participants who received at least 1 dose of the study intervention to which they |
| , , | are randomized and have post-vaccination data, minus participants with protocol |
| | deviations that lead to exclusion. |

The primary analysis for immunogenicity will be performed on the Per Protocol set (PPS). If the percentage of vaccinated participants with serological results excluded from the PPS for immunogenicity is at least 5% for at least 1 visit and at least 1 group, a second analysis will be performed on the Exposed Set (ES). The immunogenicity analysis will be performed overall, by sex, by age category (age at Dose  $1: \ge 65 \text{ YOA}, \ge 70 \text{ YOA}, \ge 80 \text{ YOA}, 60-69 \text{ YOA}$  and 70-79 YOA, and by region (North America, Europe, Asia).

# 4.2. Criteria for eliminating data from Analysis Sets

#### 4.2.1. Elimination from ES

Code 1030 (Study intervention not administered at all), 800 (Fraudulent data) and code 900 (Invalid informed consent) will be used for identifying participants eliminated from the ES.

# 4.2.2. Elimination from Per-protocol analysis Set (PPS)

## 4.2.2.1. Excluded participants

A participant will be excluded from the populations of analysis under the following conditions

- For codes 800, 900, 1030 and 1050: participants will be eliminated for all visits.
- For codes 1040, 1070, 1080, 1090, 2010, 2040, 2050, 2080: participants will be eliminated from a specific visit (at which the condition is met) onwards.
- For codes 2090, 2100, 2120: participants will be eliminated at the specific visit at which the condition is met.

# Table 6 List of elimination codes

| Code | Condition under which the code is used | Visit (timepoints) where the code is checked | Applicable for analysis set |
|---|---|---|---|
| 800 | Fraudulent data | All | ES and PPS |
| 900 | Invalid informed consent | All | ES and PPS |
| 1030 | Study intervention not administered at all | All | ES and PPS |
| 1040 | Administration of concomitant vaccine(s) forbidden in the protocol | All | PPS |
| | Any investigational or non-<br>registered vaccine other than<br>the study vaccine used during<br>the study period beginning 30<br>days before the first dose of<br>study vaccine, or planned use<br>during the study period. | | |
| | • Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before each dose and ending 30 days after each dose of study vaccine administration, with the exception of inactivated, split virion and subunit influenza vaccines which can be administered up to 14 days before or from 14 days after each study vaccination. | | |
| | Previous vaccination with an<br>RSV vaccine | | |
| 1050 | Randomization failure | Day 1 | PPS |
| 1070 | Vaccine administration not according to protocol | Vaccination visits at Day 1, Month 12, and 24 | PPS |
| | <ul> <li>Incomplete vaccination course</li> <li>Participant was vaccinated with the correct vaccine but containing a lower volume</li> </ul> | Months 12 and 24 are applicable to the RSV_annual group and Month 24 applies | |

| <u> </u> | Statistical Analysis Plan Amendmen | | |
|---|---|---|---|
| Code | Condition under which the code is used | Visit (timepoints) where the code is checked | Applicable for analysis set |
| | Participant was re-vaccinated while it was not planned | to the RSV_flexible revaccination group | |
| | Route of the study intervention is not intramuscular | | |
| | Wrong reconstitution of<br>administered vaccine | | |
| 1080 | Vaccine administration after a Temperature deviation | Day 1, Month 12, and 24 | PPS |
| | Vaccine administered despite<br>a Good Manufacturing<br>Practices (GMP) no-go<br>temperature deviation | Months 12 and 24 are applicable to the RSV_annual group and Month 24 applies to RSV_flexible revaccination group | |
| 1090 | Vaccine administration after expiration | Day 1, Month 12, and 24 Months 12 and 24 are applicable to the RSV_annual group and Month 24 belongs to the RSV_flexible revaccination group | PPS |
| 2010 | Protocol deviation linked to inclusion/exclusion criteria | All | PPS |
| 2040 | <ul> <li>Administration of any medication forbidden by the protocol</li> <li>Any investigational or non-registered medication used during the study period</li> <li>Administration of long-acting immune-modifying drugs at any time during the study period (e.g. <i>infliximab</i>)</li> <li>Immunoglobulins and/or any blood products administered during the study period</li> </ul> | All | PPS |

| | | Statistical Analysis Plan Amendmen | |
|---|---|---|---|
| Code | Condition under which the code | Visit (timepoints) | Applicable for |
| | is used | where the code is | analysis set |
| | | checked | |
| | • Chronic administration (defined as more than 14 consecutive days in total) of immunosuppressants or other immune-modifying drugs during the period starting 90 days prior to the study vaccine administration or planned administration during the study period. For corticosteroids, this will mean prednisone ≥20 mg/day, or equivalent. | | |
| 2050 | Intercurrent medical condition | All | PPS |
| | • Participants may be eliminated from the PPS for immunogenicity if, during the study, they incur a condition that has the capability of altering their immune response (intercurrent medical condition) or are confirmed to have an alteration of their initial immune status. | | |
| 2080 | Participants did not comply with dosing schedule | Month 12 and 24 | PPS |
| | RSV_annual: number of days between dose 1 and revaccination dose at Month 12 is outside [350-380 days] | | |
| | • RSV_annual and RSV_flexible revaccination: number of days between dose 1 and revaccination dose at Month 24 is outside [715-745 days] | | |
| 2090 | Participants did not comply with blood sample schedule | Day 31, Month 6, 12, 13, 18, 24, 25, 30, 36 | PPS |
| | • Number of days between dose 1 and Day 31 blood sample is outside [30-42 days] | | |

| | Statistical Analysis Plan Amendme | | |
|---|---|---|---|
| Code | Condition under which the code | Visit (timepoints) | Applicable for |
| | is used | where the code is | analysis set |
| | | checked | |
| | • Number of days between dose 1 and Month 6 blood sample is outside [180-210 days] | | |
| | • Number of days between dose 1 and Month 12 blood sample is outside [350-380 days] | | |
| | Number of days between Month 12 and Month 18 blood sample is outside [180-210 days] | | |
| | Number of days between dose 1 and Month 24 blood sample is outside [715-745 days] | | |
| | Number of days between Month 24 and Month 30 blood sample is outside [180-210 days] | | |
| | Number of days between dose<br>1 and Month 36 blood sample<br>is outside [1080-1110 days] | | |
| | For RSV_annual group only: | | |
| | Number of days between<br>revaccination at Month 12 and<br>Month 13 blood sample is<br>outside [30-42 days] | | |
| | For RSV_annual and RSV_flexible | | |
| | groups: | | |
| | Number of days between<br>revaccination at Month 24 and<br>Month 25 blood sample is<br>outside [30-42 days] | | |
| 2600* | Participants not included in the humoral immunogenicity subset | Day 1, 31, Month 6, 12, 13, 18, 24, 25, 30, 36 | PPS |
| 2700* | Participants not included in the cell-mediated immune response subset | Day 1, 31, Month 6, 12, 13, 18, 24, 25, 30, 36 | PPS |
| 2100 | <ul> <li>Serological results not available</li> <li>No immunological result at visit x for all the following</li> </ul> | Day 1, Day 31,<br>Month 6, 12, 13, 18,<br>24, 25, 30, 36 | PPS |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 2

| Code | Condition under which the code | Visit (timepoints) | Applicable for |
|---|---|---|---|
| | is used | where the code is checked | analysis set |
| | tests: RSV A/B Neutralizing antibody titer, RSVPreF3-specific IgG antibody concentration and RSVPreF3-specific CD4+/CD8+ T cells frequency | Month 13 and 25 are applicable to the RSV_annual and only Month 25 is applicable to the RSV_flexible revaccination group | |
| 2120 | Obvious incoherence or abnormality or error in laboratory data • Unreliable released data as a result of confirmed sample mismatch or confirmed inappropriate sample handling at laboratory | Day 1, 31, Month 6, 12, 13, 18, 24, 25, 30, 36 | PPS |

<sup>\*</sup> codes 2600 and 2700 are not considered as protocol deviations, but those codes will be used to identify participants that are not part of the immunogenicity subsets.

#### 5. STATISTICAL ANALYSES

Standard data derivation rules and stat methods are described in Section 10.1 while the study specific data derivation rules and stat methods are described in Section 9.

For the sake of analysis, data up to Month 12 will be analyzed by group (RSV\_annual, RSV\_flexible revaccination and RSV\_1dose), and also the 3 groups will be pooled. For Month 13, Month 18 and Month 24, the analyses will be tabulated for RSV\_annual group versus the pooled RSV\_flexible revaccination and RSV\_1dose groups. From Month 25 up to study end, the analyses will be performed by group

If more than 5% of participants in the RSV\_annual and RSV\_flexible revaccination groups receive different number of doses, an analysis by subgroup according to the number of dose(s) administered might be performed. The goal of this analysis is to describe the characteristics of participants in the RSV\_annual and RSV\_flexible revaccination groups who ultimately receive different numbers of revaccination doses in order to rule out the possibility of systematic differences between these subgroups.

#### 5.1. General considerations

## 5.1.1. Demography

For a given participant and a given demographic variable, missing measurements will not be replaced.

# 5.1.2. Immunogenicity

- Any missing or non-evaluable immunogenicity measurement will not be replaced. The descriptive analysis performed for each assay at each timepoint will exclude participants with a missing or non-evaluable measurement. This is applicable to the standard way of computing geometric mean titers/concentrations (GMTs/GMCs).
- During the computation of GMTs/GMCs from the mixed effects model (Section 5.4.3.1). Multiple imputation (MI) technique will not be applied for any missing immunogenicity measurement. This is because the mixed effects model inherently accounts for the missingness, under the assumption that the missing data are missing at random (MAR). Thus considering that missing data are MAR is a reasonable assumption for this descriptive clinical trial, then it is not necessary to perform MI [Rubin et al., 1995]
- The GMTs/GMCs will be computed by taking the anti-logarithm of the arithmetic mean of the log<sub>10</sub> transformed titers/concentrations.
- A seronegative participant will be defined as a participant whose antibody titer/concentration is below the technical cut-off value of the assay. A seropositive participant is a participant whose antibody titer/concentration is greater than or equal to the technical cut-off value of the assay.
- Antibody titers/concentrations below the technical assay cut-off will be given an arbitrary value of half the technical assay cut-off for the purpose of GMT/GMC calculation.
- Antibody titers/concentrations above the Upper Limit of Quantification (ULOQ) value will be given the ULOQ value for the purpose of GMT/GMC calculation.
- The mean geometric increase (MGI) is calculated by the geometric mean of ratios of antibody titers/concentrations of each post vaccination time point over pre vaccination (Day 1).

# 5.1.3. Reactogenicity/Safety

- For a given participant and the analysis of solicited events within 4 days post-vaccination, missing or non-evaluable measurements will not be replaced. Therefore, the analysis of solicited events will include only vaccinated participants with documented solicited safety data (i.e., paper diary completed).
- For analysis of unsolicited AEs, serious adverse events (SAEs), potential immunemediated diseases (pIMDs) and concomitant medications, all vaccinated participants will be considered. Participants who did not report an event or concomitant medication will be considered as participants without the event or the concomitant medication, respectively.

# 5.2. Analysis of demography and baseline characteristics

# 5.2.1. Analysis planned in the protocol

Descriptive summaries will be performed for each group (RSV\_annual, RSV\_flexible revaccination and RSV\_1dose) and overall. The same will be performed in each subset (humoral immune subset and CMI subset).

Demographic/baseline characteristics (age at vaccination in years, sex, race, ethnicity, type of residence (CD/LTCF) and smoking status) will be summarized using descriptive statistics:

- Frequency tables will be generated for categorical variables such as race.
- Mean, median, standard deviation and range will be provided for continuous data such as age.

The distribution of participants will be tabulated as a whole and per group, for each age category, and for each subset.

The number of doses of the study intervention administered will be tabulated by group and by visit.

Withdrawal status will be summarized by group using descriptive statistics:

- The number of participants enrolled into the study as well as the number of participants excluded from Per Protocol (PP) analyses will be tabulated.
- The numbers of participants withdrawn from the study will be tabulated according to the reason for withdrawal.

Participant disposition in the ES and PPS will be reported as a whole and per group

The number and percentage of participants using concomitant medication (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) during the 4-day follow-up period (i.e., on the day of vaccination and 3 subsequent days) and during the 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) will be summarized by group after each vaccine dose and after the revaccination.

#### 5.2.2. Additional considerations

- The analysis of demographic characteristics by group will be performed on the ES and on the PPS.
- Demography and baseline characteristics will also be summarized by sex and region.
- A summary of important protocol deviations leading to elimination from any analyses will be provided by group, based on the Enrolled Set.
- Medical history will be tabulated by System Organ Class (SOC), High Level Term (HLT) and Preferred Term (PT).

# 5.3. Primary endpoint(s)

#### 5.3.1. Analysis planned in the protocol

The primary analysis for immunogenicity will be performed on the PPS. If the percentage of vaccinated participants with serological results excluded from the PPS for immunogenicity is at least 5% for at least 1 visit and at least 1 group, a second analysis will be performed on the ES.

#### 5.3.1.1. Humoral immune response – up to Month 12

The analysis of the primary vaccination timepoints up to Month 12 will be performed for each group and for the 3 groups pooled. For each timepoint with blood sample collection for humoral immune response up to Month 12 and for each assay (RSV-A/-B neutralization assays), unless otherwise specified, the following analyses will be performed:

#### Within groups evaluation:

- Percentage of participants with antibody titers/concentrations above or equal to the technical assay cut-off and their exact 95% confidence interval (CI) will be tabulated.
- GMTs/GMCs and their 95% CI will be tabulated and represented graphically. Furthermore, to account for all the timepoints at which the blood samples are collected, a mixed effects model (see Section 5.4.3.1) will be fitted, from which the GMTs/GMCs will be computed.
- Antibody titers/concentrations will be displayed using reverse cumulative curves.
- The MGI i.e. geometric mean of ratios of antibody titer/concentrations will be tabulated with 95% CI.

# 5.4. Secondary endpoint(s)

# 5.4.1. Humoral immune response

The same analyses as described above for the primary endpoint will be performed for RSVPreF3-specific IgG ELISA up to Month 12 and for each timepoint with blood sample collection for humoral immune response **from study Month 13 up to study end** and for each assay (RSVpreF3-specific IgG **ELISA and RSV-A/-B neutralization assays**). For Month 13, Month 18, and Month 24, the analyses will be tabulated for RSV\_annual group versus the pooled RSV\_flexible revaccination and RSV\_1dose groups. From Month 25 up to study end, the analyses will be performed by group.

Only the analyses requiring further clarification of the exact timepoints analyzed are summarized below:

#### Within groups evaluation:

- The MGI i.e. geometric mean of ratios of antibody titer/concentrations will be tabulated with 95% CI:
  - For each post-primary vaccination time point (at Months 18, 24, 30 and 36 when applicable) over pre-primary vaccination (Day 1),
  - For each post-revaccination time point over corresponding pre-revaccination (Months 12 and 24) in the RSV annual group,
  - For each post-revaccination timepoint over corresponding pre-revaccination (Month 24) in the RSV flexible revaccination group,
  - For 1 month post-revaccination at Month 12 (Month 13) over 1 month post-Dose 1 vaccination (Day 31) in RSV\_annual group.
  - For 1 month post-revaccination at Month 24 (Month 25) over 1 month post-revaccination at Month 12 (Month 13) in RSV annual group
  - For 1 month post-revaccination at Month 24 (Month 25) over 1 month post-Dose 1 vaccination (Day 31) in RSV\_flexible revaccination group.

In addition, the following evaluation will be performed:

• The kinetics of GMTs/GMCs will be plotted as a function of time for participants with results available at all post vaccination timepoints.

The immunogenicity analysis will be performed overall, by sex, age category (age at Dose  $1: \ge 65 \text{ YOA}, \ge 70 \text{ YOA}, \ge 80 \text{ YOA}, 60-69 \text{ YOA}$  and 70-79 YOA), and region (North America, Europe, Asia).

#### 5.4.2. Cell-mediated immune response

#### Within groups evaluation:

The following parameters will be summarized by group at each timepoint for which blood samples are collected, for the 3 groups pooled for time points up to study Month 12, for Month 13, Month 18 and Month 24, the analyses will be tabulated for RSV\_annual group versus the pooled RSV\_flexible revaccination and RSV\_1dose groups. From Month 25 up to study end, the analyses will be performed by group using descriptive statistics (N, geometric mean, min, Q1, median, Q3, max) in the CMI subset:

- Frequency of RSVPreF3-specific CD4+ and/or CD8+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13, IL-17, measured by intracellular cytokine staining (ICS) using peripheral blood mononuclear cells PBMCs.
- The kinetics of RSVPreF3-specific CD4+ T cells frequencies will be plotted as a function of time for participants with results available at all timepoints.
- Fold increase of the frequency of RSVPreF3-specific CD4+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13, IL-17, measured by ICS at each post-primary vaccination timepoint over pre-vaccination (Day 1) by group, at each post-

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 2

revaccination over the corresponding pre-revaccination (Month 12/Month 24 in the RSV\_annual group and Month 24 in the RSV\_flexible revaccination group), at one month post-revaccination over 1 month post-previous dose in the RSV\_annual group [one month post-revaccination at Month 12 (Month 13) over one month post-Dose 1 vaccination (Day 31) and one month post-revaccination at Month 24 (Month 25) over one month post-revaccination at Month 12 (Month 13)] and in the RSV\_flexible revaccination group [one month post-revaccination at Month 24 (Month 25) over one month post-Dose 1 vaccination (Day 31)].

The immunogenicity analysis will be performed overall, by sex, age category (age at Dose  $1: \ge 65 \text{ YOA}, \ge 70 \text{ YOA}, \ge 80 \text{ YOA}, 60-69 \text{ YOA}$  and 70-79 YOA, and region (North America, Europe, Asia).

#### 5.4.3. Additional considerations

#### 5.4.3.1. Mixed effects model

For the GMTs/GMCs calculation based on the mixed effects model mentioned in Section 5.3.1.1, repeated measures analysis of covariance (ANCOVA) model will be fitted including age category (60-69 YOA, 70-79 YOA and ≥80 YOA,), study group (RSV\_annual, RSV\_flexible revaccination and RSV\_1dose), sex (male and female), visit (Day 31, Months 6, 12, 13, 18, 24, 25, 30, 36), as fixed effects, pre-vaccination log10-transformed titers/concentrations as a covariate and the response variable is the post-vaccination log10-transformed titers/concentrations. The PROC MIXED procedure in SAS® will be used to carry out the ANCOVA.

The following SAS codes will be used:

For the analysis by study group, study group and visit will be included as the fixed effects in the model

```
Analysis by group
PROC MIXED DATA=SERO method=reml empirical;
CLASS subjid group visit;
MODEL post-vac=pre-vacc group visit visit*group/ noint s cl;
RANDOM intercept/ subject=usubjid g v vcorr type = un;
REPEATED visit/type=unsubject=subjid;
LSMEANS visit*group/ E cl;
ODS OUTPUT LSMEANS=LS;
RUN;
```

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 2

For the analysis by age category, age category and visit will be included as the fixed effects in the model. However, this is only applicable at timepoints where the 3 study groups will be pooled. Otherwise for the timepoints where pooling of the 3 groups is not possible, the fixed effects will include study group, age category and visit.

#### Analysis by age-category

```
PROC MIXED DATA=SERO method=reml empirical;
CLASS subjid visit agecat;
MODEL post-vac=pre-vacc agecat visit visit* agecat /noint s cl;
RANDOM intercept/ subject=usubjid g v vcorr type = un;
REPEATED visit/type=un subject=subjid;
LSMEANS visit*agecat/ E cl;
ODS OUTPUT LSMEANS=LS;
RUN;
```

For the analysis by sex, sex and visit will be included as the fixed effects in the model. However, this is only applicable at timepoints where the 3 study groups will be pooled. Otherwise for the timepoints where pooling of the 3 groups is not possible, the fixed effects will include study group, sex and visit.

#### Analysis by sex

```
PROC MIXED DATA=SERO method=reml empirical;
CLASS subjid visit agecat;
MODEL post-vac=pre-vacc sex visit visit* sex / noint s cl;
RANDOM intercept/ subject=usubjid g v vcorr type = un;
REPEATED visit/type=un subject=subjid;
LSMEANS visit*sex/ E cl;
ODS OUTPUT LSMEANS=LS;
RUN;
```

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 2

For the analysis by region, region and visit will be included as the fixed effects in the model. However this is only applicable at timepoints where the 3 study groups will be pooled. Otherwise for the timepoints where pooling of the 3 groups is not possible, the fixed effects will include study group, region and visit.

#### Analysis by region

```
PROC MIXED DATA=SERO method=reml empirical;
CLASS subjid visitregion;
MODEL post-vac=pre-vacc region visit visit* region / noint scl;
RANDOM intercept/ subject=usubjid g v vcorr type = un;
REPEATED visit/type=un subject=subjid;
LSMEANS visit*region/ E cl;
ODS OUTPUT LSMEANS=LS;
RIIN:
```

The GMTs/GMCs, lower and upper confidence limits are obtained from the following data step:

```
DATA LS;
   SET LS;
   gm=10**estimate;
   ll=10**lower;
   ul=10**upper;
RUN;
```

The above SAS codes may be adapted in case of convergence issues.

#### 5.4.3.2. Cell-mediated immune response

#### Within groups evaluation

- The frequency of RSVPreF3 specific-CD4+ T cells will be displayed graphically using boxplots (min, Q1, median, Q3, max), by group and timepoint.
- The RSVPreF3-specific CD4+/ CD8+ T cell frequencies will be obtained by subtracting the background value to the antigen-induced value, and by setting to 1 all values less than or equal to zero for geomean calculation and graphical representation. Frequencies will be expressed as the number of cells per million of CD4+ T cells.
- More specifically, the frequencies of RSVPreF3-specific CD4+/ CD8+ T cells expressing at least 2 activation markers including at least one cytokine [Freq<sup>2+</sup>] will be computed as follows:

$$Freq_{Background}^{2+} = \frac{n_{background}^{2+}}{N_{Background}^{CD4}} \quad \text{and} \quad Freq_{Induction}^{2+} = \frac{n_{Induction}^{2+}}{N_{Induction}^{CD4}},$$

And

$$Freq_{Specific}^{2+} = Freq_{Induction}^{2+} - Freq_{Background}^{2+}$$

where

 $n_{Background}^{2+}$  = number of CD4+ T cells expressing at least 2 activation markers including at least one cytokine after stimulation with medium only (background),

 $n_{Induction}^{2+}$  = number of CD4+ T cells expressing at least 2 activation markers including at least one cytokine after stimulation with a pool of peptides covering RSVPreF3 (induction),

 $N_{\it Back/Ind}^{\it CD4}$  = Total number of CD4 T cells involved in the assay (background or induction).

For the computation of the fold increase (post- over pre-vaccination) of the frequency of RSVPreF3-specific CD4+ T-cells identified as expressing **at least 2 activation marker(s) including at least one cytokine** among CD40L, 4-1BB, IL-2, TNF-α, IFN-γ, IL-13, IL-17.the results **below the LLOQ** of the assay will be replaced by the value of the LLOQ.

# 5.4.3.3. Assessment of long-term persistence of the immune response at Months 18, 24 and 36 after dose 1

The exploratory analysis for modelling the long-term persistence of immune response (humoral and cellular) post dose 1 vaccination will constitute of the following;

- A piece-wise linear mixed model, power law model and modified power law model [David et al, 2009] for repeated measurements (all data available from Day 1, 31 and Month 6, 12, 18, 24, 30, 36 post-Dose 1 vaccination, will be used to model over time
  - the frequency of RSVPreF3-specific CD4+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 4-1BB, IL-2, TNF-α, IFN-γ, IL-13, IL-17.
  - the neutralizing antibody titers against RSV-A, RSV-B and RSVPreF3-specific IgG antibody concentrations.

The *piece-wise linear mixed model* is expressed as follows

The piece-wise model fits the data on three non-overlapping time intervals. This corresponds to the observed decay of humoral and cellular antibodies. Each piece of the model uses a linear function. Three break points, Months x, xx and xxx, will be selected on the basis of Akaike's Information Criterion (AIC) [Pan, 2001].

$$(ft) = \beta_0 + \beta_1 t \qquad \text{if } x \le t < xx \text{ months}$$

$$(ft) = \beta_0 + \beta_1 t + \beta_2 (t - xx) \quad \text{if } xx \le t < xxx \text{ months}.$$

$$(ft) = \beta_0 + \beta_1 t + \beta_2 (t - xx) + \beta_3 (t - xxx) \quad \text{if } t \ge xxx \text{ months}$$

where f(t) is the log-10 transformed antibody titer/concentration/ RSVPreF3-specific CD4+ T cells at time t post-vaccination,  $\beta_0$  is the intercept and  $\beta_1(i=1,2,3)$  are the parameters corresponding to the three time intervals, respectively. All three model effects

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 2

will be fitted using the SAS PROC MIXED standard code for linear regression methodology

```
ODS OUTPUT FitStatistics= stat;
ODS OUTPUT ConvergenceStatus= conv;
PROC MIXED DATA=kin&i.&j. EMPIRICAL COVTEST NOCLPRINT IC;
CLASS pid;
MODEL log_val = int_m int_m_pw_m&i.*m&i. int_m_pw_m&j.*m&j./s cl
covb outp=pred outpm=predm;
RANDOM intercept/SUBJECT=pid;
MAKE "solutionF" out=est;
RUN;
```

The *power-law model* is expressed as follows:

$$f(t) = k - a \log(c + t)$$

where f(t) is the log-10 transformed antibody titer/concentration/RSVPreF3-specific CD4+ T cells at time t post-vaccination, k is the peak log level, a is the decay rate, and c is an arbitrary small constant (set to zero in this case). The estimated maximum likelihood (ML) values for the model parameters will be obtained using the PROC NLMIXED SAS procedure.

```
PROC NLMIXED DATA=kineticm;

PARMS se=&se a0 =&a k0 =&k sk=&sk sa=&sa ska=&ska;

q = (1/&time) **a;

lg=&log(q);

mean = k + lg;

MODEL log_val ~ NORMAL(mean, se*se);

RANDOM k a ~ NORMAL([k0,a0], [sk*sk, ska, sa*sa]) SUBJECT=pid out=indiv;

RUN;
```

The *modified power-law model* is expressed as follows:

It is an extension of the power law model, and it is expressed as follows.

$$f(t) = k + \log[(1 - \pi)(c + t)^{a} + \pi]$$

The quantity  $\pi$  (between 0 and 1) represents the proportion of antibodies that are produced in the long term. When the value of  $\pi$  is positive, this implies long-term antibody persistence, as noted by [Fraser et al, 2007]. If  $\pi = 0$ , then the modified power-law model reduces to the standard power-law model. The estimated maximum likelihood (ML) values for the model parameters will be obtained using the PROC NLMIXED SAS procedure.

```
PROC NLMIXED DATA=kineticm; 

PARMS pi=&pi se=&se a0 =&a k0 =&k sk=&sk sa=&sa ska=&ska; 

q = (1-pi)*(1/\&time)**a; 

lg=\&log(q+pi); 

mean = k + lg; 

MODEL log_val ~ NORMAL(mean, se*se); 

RANDOM k a ~ NORMAL([k0,a0], [sk*sk, ska, sa*sa]) SUBJECT=pid out =indiv RUN;
```

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 2

- The three models based on data up to Month 36 will be presented graphically. Models based on data up to Month 18 vs. Month 24, Month 24 vs. Month 30 and Month 30 vs. Month 36 will be presented side by side.
- The above models and SAS codes may be adapted in case of convergence issues.

#### 5.4.3.4. Sensitivity analyses

- In case the COVID-19 pandemic is still ongoing during the study conduct, the following sensitivity analyses might be considered.
  - During the assessment of long-term persistence of the immune response, the models described in Section 5.4.3.3 might be fitted taking into account participants who received the first dose of study vaccine and with full follow-up (attending all study visits).
  - Similarly, a mixed model might be fitted for the evaluation of GMT/GMC based on participants with full follow-up (attending all study visits).

The goal of this sensitivity analysis is to determine the extent to which results might be impacted by considering the different scenarios.

#### 5.4.4. Safety analysis

## Primary vaccination and revaccination dose:

The safety analysis will be performed on the ES. A descriptive analysis by group, for the 3 groups pooled up to Month 12, for the RSV\_flexible revaccination and RSV\_1dose groups pooled vs RSV\_annual group for Month 13, Month 18 and Month 24, and by group from Month 25 up to study end, will present a summary of:

- The number and percentage of participants with at least one administration site event (solicited and unsolicited), with at least one systemic event (solicited and unsolicited) and with any AE during the 4-day or 30-day follow-up period will be tabulated with exact 95% CI after each dose. The same computations will be done for Grade 3 AEs, and for Grade 3 non-serious AEs and for AEs resulting in medically attended visit.
- The number and percentage of participants reporting each individual solicited administration site event (any grade, Grade 3 and resulting in medically attended visit) and solicited systemic event (any grade, Grade 3 and resulting in medically attended visit) during the 4-day follow-up period (i.e., on the day of vaccination and 3 subsequent days) will be tabulated for each group after each dose.
- For fever, the number and percentage of participants reporting fever by half degree (°C) cumulative increments during the 4-day follow-up period (i.e., on the day of vaccination and 3 subsequent days) will be tabulated for each group after each dose.
- The incidence of each solicited administration site event and solicited systemic event (any grade and grade 3) will be represented graphically after each dose.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 2

- The number and percentage of participants with any unsolicited AEs during the 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) with its exact 95% CI will be tabulated for each dose by group and by Medical Dictionary for Regulatory Activities (MedDRA) Primary System Organ Class (SOC), High Level Term (HLT) and preferred term (PT). Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs, for Grade 3 causally related unsolicited AEs and for unsolicited AEs resulting in a medically attended visit. The verbatim reports of unsolicited AEs will be reviewed by a qualified person and the signs and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. Every verbatim term will be matched with the appropriate Preferred Term.
- The number and percentage of participants with at least one report of SAE classified by the MedDRA Primary SOC, HLT and PTs and reported from Dose 1 up to 6 months post-Dose 1 and from revaccination dose up to 6 months post-revaccination will be tabulated with exact 95% CI. The same tabulation will be presented for causally related SAEs and fatal SAEs..
- The number and percentage of participants with at least one report of causally related SAEs classified by the MedDRA Primary SOC, HLT and PTs will be reported after each dose and from Day 1 up to study end with exact 95% CI. The same tabulation will be presented for fatal SAEs.
- All SAEs will also be described in detail in a tabular listing.
- All AEs/SAEs leading to study/intervention discontinuation from dose 1 up to study end will be tabulated.
- The number and percentage of participants with at least one report of pIMD classified by the MedDRA Primary SOC, HLT and PTs and reported from Dose 1 up to 6 months post-Dose 1 and from revaccination dose up to 6 months post-revaccination will be tabulated with exact 95% CI. The same tabulation will be presented for causally related pIMDs
- The number and percentage of participants with at least one causally related pIMD classified by the MedDRA Primary SOC, HLT and PTs will be reported after each dose and from Day 1 up to study end with exact 95% CI.
- All pIMDs will also be described in detail in a tabular listing.
- The analyses of unsolicited AEs will include SAEs (unless otherwise specified).

The analysis of safety will also be performed by age category (age at Dose  $1: \ge 65$  YOA,  $\ge 70$  YOA,  $\ge 80$  YOA, 60-69 YOA and 70-79 YOA) and region (North America, Europe, Asia).

#### 5.4.5. Additional considerations

- Compliance in completing solicited events information will be tabulated after each dose.
- The number and percentage of participants with at least one administration site event (solicited only), with at least one systemic event (solicited only) and with any solicited event during the 4-day follow-up period after each dose will be tabulated with exact 95% CI. The same computations will be done for Grade 3 AEs and for AEs resulting in a medically attended visit.
- The number of days with solicited events reported during the 4-day follow-up period will be tabulated for each solicited event, after each dose using descriptive statistics (mean, min, Q1, median, Q3, maximum).
- The number of each solicited events (any and Grade 3) that are ongoing beyond the 4-day follow-up period will be reported with the duration in days (mean, min, Q1, median, Q3, maximum).
- The list of solicited administration site and systemic events, and definition of intensity are described in Section 10.3.3 and 10.3.9.1 of the protocol.
- The number and percentage of participants with at least one report of SAE classified by the MedDRA Primary SOC, HLT and PTs and reported within 30 days following each vaccination will be tabulated with the exact 95% CI. The same tabulation will be presented for pIMDs.

The measurement of erythema/swelling (in mm) and fever (in °C/F) will be categorized as follows:

Table 7 Intensity grading scale for solicited events

| Grading | Erythema/swelling | Fever |
|---------|-------------------|---------------------------------------|
| 0: | ≤ 20 mm | < 38.0°C (100.4°F) |
| 1: | > 20 - ≤ 50 mm | ≥ 38.0°C(100.4°F) - ≤ 38.5°C(101.3°F) |
| 2: | > 50 - ≤ 100 mm | > 38.5°C(101.3°F) - ≤ 39.0°C(102.2°F) |
| 3: | > 100 mm | > 39.0°C(102.2°F) |

#### Combined Solicited events and Unsolicited AEs

For clinicaltrials.gov and EudraCT posting purposes, a summary of combined solicited and unsolicited non-serious adverse events will be produced by System Organ Class and preferred terms and according to occurrence of each event.

Solicited events will be coded by MedDRA as per the following codes:

| Solicited event | Lower level term code | Corresponding Lower |
|-----------------|-----------------------|-------------------------|
| | | level term decode |
| Pain | 10022086 | Injection site pain |
| Erythema | 10022061 | Injection site erythema |
| Swelling | 10053425 | Injection site swelling |
| Fever | 10016558 | Fever |
| Headache | 10019211 | Headache |
| Fatigue | 10016256 | Fatigue |
| Myalgia | 10028411 | Myalgia |
| Arthralgia | 10003239 | Arthralgia |

#### **Concomitant Medication** 5.4.5.1.

Medications will be coded using the GSKDRUG dictionary.

#### 5.4.6. **Sensitivity Analyses**

If more than 10% of participants miss the revaccination dose or don't have safety data reported after revaccination, the safety analysis described in section 5.4.4 will also be conducted on participants with full follow-up (attending all study visits).

The goal of this sensitivity analysis is to determine the extent to which results might be impacted by considering the different scenarios.

#### 6. ANALYSIS INTERPRETATION

All analyses are descriptive.

#### 7. INTERIM ANALYSES

#### 7.1. Sequence of analyses

Analyses to evaluate objectives and endpoints will be performed stepwise:

- Month 6: A first analysis will be performed on all reactogenicity, safety and immunogenicity data available and as clean as possible, when data for at least primary and secondary endpoints up to Month 6 are available for all participants. This analysis will be considered as final for those endpoints. \*
- Month 13: A second analysis will be performed on all reactogenicity, safety and immunogenicity data available and as clean as possible, when data for at least primary and secondary endpoints up to Month 12 are available for all participants, as well as data up to 1 month after the first revaccination (Month 13) in the RSV annual group. This analysis will be considered as final for those endpoints \*.
- Month 18: A third analysis will be performed on all safety and/or immunogenicity data available and as clean as possible, when data for secondary endpoints up to

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 2

Month 18 are available for all participants. This analysis will be considered as final for those endpoints \*. Safety and immunogenicity analysis may be performed at different time depending on data availability.

- Month 25: A fourth analysis will be performed on all safety, reactogenicity and immunogenicity data available and as clean as possible, when data for at least primary and secondary endpoints up to Month 24 are available for all participants, as well as data up to 1 month after the second revaccination (Month 25) in the RSV\_annual group and up to 1 month after the first revaccination (Month 25) in the RSV\_flexible revaccination group. This analysis will be considered as final for those endpoints \*.
- The final **End of Study** analysis will be performed when all reactogenicity, safety and immunogenicity data for at least primary and secondary endpoints up to study conclusion are available for all participants (Month 36).
- If the data for tertiary endpoints become available at a later stage, (an) additional analysis/analyses will be performed.
- \*Each analysis can be considered as final, as it is based on data that is as clean as possible. However, the consecutive analysis of the same time point might slightly differ at the next analysis e.g when M6 data are re-analyzed at the time of M13 analysis. If major changes are identified, they will be described in the clinical study report.

| Description | Analysis | Disclosure Purpose |
|---|---|---|
| | ID | (CTRS=public posting, SR=study report, internal) |
| End of study analysis | E1_01 | CTRS, SR |
| Analysis up to Month 6 | E1_02 | SR |
| Analysis up to Month 13 | E1_03 | CTRS, SR |
| Analysis up to Month 18 | E1_04 | Internal |
| Analysis up to Month 25 | E1 05 | Internal |

# 7.2. Statistical considerations for interim analyses

All analyses will be conducted on final data (as clean as possible) and therefore no statistical adjustment for interim analyses is required.

# 8. CHANGES TO THE PROTOCOL DEFINED STATISTICAL ANALYSIS

This statistical analysis plan complements the analyses described in the protocol.

The changes compared to the planned statistical analysis specified in the Protocol amendment 1 (Dated: 01 April 2022) are described below:

- The number and percentage of participants with at least one administration site event (solicited only), with at least one systemic event (solicited only) and with any solicited event during the 4-day follow-up period after vaccination
- Related SAEs/pIMDs and Fatal SAEs will be tabulated after each dose.
- SAEs/pIMDs within 30 days following each vaccination.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 2

# 9. NON-STANDARD DATA DERIVATION RULES AND STATISTICAL METHODS

The following sections describe additional derivation rules and statistical methods which are not presented in Section 10.1 (Business rules for standard data derivations and statistical methods).

# 9.1. Handling of missing data

#### 9.1.1. Dates

When partially completed dates (i.e. with missing day or month) are used in calculations, the following rules will be applied:

- AE start dates with missing day:
  - If the month is not the same as the vaccine dose, then the imputed start date will be the 1<sup>st</sup> of the month
  - If the event starts in the same month as the vaccine dose, the flag indicating if the event occurred before or after vaccination (AE.AESTRTPT) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the vaccine dose given during that month. If 'before vaccination' is selected, the imputed date will be one day before the vaccine dose given during that month.
- AE start dates with missing day and month:
  - If the year is not the same as the vaccine dose, then the imputed start date will be the 1<sup>st</sup> of January.
  - If the event starts in the same year as the vaccine dose, the flag indicating if the event occurred before or after vaccination (AE.AESTRTPT) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first vaccine dose given during that year. If 'before vaccination' is selected, the imputed date will be one day before the first vaccine dose given during that year.
- AE end dates with missing day: the imputed end date will be the last day of the month (30 or 31) or the study conclusion date whichever comes first.
- AE end dates with missing day and month: the imputed end date will be the last day of the year (31st of December) or the study conclusion date whichever comes first.

All incomplete concomitant medication/vaccination start/end date will follow the rules above.

#### 10. ANNEXES

# 10.1. Business rules for standard data derivations and statistical methods

This section contains standard rules for data display and derivation for clinical and epidemiological studies.

#### 10.1.1. Attributing events to vaccine doses

The dose relative to an event is the most recent study dose given to a participant prior to the start of a given event. For example, if the start date of an AE is between Dose 1 and Dose 2, the relative dose will be Dose 1.

If an event starts on the same day as a study dose, the relative dose will be derived from the additional information provided in the case report form (CRF) using the contents of the flag indicating if the event occurred before or after study dose. If 'after vaccination is selected, the relative dose for the event will be the one administered on the start day of the event. If 'before vaccination is selected, the relative dose for the event will be the dose prior to this one.

#### 10.1.2. Handling of missing data

#### 10.1.2.1. Dates

When partially completed dates (i.e. dates missing a day and/or month) are used in calculations, the following standard rules will be applied:

- A missing day will be replaced by 15<sup>th</sup>
- A missing day and month will be replaced by June 30<sup>th</sup>.

See also exceptions in Section 9.1.

#### 10.1.2.2. Laboratory data

Refer to Section 5.1.2 for more details.

#### 10.1.2.3. Daily recording of solicited events

#### 10.1.2.3.1. Studies with paper diaries

For studies using paper diaries which have questions in the CRF indicating the presence or absence of solicited events, the following rules are applicable:

• Denominators for the summary of administration site (or systemic) solicited events will be calculated using the number of participants who respond "Yes" or "No" to the question concerning the occurrence of administration site (or systemic) events.
212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 2

- When a specific solicited event is marked as having not occurred following a specific study dose (i.e. SDTM CE.CEOCCUR=N for the specified post-dose period for the event in question), all daily measurements will be imputed as Grade 0.
- When a specific solicited event is marked as having occurred following a specific study dose (i.e. SDTM CE.CEOCCUR=Y for the specified post-dose period for the event in question), any missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the solicited event summary tables.
- When the occurrence of a specific solicited event is not present (i.e. SDTM CE.CEOCCUR is neither Y nor N for the specified post-dose period for the event in question) but the group of solicited events (administration site or systemic) is marked as having occurred (i.e. SDTM CE.CEOCCUR=Y), all missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the solicited event summary tables.

The following table shows how participants contribute to each category for a specific solicited event over the Day X to Day Y post-dose period:

| Solicited event category | Participants included in the calculation of the numerator |
|---|---|
| Any | All participants with at least one occurrence of the adverse event at grade 1, grade 2, or grade 3 between Day X and Day Y or with the adverse event marked as present and at least one missing daily recording between Day X and Day Y |
| At least grade 1 | All participants with at least one occurrence of the adverse event at grade 1, grade 2, or grade 3 between Day X and Day Y |
| At least grade 2 | All participants with at least one occurrence of the adverse event at grade 2 or grade 3 between Day X and Day Y |
| At least grade 3 | All participants with at least one occurrence of the adverse event at grade 3 between Day X and Day Y |

#### 10.1.2.4. Unsolicited adverse events

Unsolicited AE summaries are including SAEs unless specified otherwise.

Missing severity, relationship with study vaccine, and outcome of unsolicited AEs will not be replaced and will appear as 'UNKNOWN' when displayed in a statistical output.

#### 10.1.3. Data derivation

#### 10.1.3.1. Age at first dose in years

When age at first dose is to be displayed in years, it will be calculated as the number of complete calendar years between the date of birth and the date of first dose. For example:

DOB = 
$$10$$
SEP1983, Date of first dose =  $09$ SEP2018 -> Age = 34 years

DOB = 
$$10$$
SEP1983, Date of first dose =  $10$ SEP2018 -> Age = 35 years

In this study, we will collect only the year of birth. The rules for handling missing day and/or month in the DOB are given in Section 10.1.2.1.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 2

Since only the year of birth will be collected in the eCRF, there might be some discrepancies between the age computed using standard derivation rules and the age category used in SBIR for the minimization.

Therefore, for the analysis by age, the age categories defined in Table 4 will be determined according to the information entered in SBIR (variable AGEGRP in SDTM SUPPDM), except for " $\geq$ 65 YOA" category which will be obtained using the derived age because this category is not used in SBIR for minimization

### 10.1.3.2. Temperature

Temperatures will be presented in degrees Celsius (°C). Temperatures reported in degrees Fahrenheit (°F) will be converted as follows:

Temperature (Celsius) =  $((Temperature (Fahrenheit) - 32) \times 5)/9$ 

### 10.1.3.3. Numerical serology results

Numerical serology results will be derived from the content of IS.ISORRES in the SDTM dataset. For humoral assays with a specific cut-off, the following derivation rules apply:

| IS.ISORRES | Derived value |
|-----------------------------------------------------|---------------|
| "NEG", "-", or "(-)" | cut-off/2 |
| "POS", "+", or "(+)" | cut-off |
| "< value" and value is <= assay cut-off | cut-off/2 |
| "< value" and value is > assay cut-off | Value |
| "> value" and value is < assay cut-off | cut-off/2 |
| "> value" and value is >= assay cut-off | Value |
| "value" and value is < cut-off | cut-off/2 |
| "value" and value is >= cut-off and value is <=ULOQ | value |
| "value" and value is > ULOQ | ULOQ* |
| All other cases | Missing |

<sup>\*</sup>This rule will be used to compute descriptive statistics (GMTs, fold increase etc).

### 10.1.3.4. Geometric mean titers (GMTs) and concentrations (GMCs)

GMT or GMC calculations are performed by taking the inverse logarithm of the mean of the log titer or concentration transformations. Non quantifiable antibody titers or concentrations will be converted as described in Section 10.1.3.3 for the purpose of GMT/GMC calculation. Cut-off values are defined by the laboratory before the analysis.

#### 10.1.3.5. Onset day

The onset day for an event (e.g. AE, concomitant medication/vaccination) is the number of days between the last study dose and the start date of the event. This is 1 for an event occurring on the same day as a study dose (and reported as starting after study dose).

#### 10.1.3.6. Duration of events

The duration of an event with a start and end date will be the difference between the start and end date plus one day, i.e. an event that starts on 3 March 2018 and ends on 12 March 2018 has a duration of 10 days.

The duration of solicited events will be calculated as the sum of the individual days with the event reported at grade 1 or higher or reported as missing ("NOT DONE"), during the solicited event period. The duration of solicited events ongoing beyond the solicited period will be calculated as end date – start date + 1. The goal of this change was to align this text with the standard programs.

### 10.1.3.7. Counting rules for combining solicited and unsolicited AEs

For output combining solicited and unsolicited AEs, all SAEs will be considered systemic events since the administration site flag is not included in the Expedited Adverse Event CRF pages. Unsolicited AEs with missing administration site flag will also be considered systemic.

Multiple events with the same PT which start on the same day are counted as only one occurrence.

In case a solicited event is worsening to Grade 3 after the solicited period, it should be reported only in the following table.

Summary of grade 3 AEs (solicited and unsolicited) within 30 days following each dose and overall

### 10.1.3.8. Counting rules for occurrences of solicited events

When the occurrences of solicited events are summarized, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurs. Also, in the case of co-administered study interventions, an administration site event recorded for a participant following multiple study interventions will be counted as only one occurrence.

### 10.1.4. Display of decimals

### 10.1.4.1. Percentages

Percentages and their corresponding confidence limits will be displayed with one decimal except for 100% in which case no decimal will be displayed.

### 10.1.4.2. Demographic/baseline characteristics statistics

The mean, median, and SD for continuous baseline characteristics will be presented with one decimal.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 2

The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values.

The maximum and minimum of transformed body temperatures will be displayed with one decimal.

### 10.1.4.3. Serological summary statistics

For each assay, GMT or GMC and their confidence limits will be presented with one decimal, as well as GMT/GMC fold increase from pre-dose.

The mean, median, SD and quartile values for frequency of RSVPreF3-specific-CD4+ and CD8+ T cells and for the fold increase (post- over pre-vaccination) will be presented with one decimal. The minimum and maximum values will be presented with no decimal.

### 10.1.5. Statistical methodology

### 10.1.5.1. Exact confidence intervals around proportions

The exact confidence intervals around within-group proportions are derived using the method of Clopper and Pearson [Clopper, 1934].

# 11. ADDITIONAL ANALYSES DUE TO THE COVID-19 PANDEMIC

Depending on how the COVID-19 situation evolves, the SAP might be amended to reflect the analysis corresponding to COVID-19.

### 12. REFERENCES

Clopper CJ, Pearson E. The Use of Confidence or Fiducial Limits Illustrated in the case of the Binomial. *Biometrika*. 1934;26:404-13.

David M-P, Van Herck K, Hardt K, Tibaldi F, Dubin G, Descamps D, et al. Long-term persistence of anti-HPV-16 and-18 antibodies induced by vaccination with the AS04-adjuvanted cervical cancer vaccine: modeling of sustained antibody responses. GYNECOLOGIC ONCOLOGY. 2009;115(3):S1–6.

Fraser C, Tomassini JE, Xi L, Golm G, Watson M, Giuliano AR, et al. Modeling the long-term antibody response of a human papillomavirus (HPV) virus-like particle (VLP) type 16 prophylactic vaccine. Vaccine 2007 May 22;25(21):4324-33

Pan W Akaike's information criterion in generalized estimating equations Biometrics, 57 (1) (2001), pp. 120-125

Rubin, D. B., Stern, H. S. AND Vehovar, V. Handling "don't know" survey responses: the case of the Slovenian plebiscite. Journal of the American Statistical Association 90, 1995, 822–828

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

| | Statistical Analysis Plan Amendment 1 |
|---|---|
| gsk | Statistical Analysis Plan |
| Title: | A phase 3, randomized, open-label, multi-country study to evaluate the immunogenicity, safety, reactogenicity and persistence of a single dose of the RSVPreF3 OA investigational vaccine and different revaccination schedules in adults aged 60 years and above. |
| eTrack study number and<br>Abbreviated Title | 212496 (RSV OA=ADJ-004) |
| Scope: | All data pertaining to the above study except the Safety Review Team analyses for the first 50 participants aged 80 years and above |
| Date of Statistical Analysis<br>Plan | Amendment 1 Final: 04 Mar 2022 |

APP 9000058193 Statistical Analysis Plan Template V5 (Effective date: 1July2020)

04 Mar 2022 Page 1 of 38

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

### **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| LIS | ST OF A | ABBREV | IATIONS | 6 |
| 1. | DOCU | JMENT H | HISTORY | 7 |
| 2. | OBJE | CTIVES | ENDPOINTS | 8 |
| 3. | STUD<br>3.1. | | GNdesign | |
| 4. | ANAL<br>4.1.<br>4.2. | Definition | frs | 12<br>12<br>12 |
| 5. | STAT<br>5.1. | | Immunogenicity | 17<br>17<br>17 |
| | 5.2. | Analysis 5.2.1. 5.2.2. | s of demography and baseline characteristics | 18<br>18 |
| | 5.3. | | endpoint(s) Analysis planned in the protocol 5.3.1.1. Humoral immune response – up to Month 12 | 19<br>19 |
| | 5.4. | Second 5.4.1. 5.4.2. 5.4.3. | ary endpoint(s) | 20<br>21<br>21<br>21 |
| | | 5.4.4.<br>5.4.5.<br>5.4.6. | after dose 1 | 26<br>26<br>27 |
| 6 | ΔΝΔΙ | YSIS IN | TERPRETATION | 28 |

| 7. | INTERIM ANA<br>7.1. Seque | LYSES | /ses | 29 |
|---|---|---|---|---|
| | 7.2. Statisti | cal conside | rations for interim analyses | 29 |
| 8. | CHANGES TO | O THE PRO | DTOCOL DEFINED STATISTICAL | |
| • | | | | 30 |
| | | | the SAP | |
| 9. | NON-STAND | ARD DATA | DERIVATION RULES AND STATISTICAL | |
| • | | | | 32 |
| | | | ng data | |
| | 9.1.1. | _ | <u> </u> | |
| 10. | ANNEXES | | | 33 |
| | | ss rules for | standard data derivations and statistical | |
| | method | ek | | 33 |
| | 10.1.1. | Attributing | g events to vaccine doses | 33 |
| | 10.1.2. | Handling | of missing data | 33 |
| | | 10.1.2.1. | Dates | 33 |
| | | 10.1.2.2. | Laboratory data | 33 |
| | | 10.1.2.3. | Daily recording of solicited events | 33 |
| | | | 10.1.2.3.1. Studies with paper diaries | 33 |
| | | 10.1.2.4. | Unsolicited adverse events | |
| | 10.1.3. | Data deri | vation | 35 |
| | | 10.1.3.1. | Age at first dose in years | 35 |
| | | | Temperature | |
| | | 10.1.3.3. | Numerical serology results | 35 |
| | | | Geometric mean titres (GMTs) and | |
| | | | concentrations (GMCs) | 36 |
| | | 10.1.3.5. | Onset day | 36 |
| | | 10.1.3.6. | Duration of events | 36 |
| | | | Counting rules for combining solicited and | |
| | | | unsolicited adverse events | 36 |
| | | 10.1.3.8. | Counting rules for occurrences of solicited | |
| | | | events | 36 |
| | 10.1.4. | Display of | f decimals | |
| | | | Percentages | |
| | | | Demographic/baseline characteristics | |
| | | | statistics | 37 |
| | | 10.1.4.3. | Serological summary statistics | |
| | 10.1.5. | | I methodology | |
| | | 10.1.5.1. | Exact confidence intervals around | |
| | | | proportions | 37 |
| 11. | ADDITIONAL | ANALYSE: | S DUE TO THE COVID-19 PANDEMIC | 37 |
| 12. | KEFEKENCE | .5 | | 38 |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

### **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | Study groups, intervention and blinding foreseen in the study | 10 |
| Table 2 | Group names and definition for footnote in the TFLs | 10 |
| Table 3 | Pooled group names and definition for footnote in the TFLs | 11 |
| Table 4 | Sub-group names and definitions for footnote in the TFLs | 11 |
| Table 5 | Populations for analyses | 12 |
| Table 6 | List of elimination codes | 13 |
| Table 7 | Intensity grading scale for solicited events | 28 |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

### **LIST OF FIGURES**

| | | PAGE |
|----------|-----------------------|------|
| Figure 1 | Study design overview | g |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

### LIST OF ABBREVIATIONS

**AE** Adverse event

**AESI** Adverse Events of Special Interest

**ANCOVA** Analysis of Covariance

**CD** Community Dwelling

CI Confidence Interval

**COVID-19** Coronavirus Disease 2019

**CRF** Case Report Form

CTRS Clinical Trial Registry Summary

Eli Type Internal database code for type of elimination code

**ELISA** Enzyme-linked immunosorbent assay

ELU/mL ELISA unit per milliliter

**ES** Exposed Set

**GMC** Geometric mean antibody concentration

**GMT** Geometric mean antibody titre

**GSK** GlaxoSmithKline

IU/mL International units per milliliter

LL Lower Limit of the confidence interval

LTCF Long Term Care Facility

**MedDRA** Medical Dictionary for Regulatory Activities

NA Not Applicable

**PD** Protocol Deviation

**PPS** Per-Protocol Set

**SAE** Serious adverse event

**SAP** Statistical Analysis Plan

SBIR GSK Biologicals Internet Randomization System

**SD** Standard Deviation

**SDTM** Study Data Tabulation Model

UL Upper Limit of the confidence interval

# 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|---|---|---|
| 15 February 2021<br>04 Mar 2022 | First version Amendment 1: The percentage has been changed to 5% in this statement: If in any study group the percentage of vaccinated participants with serological results excluded from the PPS for immunogenicity is at least 5%, a second analysis will be performed on the Exposed Set (section 4) The definition of randomized set and elimination code 1010 were deleted (section 4.2.1) Changes in the demography and baseline characteristics (section 5.2) Addition of demography analysis by sex and region Clarify that study intervention administered will also be tabulated by visit Deletion of participant disposition analysis in the ES and PPS by age category. Changes in the immunogenicity analysis section 5.4.1 and section 5.4.2 Deletion of some analyses Changes in the safety analysis (section 5.4.1 and section 5.4.2) Deletion of some analyses Unsolicited AEs, SAEs, pIMDs to also be presented by High Level Term (HLT) Solicited events (any and Grade 3) that are ongoing beyond the 4-day follow-up period to be considered Safety analysis to be presented also by region Additional details about persistence modelling have been added (section 5.4.3.3) | Final: 28 October 2020 Final: 28 October 2020 |

### 2. OBJECTIVES/ENDPOINTS

| Objectives | Endpoints |
|---|---|
| Prim | |
| To evaluate the humoral immune response following a 1-dose primary schedule of RSVPreF3 OA investigational vaccine up to 12 months post-Dose 1. | Humoral immune response at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), and at 6 and 12 months post-Dose 1 (Months 6 and 12), in a subset of participants: Neutralizing antibody titers against RSV-A Neutralizing antibody titers against RSV-B. |
| Secondary | |
| To further evaluate the humoral immune response following a 1-dose primary schedule of RSVPreF3 OA investigational vaccine up to 12 months post-Dose 1. | Humoral immune response at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), and at 6 and 12 months post-Dose 1 (Months 6 and 12), in a subset of participants: RSVPreF3-specific Immunoglobulin G (IgG) antibody concentrations. |
| To evaluate the humoral immune response following 1 dose of the RSVPreF3 OA investigational vaccine and following revaccination doses, up to study end. | Humoral immune response at Months 18, 24, 30 and 36 post-Dose 1, and at 1 month after each revaccination dose (Months 13 and 25), in a subset of participants: Neutralizing antibody titers against RSV-A and RSV-B RSVPreF3-specific IgG antibody concentrations. |
| To evaluate the cell-mediated immune (CMI) response following 1 dose of the RSVPreF3 OA investigational vaccine and following revaccination doses up to study end. | <ul> <li>CMI response at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), at Months 6, 12, 18, 24, 30 and 36 post-Dose 1, and at 1 month after each revaccination dose (Months 13 and 25), in a subset of participants:</li> <li>Frequency of RSVPreF3-specific CD4+ and/or CD8+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 4-1BB, IL-2, TNF-α, IFN-γ, IL-13, IL-17.</li> </ul> |
| To evaluate the safety and reactogenicity of each vaccination schedule of the RSVPreF3 OA investigational vaccine in all participants. | <ul> <li>Occurrence of each solicited administration-site and systemic event during a 4-day follow-up period (i.e., on the day of vaccination and 3 subsequent days) after each vaccination.</li> <li>Occurrence of any unsolicited AE during a 30-day follow up period (i.e., on the day of vaccination and 29 subsequent days) after each vaccination.</li> <li>Occurrence of all SAEs and pIMDs up to 6 months after each vaccination.</li> <li>Occurrence of fatal SAEs, related SAEs and related pIMDs from first vaccination (Day 1) up to study end (Month 36).</li> </ul> |
| Terti | ary |
| To further characterize immune responses to the RSVPreF3 OA investigational vaccine. | Any further exploratory immunology in a subset of participants, such as, but not limited to: Antibodies against specific protein F epitopes. Potential new immunological markers for protection. Frequency of RSVPreF3-specific CD4+ and/or CD8+ T cells expressing one or any combination of immune marker(s) **SAF = periods adverse event in IMD = petential immune mediated.** |

CMI = cell-mediated immunity, AE = adverse event, SAE = serious adverse event, pIMD = potential immune-mediated disease.

### STUDY DESIGN

### 3.1. Overall design

Figure 1 Study design overview



N = number of participants; D = Day; M = Month; AE = adverse event; HI = humoral immunity; CMI = cell-mediated immunity; pIMD = potential immune-mediated disease; SAE = serious adverse event.

- = blood sample for humoral immune responses (only applicable for the 345 participants of the RSV\_annual group; and for all participants of the RSV\_flexible revaccination and RSV\_1dose groups)
- = blood sample for CMI (only applicable for the ~345 participants of the RSV\_annual group, and ~115 participants each from the RSV\_flexible revaccination and RSV\_1dose groups).

Note: For group RSV\_annual, Revaccination Year 1 = Month 12; Revaccination Year 2 = Month 24.

- \* Visit and follow-up of solicited events, unsolicited AEs, SAEs and pIMDs only applicable for RSV\_annual group
- \*\* For the RSV\_annual group, the same ~345 participants will be part of both the HI and CMI subsets. The remaining ~645 participants will have no blood draws, and will only be followed up for safety and reactogenicity.
- \*\*\*For those participants in the RSV\_annual group without blood sample collections, visits at Months 6, 18, 30 and 36 may be through a phone contact. However, phone contact should be attempted only if site visit is not possible at Months 6, 18, 30 and 36.
- Type of study: self-contained.
- **Experimental design**: Phase 3, randomized, open-label, multi-country study with 3 parallel groups (see Figure 1).
- **Duration of the study**: ~ 36 months for each participant.
- **Primary completion date**: Month 12.
- Control: none.
- **Blinding**: open-label. Refer to the protocol for details.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

- **Data collection**: standardized electronic Case Report Form (eCRF). Solicited events and unsolicited AEs will be collected using a participant Diary card (paper Diary card).
- Safety monitoring: the study will be conducted with oversight by the project Safety Review Team (SRT). Please refer to protocol for the description of review of safety data by the SRT.
- **Study groups**: refer to Figure 1 and Table 1 for an overview of the study groups

Table 1 Study groups, intervention and blinding foreseen in the study

| | | | | Intervention | | |
|---|---|---|---|---|---|---|
| Study Groups | Number of participants | Age | Primary vaccination | Revaccination<br>Year 1 (Month<br>12) | Revaccination<br>Year 2 (Month<br>24) | Open |
| RSV_annual* | ~990 | ≥60 years | RSVPreF3 OA investigational vaccine | RSVPreF3 OA investigational vaccine | RSVPreF3 OA investigational vaccine | Х |
| RSV_flexible revaccination** | ~330 | ≥60 years | RSVPreF3 OA investigational vaccine | | | Х |
| RSV_1dose | ~330 | ≥60 years | RSVPreF3 OA investigational vaccine | (none) | (none) | Х |

<sup>\*</sup> RSV\_annual group will be split in 3 technical groups in SBIR in order to have a randomization ratio of 1:1:1:1:1: for treatment allocation and avoid predictability.

Groups and sub-groups definition for analysis: Refer to the tables below for a description of the groups and subgroups labels that will be used in the Tables Figures and Listings (TFLs).

For some of the analyses up to 12 months post dose 1, the 3 study groups will be pooled, and from Month 13, the RSV flexible revaccination and RSV 1dose groups will be pooled, at applicable timepoints. The following group names will be used in the TFLs:

Table 2 Group names and definition for footnote in the TFLs

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | RSV_annual | Participants receiving the first dose (Dose 1) of RSVPreF3 OA investigational vaccine at Day 1, followed by a revaccination dose at 12 months post-Dose 1 and at 24 months post-Dose 1 |
| 2 | RSV_flexible revaccination | Participants receiving the first dose (Dose 1) of RSVPreF3 OA investigational vaccine at Day 1 and a revaccination dose will be given whenever a revaccination would be needed |
| 3 | RSV_1dose | Participants receiving a single dose (Dose 1) of RSVPreF3 OA investigational vaccine at Day 1 |

<sup>\*\*</sup>Based on immunogenicity data from this study and efficacy results from the Phase 3 study RSV OA=ADJ-006, a revaccination might be decided for this group.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

Table 3 Pooled group names and definition for footnote in the TFLs

| Pooled Group label in tables | Groups to be pooled | Pooled definition for footnote | Comment |
|---|---|---|---|
| Total | RSV_annual,<br>RSV_flexible<br>revaccination and<br>RSV_1dose | Participants receiving one dose of RSVPreF3 OA investigational vaccine in all three groups | Applicable on data reported up to Month 12 |
| Flexible+1dose | RSV_flexible<br>revaccination, and<br>RSV_1dose | Participants receiving one dose of RSVPreF3 OA investigational vaccine in the RSV_flexible revaccination, and RSV_1dose groups | Applicable on data reported from Month 13 |

Table 4 Sub-group names and definitions for footnote in the TFLs

| Sub-analysis | Subgroup order in tables | Subgroup label in tables | Subgroup definition for footnote |
|---|---|---|---|
| By age | 1 | ≥65YOA | ≥65 years old participants |
| | 2 | ≥70YOA | ≥70 years old participants |
| | 3 | ≥80YOA | ≥80 years old participants |
| | 4 | 60-69YOA | 60-69 years old participants |
| | 5 | 70-79YOA | 70-79 years old participants |
| By sex | 1 | Female | Female |
| | 2 | Male | Male |
| By region | 1 | North America | Participants from North America (United States of America) |
| | 2 | Europe | Participants from Europe (Finland, Germany) |
| | 3 | Asia | Participants from Asia (Japan, Taiwan) |

YOA = Years of age

### Allocation of participants to assay subsets

Allocation of participants to assay subsets will be performed using SBIR. The subsets are detailed below.

| | RSV_annual | RSV_flexible revaccination | RSV_1dose |
|---|---|---|---|
| HI subset | ~345* | All participants (~330) | All participants (~330) |
| CMI subset | ~345* | ~115 | ~115 |

<sup>\*</sup>For the RSV\_annual group, the same ~345 participants will be part of both the HI and CMI subsets. The remaining ~645 participants will have no blood draws, and will only be followed up for safety and reactogenicity.

- HI subset: ~345 participants from the RSV annual group, and all participants from the RSV flexible revaccination and RSV 1dose groups. These participants will have blood samples collected for testing of humoral immunity at each visit applicable for their study group.
- CMI subset: ~345 participants from the RSV annual group, and ~115 participants each from the RSV flexible revaccination and RSV 1dose groups. These participants will have additional blood samples collected for CMI testing at each visit applicable for their study group.

### 4. ANALYSIS SETS

### 4.1. Definition

Table 5 Populations for analyses

| Analysis set | Description |
|---|---|
| Enrolled set | Participants who agreed to participate in a clinical study after completion of the |
| | informed consent process. |
| Exposed set (ES) | All participants who received at least 1 dose of the study intervention. The |
| | allocation in a group is done in function of the administered intervention. |
| Per Protocol set (PPS) | PPS) All participants who received at least 1 dose of the study intervention to which the |
| , , | are randomized and have post-vaccination data, minus participants with protocol |
| | deviations that lead to exclusion. |

The primary analysis for immunogenicity will be performed on the Per Protocol set (PPS). If in any study group the percentage of vaccinated participants with serological results excluded from the PPS for immunogenicity is at least 5%, a second analysis will be performed on the Exposed Set (ES). The immunogenicity analysis will be performed overall, by sex, by age category (age at Dose  $1: \ge 65 \text{ YOA}, \ge 70 \text{ YOA}, \ge 80 \text{ YOA}, 60-69 \text{ YOA}$  and 70-79 YOA, and by region (North America, Europe, Asia).

### 4.2. Criteria for eliminating data from Analysis Sets

### 4.2.1. Elimination from Exposed Set (ES)

Code 1030 (Study intervention not administered at all), 800 (Fraudulent data) and code 900 (invalid informed consent) will be used for identifying participants eliminated from the ES.

### 4.2.2. Elimination from Per-protocol analysis Set (PPS)

### 4.2.2.1. Excluded participants

A participant will be excluded from the populations of analysis under the following conditions

- For codes 800, 900, 1030 and 1050: participants will be eliminated for all visits
- For codes 1040, 1070, 1080, 1090, 2010, 2040, 2050, 2080: participants will be eliminated from a specific visit (at which the condition is met) onwards.
- For codes 2090, 2100, 2120, 2130: participants will be eliminated at the specific visit at which the condition is met.

# Table 6 List of elimination codes

| Code | Condition under which the code is used | Visit (timepoints) where the code is checked | Applicable for analysis set |
|---|---|---|---|
| 800 | Fraudulent data | All | ES and PPS |
| 900 | Invalid informed consent | All | ES and PPS |
| 1030 | Study intervention not administered at all | All | ES and PPS |
| 1040 | Administration of concomitant vaccine(s) forbidden in the protocol | All | PPS |
| | <ul> <li>Any investigational or non-registered vaccine other than the study vaccine used during the study period beginning 30 days before the first dose of study vaccine, or planned use during the study period.</li> <li>Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before each dose and ending 30 days after each dose of study vaccine administration, with the exception of inactivated, split virion and subunit influenza vaccines which can be administered up</li> </ul> | | |
| | <ul><li>to 14 days before or from 14 days after each study vaccination.</li><li>Previous vaccination with an</li></ul> | | |
| | RSV vaccine | | |
| 1050 | Randomization failure | Day 1 | PPS |
| 1070 | Vaccine administration not according to protocol Incomplete vaccination course | Vaccination visits at Day 1, Month 12, and 24 | PPS |
| | Participant was vaccinated with the correct vaccine but containing a lower volume | Months 12 and 24 are applicable to the RSV_annual group only | |

| Cada | Condition under which the code Visit (timepoints) Applicable for | | |
|---|---|---|---|
| Code | | Visit (timepoints) | Applicable for |
| | is used | where the code is | analysis set |
| | | checked | |
| | Participant was re-vaccinated while it was not planned | | |
| | Route of the study intervention is not intramuscular | | |
| | Wrong reconstitution of<br>administered vaccine | | |
| 1080 | Vaccine administration after a<br>Temperature deviation | Day 1, Month 12, and 24 | PPS |
| | Vaccine administered despite a Good Manufacturing Practices (GMP) no-go temperature deviation | Months 12 and 24 are applicable to the RSV_annual group only | |
| 1090 | Vaccine administration after expiration | Day 1, Month 12, and 24 | PPS |
| | | Months 12 and 24 are applicable to the RSV_annual group only | |
| 2010 | D . 11 11 1 | • | DDC. |
| 2010 | Protocol deviation linked to | All | PPS |
| | inclusion/exclusion criteria | | |
| 2040 | Administration of any medication forbidden by the protocol | All | PPS |
| | Any investigational or non-<br>registered medication used<br>during the study period | | |
| | • Administration of long-acting immune-modifying drugs at any time during the study period (e.g. <i>infliximab</i> ) | | |
| | Immunoglobulins and/or any<br>blood products administered<br>during the study period | | |
| | Chronic administration (defined as more than 14 consecutive days in total) of immunosuppressants or other immune-modifying drugs during the period starting 90 days prior to the study | | |

| α. | Statistical Analysis Plan Amendment | | |
|---|---|---|---|
| Code | Condition under which the code | Visit (timepoints) | Applicable for |
| | is used | where the code is | analysis set |
| | | checked | |
| | vaccine administration or | | |
| | planned administration during | | |
| | the study period. For | | |
| | corticosteroids, this will mean | | |
| | prednisone ≥20 mg/day, or | | |
| | equivalent. | | |
| 2050 | Intercurrent medical condition | All | PPS |
| | Participants may be eliminated from the PPS for immunogenicity if, during the study, they incur a condition that has the capability of | | |
| | altering their immune response (intercurrent medical condition) or are confirmed to have an alteration of their initial immune status. | | |
| 2000 | | 26 1 10 101 | 77.0 |
| 2080 | Participants did not comply with | Month 12 and 24 | PPS |
| | dosing schedule | | |
| | • RSV_annual: number of days between dose 1 and | | |
| | revaccination dose at Month<br>12 is outside [350-380 days] | | |
| | • RSV_annual: number of days between dose 1 and revaccination dose at Month 24 is outside [715-745 days] | | |
| 2090 | Participants did not comply with | Day 31, Month 6, 12, | PPS |
| | blood sample schedule | 13, 18, 24, 25, 30, 36 | |
| | Number of days between dose 1 and Day 31 blood sample is outside [30-42 days] | | |
| | Number of days between dose<br>1 and Month 6 blood sample is<br>outside [180-210 days] | | |
| | • Number of days between dose 1 and Month 12 blood sample is outside [350-380 days] | | |
| | Number of days between Month 12 and Month 18 blood | | |

| G : | Statistical Analysis Plan Amendment | | |
|---|---|---|---|
| Code | Condition under which the code | Visit (timepoints) | Applicable for |
| | is used | where the code is | analysis set |
| | | checked | |
| | sample is outside [180-210 days] | | |
| | Number of days between dose 1 and Month 24 blood sample is outside [715-745 days] | | |
| | Number of days between Month 24 and Month 30 blood sample is outside [180-210 days] | | |
| | Number of days between dose<br>1 and Month 36 blood sample<br>is outside [1080-1110 days] | | |
| | For RSV_annual group only: | | |
| | Number of days between<br>revaccination at Month 12 and<br>Month 13 blood sample is<br>outside [30-42 days] | | |
| | Number of days between<br>revaccination at Month 24 and<br>Month 25 blood sample is<br>outside [30-42 days] | | |
| 2600* | Participants not included in the humoral immunogenicity subset | Day 1, 31, Month 6, 12, 13, 18, 24, 25, 30, 36 | PPS |
| 2700* | Participants not included in the cell-mediated immune response subset | Day 1, 31, Month 6, 12, 13, 18, 24, 25, 30, 36 | PPS |
| 2100 | Serological results not available post-vaccination | Day 31, Month 6, 12, 13, 18, 24, 25, 30, 36 | PPS |
| | No immunological result at visit x for all the following tests: RSV A/B Neutralizing antibody titer, RSVPreF3-specific IgG antibody concentration and RSVPreF3-specific CD4+/CD8+ T cells frequency | Month 13 and 25 are applicable to the RSV_annual group only | |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

| Code | Condition under which the code is used | Visit (timepoints) where the code is checked | Applicable for analysis set |
|---|---|---|---|
| 2120 | Obvious incoherence or abnormality or error in laboratory data | Day 1, 31, Month 6, 12, 13, 18, 24, 25, 30, 36 | PPS |
| | Unreliable released data as a result of confirmed sample mismatch or confirmed inappropriate sample handling at laboratory | | |

<sup>\*</sup> codes 2600 and 2700 are not considered as protocol deviations, but those codes will be used to identify participants that are not part of the immunogenicity subsets.

### 5. STATISTICAL ANALYSES

Standard data derivation rules and stat methods are described in section 10.1 while the study specific data derivation rules and stat methods are described in section 9.

For the sake of analysis, data up to Month 12 will be analyzed by group (RSV\_annual, RSV\_flexible revaccination and RSV\_1dose), and also the 3 groups will be pooled. From Month 13, the analysis will be tabulated by group, and also for RSV\_annual versus the pooled RSV\_flexible revaccination and RSV\_1dose groups, at applicable time points.

If more than 5% of participants in the RSV\_annual group received only 1 dose or only 2 doses, an analysis by subgroup according to the number of dose(s) administered will be performed. The goal of this analysis is to describe the characteristics of participants in the RSV\_annual group who ultimately receive different numbers of revaccination doses in order to rule out the possibility of systematic differences between these subgroups.

### 5.1. General considerations

### 5.1.1. Demography

For a given participant and a given demographic variable, missing measurements will not be replaced.

### 5.1.2. Immunogenicity

- Any missing or non-evaluable immunogenicity measurement will not be replaced. The descriptive analysis performed for each assay at each time point will exclude participants with a missing or non-evaluable measurement. This is applicable to the standard way of computing GMTs/GMCs.
- During the computation of GMTs/GMCs from the mixed effects model (section 5.4.3.1). Multiple imputation (MI) technique will not be applied for any missing immunogenicity measurement. This is because the mixed effects model inherently

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

accounts for the missingness, under the assumption that the missing data are missing at random (MAR). Thus considering that missing data are MAR is a reasonable assumption for this descriptive clinical trial, then it is not necessary to perform MI [Rubin et al., 1995]

- The geometric mean titers/concentrations (GMTs/GMCs) will be computed by taking the anti-logarithm of the arithmetic mean of the log<sub>10</sub> transformed titers/concentrations.
- A seronegative participant will be defined as a participant whose antibody titer/concentration is below the cut-off value of the assay. A seropositive participant is a participant whose antibody titer/concentration is greater than or equal to the cut-off value of the assay.
- Antibody titers/concentrations below the assay cut-off will be given an arbitrary value of half the assay cut-off for the purpose of GMT/GMC calculation.
- Antibody titers/concentrations above the Upper Limit of Quantification (ULOQ) value will be given the ULOQ value for the purpose of GMT/GMC calculation.
- The mean geometric increase (MGI) is calculated by the geometric mean of ratios of antibody titers/concentrations of each post-primary vaccination time point over preprimary vaccination (Day 1).

### 5.1.3. Reactogenicity/Safety

- For a given participant and the analysis of solicited events within 4 days post-vaccination, missing or non-evaluable measurements will not be replaced. Therefore, the analysis of solicited events will include only vaccinated participants with documented solicited safety data (i.e., paper diary completed).
- For analysis of unsolicited AEs, SAEs, pIMDs and concomitant medications, all vaccinated participants will be considered. Participants who did not report an event or concomitant medication will be considered as participants without the event or the concomitant medication, respectively.

# 5.2. Analysis of demography and baseline characteristics

### 5.2.1. Analysis planned in the protocol

Descriptive summaries will be performed for each group (RSV\_annual, RSV\_flexible revaccination and RSV\_ldose) and overall. The same will be performed in each subset (humoral immune subset and CMI subset).

Demographic/baseline characteristics (age at vaccination in years, sex, race, ethnicity, type of residence (CD/LTCF) and smoking status) will be summarized using descriptive statistics:

- Frequency tables will be generated for categorical variables such as race.
- Mean, median, standard deviation and range will be provided for continuous data such as age.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

The distribution of participants will be tabulated as a whole and per group, for each age category, and for each subset.

The number of doses of the study intervention administered will be tabulated by group and by visit.

Withdrawal status will be summarized by group using descriptive statistics:

- The number of participants enrolled into the study as well as the number of participants excluded from Per Protocol (PP) analyses will be tabulated.
- The numbers of participants withdrawn from the study will be tabulated according to the reason for withdrawal.

Participant disposition in the ES and PPS will be reported as a whole and per group

The number and percentage of participants using concomitant medication (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) during the 4-day follow-up period (i.e., on the day of vaccination and 3 subsequent days) and during the 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) will be summarized by group after each vaccine dose and overall, and after the revaccination.

### 5.2.2. Additional considerations

- The analysis of demographic characteristics by group will be performed on the ES and on the PPS.
- Demography and baseline characteristics will also be summarized by sex and region

### 5.3. Primary endpoint(s)

### 5.3.1. Analysis planned in the protocol

The primary analysis for immunogenicity will be performed on the Per Protocol set (PPS). If in any study group the percentage of vaccinated participants with serological results excluded from the PPS for immunogenicity is at least 5%, a second analysis will be performed on the Exposed Set (ES).

### 5.3.1.1. Humoral immune response – up to Month 12

The analysis of the primary vaccination time points up to Month 12 will be performed for each group and for the 3 groups pooled. For each time point with blood sample collection for humoral immune response up to Month 12 and for each assay (RSV-A/-B neutralization assays), unless otherwise specified, the following analyses will be performed:

### Within groups evaluation:

- Percentage of participants with antibody titers/concentrations above a positivity cutoff and their exact 95% confidence interval (CI) will be tabulated.
- GMTs/GMCs and their 95% CI will be tabulated and represented graphically. Furthermore, to account for all the time points at which the blood samples are collected, a mixed effects model (see section 5.4.3.1) will be fitted, from which the GMTs/GMCs will be computed.
- Antibody titers/concentrations will be displayed using reverse cumulative curves.
- The MGI i.e. geometric mean of ratios of antibody titer/concentrations will be tabulated with 95% CI.

### 5.4. Secondary endpoint(s)

### 5.4.1. Humoral immune response

The same analyses as described above for the primary endpoint will be performed for PreF3 IgG ELISA up to Month 12 and for each time point with blood sample collection for humoral immune response **from study Month 13 up to study end** and for each assay (preF3 IgG **ELISA and RSV-A/-B neutralization assays**). The analysis of the post-primary vaccination time points from study Month 13 up to study end will be performed for each group and for the pooled RSV\_flexible revaccination and RSV\_ldose groups.

Only the analyses requiring further clarification of the exact time points analysed are summarized below:

### Within groups evaluation:

- The MGI i.e. geometric mean of ratios of antibody titer/concentrations will be tabulated with 95% CI:
  - For each post-primary vaccination time point (at Months 18, 24, 30 and 36 when applicable) over pre-primary vaccination (Day 1),
  - For each post-revaccination time point over corresponding pre-revaccination (Months 12/24) in the RSV annual group,
  - For 1 month post-revaccination at Month 12 (Month 13) over 1 month post-Dose 1 vaccination (Day 31) in RSV\_annual group.
  - For 1 month post-revaccination at Month 24 (Month 25) over 1 month post-revaccination at Month 12 (Month 13) in RSV annual group

In addition, the following evaluation will be performed:

• The kinetics of GMTs/GMCs will be plotted as a function of time for participants with results available at all post-primary vaccination time points.

The immunogenicity analysis will be performed overall, by sex, age category (age at Dose  $1: \ge 65 \text{ YOA}, \ge 70 \text{ YOA}, \ge 80 \text{ YOA}, 60-69 \text{ YOA}$  and 70-79 YOA), and region (North America, Europe, Asia).

### 5.4.2. Cell-mediated immune response

### Within groups evaluation:

The following parameters will be summarized by group at each time point for which blood samples are collected, for the 3 groups pooled for time points up to study Month 12, for the pooled RSV\_flexible revaccination and RSV\_1 dose up to study end using descriptive statistics (N, geometric mean, min, Q1, median, Q3, max) in the CMI subset:

- Frequency of RSVPreF3-specific CD4+ and/or CD8+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13, IL-17, measured by intracellular cytokine staining (ICS) using peripheral blood mononuclear cells PBMCs.
- The kinetics of RSVPreF3-specific CD4+ T cells frequencies will be plotted as a function of time for participants with results available at all primary vaccination time points.
- Fold increase of the frequency of RSVPreF3-specific CD4+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13, IL-17, measured by ICS at each post-primary vaccination time point over pre-vaccination (Day 1) by group, at each post-revaccination over the corresponding pre-revaccination and at one month post-revaccination over 1 month post-previous dose in the RSV annual group.

The immunogenicity analysis will be performed overall, by sex, age category (age at Dose  $1: \ge 65 \text{ YOA}, \ge 70 \text{ YOA}, \ge 80 \text{ YOA}, 60-69 \text{ YOA}$  and 70-79 YOA, and region (North America, Europe, Asia).

### 5.4.3. Additional considerations

#### 5.4.3.1. Mixed effects model

For the GMTs/GMCs calculation based on the mixed effects model mentioned in section 5.3.1.1, repeated measures analysis of covariance (ANCOVA) model will be fitted including age category (60-69 YOA, 70-79 YOA and ≥80 YOA,), study group (RSV\_annual, RSV\_flexible revaccination and RSV\_1dose), sex (male and female), visit (Day 31, Month 6, 12, 13, 18, 24, 25, 30, 36), as fixed effects, pre-vaccination log10-transformed titers/concentrations as a covariate and the response variable is the post-vaccination log10-transformed titers/concentrations. The PROC MIXED procedure in SAS® will be used to carry out the ANCOVA.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

The following SAS codes will be used:

For the analysis by study group, study group and visit will be included as the fixed effects in the model

```
Analysis by group
PROC MIXED DATA=SERO method=reml empirical;
CLASS subjid group visit;
MODEL post-vac=pre-vacc group visit visit*group/ noint s cl;
RANDOM intercept/ subject=usubjid g v vcorr type = un;
REPEATED visit/type=unsubject=subjid;
LSMEANS visit*group/ E cl;
ODS OUTPUT LSMEANS=LS;
RUN;
```

For the analysis by age category, age category and visit will be included as the fixed effects in the model. However, this is only applicable at timepoints where the 3 study groups will be pooled. Otherwise for the timepoints where pooling of the 3 groups is not possible, the fixed effects will include study group, age category and visit.

### Analysis by age-category

```
PROC MIXED DATA=SERO method=reml empirical;
CLASS subjid visit agecat;
MODEL post-vac=pre-vacc agecat visit visit* agecat /noint s cl;
RANDOM intercept/ subject=usubjid g v vcorr type = un;
REPEATED visit/type=un subject=subjid;
LSMEANS visit*agecat/ E cl;
ODS OUTPUT LSMEANS=LS;
RUN;
```

For the analysis by sex, sex and visit will be included as the fixed effects in the model. However, this is only applicable at timepoints where the 3 study groups will be pooled. Otherwise for the timepoints where pooling of the 3 groups is not possible, the fixed effects will include study group, sex and visit.

#### Analysis by sex

```
PROC MIXED DATA=SERO method=reml empirical;
CLASS subjid visit agecat;
MODEL post-vac=pre-vacc sex visit visit* sex / noint s cl;
RANDOM intercept/ subject=usubjid g v vcorr type = un;
REPEATED visit/type=un subject=subjid;
LSMEANS visit*sex/ E cl;
ODS OUTPUT LSMEANS=LS;
RUN;
```

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

For the analysis by region, region and visit will be included as the fixed effects in the model. However this is only applicable at timepoints where the 3 study groups will be pooled. Otherwise for the timepoints where pooling of the 3 groups is not possible, the fixed effects will include study group, region and visit.

### Analysis by region

```
PROC MIXED DATA=SERO method=reml empirical;
CLASS subjid visitregion;
MODEL post-vac=pre-vacc region visit visit* region / noint scl;
RANDOM intercept/ subject=usubjid g v vcorr type = un;
REPEATED visit/type=un subject=subjid;
LSMEANS visit*region/ E cl;
ODS OUTPUT LSMEANS=LS;
RIIN:
```

The Geometric mean antibody titers/concentrations, lower and upper confidence limits are obtained from the following data step:

```
DATA LS;
   SET LS;
   gm=10**estimate;
   ll=10**lower;
   ul=10**upper;
RUN;
```

The above SAS codes may be adapted in case of convergence issues.

### 5.4.3.2. Cell-mediated immune response

### Within groups evaluation

- The frequency of RSVPreF3 specific-CD4+ T cells will be displayed graphically using boxplots (min, Q1, median, Q3, max), by group and timepoint.
- The RSVPreF3-specific CD4+/ CD8+ T cell frequencies will be obtained by subtracting the background value to the antigen-induced value, and by setting to 1 all values less than or equal to zero for geomean calculation and graphical representation. Frequencies will be expressed as the number of cells per million of CD4+ T cells.
- More specifically, the frequencies of RSVPreF3-specific CD4+/ CD8+ T cells expressing at least 2 activation markers including at least one cytokine [Freq<sup>2+</sup>] will be computed as follows:

$$Freq_{Background}^{2+} = \frac{n_{background}^{2+}}{N_{Background}^{CD4}}$$
 and  $Freq_{Induction}^{2+} = \frac{n_{Induction}^{2+}}{N_{Induction}^{CD4}}$ ,

And

$$Freq_{Specific}^{2+} = Freq_{Induction}^{2+} - Freq_{Background}^{2+}$$

where

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

 $n_{Background}^{2+}$  = number of CD4+ T cells expressing at least 2 activation markers including at least one cytokine after stimulation with medium only (background)

 $n_{Induction}^{2+}$  = number of CD4+ T cells expressing at least 2 activation markers including at least one cytokine after stimulation with a pool of peptides covering RSVPreF3 (induction)

 $N_{\it Back/Ind}^{\it CD4}$  = Total number of CD4 T cells involved in the assay (background or induction)

For the computation of the fold increase (post over pre-vaccination) of the frequency of RSVPreF3-specific CD4+ T-cells identified as expressing **at least 2 marker(s)** among IL-2, CD40L, TNF- $\alpha$ , IFN- $\gamma$ , the results **below the LLOQ** of the assay will be replaced by the value of the LLOQ.

# 5.4.3.3. Assessment of long-term persistence of the immune response at Months 18, 24 and 36 after dose 1.

The exploratory analysis for modelling the long-term persistence of immune response (humoral and cellular) post dose 1 vaccination will constitute of the following;

- A piece-wise linear mixed model, power law model and modified power law model [David et al, 2009] for repeated measurements (all data available from Day 1, 31 and Month 6, 12, 18, 24, 30, 36 post dose 1 vaccination, will be used to model over time
  - the frequency of RSVPreF3-specific CD4+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 4-1BB, IL-2, TNF-α, IFN-γ, IL-13, IL-17.
  - the neutralizing antibody titers against RSV-A, RSV-B and RSVPreF3-specific IgG antibody concentrations.

### The *piece-wise linear mixed model* is expressed as follows

The piece-wise model fits the data on three non-overlapping time intervals. This corresponds to the observed decay of humoral and cellular antibodies. Each piece of the model uses a linear function. Three break points, Months x, xx and xxx, will be selected on the basis of Akaike's Information Criterion (AIC) [Pan, 2001].

$$(ft) = \beta_0 + \beta_1 t \qquad \text{if } x \le t < xx \text{ months}$$

$$(ft) = \beta_0 + \beta_1 t + \beta_2 (t - xx) \quad \text{if } xx \le t < xxx \text{ months}.$$

$$(ft) = \beta_0 + \beta_1 t + \beta_2 (t - xx) + \beta_3 (t - xxx) \quad \text{if } t \ge xxx \text{ months}$$

where f(t) is the log antibody titer/concentration/RSVPreF3-specific CD4+ T cells at time t post-vaccination,  $\beta_0$  is the intercept and  $\beta_1(i=1,2,3)$  are the parameters corresponding to the three time intervals, respectively. All three model effects will be fitted using the SAS PROC MIXED standard code for linear regression methodology

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

```
ODS OUTPUT FitStatistics= stat;
ODS OUTPUT ConvergenceStatus= conv;
PROC MIXED DATA=kin&i.&j. EMPIRICAL COVTEST NOCLPRINT IC;
CLASS pid;
MODEL log_val = int_m int_m_pw_m&i.*m&i. int_m_pw_m&j.*m&j./s cl
covb outp=pred outpm=predm;
RANDOM intercept/SUBJECT=pid;
MAKE "solutionF" out=est;
RUN;
```

The *power-law model* is expressed as follows:

$$f(t) = k - a \log(c + t)$$

where f(t) is the log antibody titer/concentration/RSVPreF3-specific CD4+ T cells at time t post-vaccination, k is the peak log level, a is the decay rate, and c is an arbitrary small constant (set to zero in this case). The estimated maximum likelihood (ML) values for the model parameters will be obtained using the PROC NLMIXED SAS procedure.

```
PROC NLMIXED DATA=kineticm;

PARMS se=&se a0 =&a k0 =&k sk=&sk sa=&sa ska=&ska;

q = (1/&time) **a;

lg=&log(q);

mean = k + lg;

MODEL log_val ~ NORMAL(mean, se*se);

RANDOM k a ~ NORMAL([k0,a0], [sk*sk, ska, sa*sa]) SUBJECT=pid out=indiv;

RIN:
```

The *modified power-law model* is expressed as follows:

It is an extension of the power law model, and it is expressed as follows.

$$f(t) = k + \log[(1 - \pi)(c + t)^{a} + \pi]$$

The quantity  $\pi$  (between 0 and 1) represents the proportion of antibodies that are produced in the long term. When the value of  $\pi$  is positive, this implies long-term antibody persistence, as noted by [Fraser et al, 2007]. If  $\pi = 0$ , then the modified power-law model reduces to the standard power-law model. The estimated maximum likelihood (ML) values for the model parameters will be obtained using the PROC NLMIXED SAS procedure.

```
PROC NLMIXED DATA=kineticm;

PARMS pi=&pi se=&se a0 =&a k0 =&k sk=&sk sa=&sa ska=&ska;

q = (1-pi)*(1/&time)**a;

lg=&log(q+pi);

mean = k + lg;

MODEL log_val ~ NORMAL(mean, se*se);

RANDOM k a ~ NORMAL([k0,a0], [sk*sk, ska, sa*sa]) SUBJECT=pid out =indiv

RIN:
```

- The three models based on data up to M36 will be presented graphically. Models based on data up to M18 vs M24, M24 vs M30 and M30 vs M36 will be presented side by side.
- The above models and SAS codes may be adapted in case of convergence issues.

### 5.4.3.4. Sensitivity analyses

- In case the COVID-19 pandemic is still ongoing during the study conduct, the following sensitivity analyses might be considered.
  - During the assessment of long-term persistence of the immune response, the models described in section 5.4.3.3 might be fitted taking into account;
     Participants who received the first dose of study vaccine and with full follow-up (attending all study visits)
  - Similarly, a mixed model will be fitted for the evaluation of GMT/GMC based on participants with full follow-up (attending all study visits).

The goal of this sensitivity analysis is to determine the extent to which results might be impacted by considering the different scenarios.

### 5.4.4. Safety analysis

### Primary vaccination and revaccination dose:

The safety analysis will be performed on the ES. A descriptive analysis by group, for the 3 groups pooled up to Month 12, for the RSV\_flexible revaccination and RSV\_1dose groups pooled vs RSV\_annual group from study Month 13 up to study end will present a summary of:

- The number and percentage of participants with at least one administration site event (solicited and unsolicited), with at least one systemic event (solicited and unsolicited) and with any AE during the 4-day or 30-day follow-up period will be tabulated with exact 95% CI after each dose. The same computations will be done for Grade 3 AEs, and for Grade 3 non-serious AEs and for AEs resulting in medically attended visit.
- The number and percentage of participants reporting each individual solicited administration site event (any grade, Grade 3 and resulting in medically attended visit) and solicited systemic event (any grade, Grade 3 and resulting in medically attended visit) during the 4-day follow-up period (i.e., on the day of vaccination and 3 subsequent days) will be tabulated for each group after each dose.
- For fever, the number and percentage of participants reporting fever by half degree (°C) cumulative increments during the 4-day follow-up period (i.e., on the day of vaccination and 3 subsequent days) will be tabulated for each group after each dose.
- The incidence of each solicited administration site event and solicited systemic event (any grade and grade 3) will be represented graphically after each dose.
- The number and percentage of participants with any unsolicited AEs during the 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) with its exact 95% CI will be tabulated for each dose by group and by Medical Dictionary for Regulatory Activities (MedDRA) Primary System Organ Class (SOC), *High Level Term (HLT) and* preferred term (PT). Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs, for Grade 3 causally related unsolicited AEs and for unsolicited AEs resulting in a medically attended

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

visit. The verbatim reports of unsolicited AEs will be reviewed by a qualified person and the signs and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. Every verbatim term will be matched with the appropriate Preferred Term.

- The number and percentage of participants with at least one report of SAE classified by the MedDRA Primary SOC, HLT and PTs and reported from Dose 1 up to 6 months post-Dose 1 and from revaccination dose up to 6 months post-revaccination will be tabulated with exact 95% CI.
- The number and percentage of participants with at least one report of causally related SAE classified by the MedDRA Primary SOC, HLT and PTs and reported during the entire study period will be tabulated with exact 95% CI.
- The same tabulation will be presented for fatal SAEs.
- All SAEs will also be described in detail in a tabular listing.
- All AEs/SAEs leading to study/intervention discontinuation from dose 1 up to study end will be tabulated.
- The number and percentage of participants with at least one report of pIMD classified by the MedDRA Primary SOC, HLT and PTs and reported from Dose 1 up to 6 months post-Dose 1 and from revaccination dose up to 6 months post-revaccination will be tabulated with exact 95% CI.
- The number and percentage of participants with at least one causally related pIMD classified by the MedDRA Primary SOC, HLT and PTs and reported during the entire study period will be tabulated with exact 95% CI.
- All pIMDs will also be described in detail in a tabular listing.
- The analyses of unsolicited AEs will include SAEs (unless otherwise specified).

The analysis of safety will also be performed by age category (age at Dose  $1: \ge 65$  YOA,  $\ge 70$  YOA,  $\ge 80$  YOA, 60-69 YOA and 70-79 YOA) and region (North America, Europe, Asia).

### 5.4.5. Additional considerations

- Compliance in completing solicited events information will be tabulated after each dose and overall.
- The number of days with solicited events reported during the 4-day follow-up period will be tabulated for each solicited event, after each dose using descriptive statistics (mean, min, Q1, median, Q3, maximum).
- The number of each solicited events (any and Grade 3) that are ongoing beyond the 4-day follow-up period will be reported with the duration in days (mean, min, Q1, median, Q3, maximum).
- The list of solicited administration site and systemic events, and definition of intensity are described in Section 10.3.3 and 10.3.9.1 of the protocol.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

The measurement of erythema/swelling (in mm) and fever (in °C/F) will be categorized as follows:

Table 7 Intensity grading scale for solicited events

| Grading | Erythema/swelling | Fever |
|---------|-------------------|---------------------------------------|
| 0: | ≤ 20 mm | < 38.0°C (100.4°F) |
| 1: | > 20 - ≤ 50 mm | ≥ 38.0°C(100.4°F) - ≤ 38.5°C(101.3°F) |
| 2: | > 50 - ≤ 100 mm | > 38.5°C(101.3°F) - ≤ 39.0°C(102.2°F) |
| 3: | > 100 mm | > 39.0°C(102.2°F) |

### **Combined Solicited events and Unsolicited AEs**

For clinicaltrials.gov and EudraCT posting purposes, a summary of combined solicited and unsolicited non-serious adverse events will be produced by System Organ Class and preferred terms and according to occurrence of each event.

Solicited events will be coded by MedDRA as per the following codes:

| Solicited event | Lower level term code | <b>Corresponding Lower</b> |
|-----------------|-----------------------|----------------------------|
| | | level term decode |
| Pain | 10022086 | Injection site pain |
| Erythema | 10022061 | Injection site erythema |
| Swelling | 10053425 | Injection site swelling |
| Fever | 10016558 | Fever |
| Headache | 10019211 | Headache |
| Fatigue | 10016256 | Fatigue |
| Myalgia | 10028411 | Myalgia |
| Arthralgia | 10003239 | Arthralgia |

#### 5.4.5.1. **Concomitant Medication**

Medications will be coded using the GSKDRUG dictionary.

#### 5.4.6. **Sensitivity Analyses**

If more than 10% of participants miss the revaccination dose or don't have safety data reported after revaccination, the safety analysis described in section 5.4.4 will also be conducted on participants with full follow-up (attending all study visits).

The goal of this sensitivity analysis is to determine the extent to which results might be impacted by considering the different scenarios.

#### ANALYSIS INTERPRETATION 6.

All analyses are descriptive.

### 7. INTERIM ANALYSES

### 7.1. Sequence of analyses

Analyses to evaluate objectives and endpoints will be performed stepwise:

- **Month 6:** A first analysis\* will be performed on all reactogenicity, safety and immunogenicity data available and as clean as possible, when data for at least primary and secondary endpoints up to Month 6 are available for all participants. This analysis will be considered as final for those endpoints.
  - \*Note: the analysis at Month 6 may be merged with the analysis at the subsequent timepoint.
- Month 13: A second analysis will be performed on all reactogenicity, safety and immunogenicity data available and as clean as possible, when data for at least primary and secondary endpoints up to Month 12 are available for all participants, as well as data up to 1 month after the first revaccination (Month 13) in the RSV\_annual group. This analysis will be considered as final for those endpoints.
- Month 18: A third analysis will be performed on all safety and/or immunogenicity data available and as clean as possible, when data for secondary endpoints up to Month 18 are available for all participants. This analysis will be considered as final for those endpoints. Safety and immunogenicity analysis may be performed at different time depending on data availability.
- Month 25: A fourth analysis will be performed on all reactogenicity, safety and immunogenicity data available and as clean as possible, when data for at least primary and secondary endpoints up to Month 24 are available for all participants, as well as data up to 1 month after the second revaccination (Month 25) in the RSV annual group. This analysis will be considered as final for those endpoints.
- The final **End of Study** analysis will be performed when all reactogenicity, safety and immunogenicity data for at least primary and secondary endpoints up to study conclusion are available for all participants (Month 36).
- If the data for tertiary endpoints become available at a later stage, (an) additional analysis/analyses will be performed.

| Description | Analysis | Disclosure Purpose |
|---|---|---|
| | ID | (CTRS=public posting, SR=study report, internal) |
| End of study analysis | E1_01 | CTRS, SR |
| Analysis up to Month 6 | E1_02 | SR |
| Analysis up to Month 13 | E1_03 | CTRS, SR |
| Analysis up to Month 18 | E1_04 | Internal |
| Analysis up to Month 25 | E1_05 | Internal |

# 7.2. Statistical considerations for interim analyses

All analyses will be conducted on final data (as clean as possible) and therefore no statistical adjustment for interim analyses is required.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

# 8. CHANGES TO THE PROTOCOL DEFINED STATISTICAL ANALYSIS

This statistical analysis plan complements the analyses described in the protocol.

Analysis sets: The percentage has been changed from 10% to 5%, the rationale for changing is to align with other phase 3 RSV OA studies (see section 4).

Randomized set: This cohort has been deleted from the SAP, simply because it is not needed when there is no screening visit and elimination code 1010 has been deleted as well (see section 4.2.1).

### Statistical analyses

The following changes have been made for the demography analyses

**Demography** (see section 5.2.1 and section 5.2.2)

Participant disposition in the ES and PPS will not be conducted by age category. The analysis by age category was considered not relevant for a phase 3 study.

Demography and baseline characteristics will also be summarized by age category, region and sex. Since the immunogenicity analyses will be conducted by these variables, it was considered relevant by the study team that the demography analyses should also be summarized by these variables.

The number of doses of the study intervention administered will be tabulated by group and by visit. This analysis will also be done by visit, since we have different vaccination schedules for the 3 study groups.

Regarding immunogenicity(see section 5.4.1 and section 5.4.2) and safety (see section 5.4.4), the following analyses are not considered relevant for a phase 3 study hence have been deleted. In addition, we aim at reducing the number of tables produced thus limiting analyses to only important tables.

**Immunogenicity** (see section 5.4.1 and section 5.4.2)

### Humoral Immunogenicity

Individual post-primary vaccination results (at Months 18, 24, 30 and 36 when applicable) versus pre-vaccination results (Day 1) by group and individual post-revaccination results versus the corresponding pre-revaccination results (Months 12/24) in the RSV annual group will be provided using scatter plots.

Distribution of the fold increase of the antibody titers/concentrations (post- over preprimary vaccination dose, post- over the corresponding pre-revaccination and 1 month post-revaccination over 1 month post-previous dose) will be tabulated when applicable.

The ratio of fold increase (pre to post-vaccination) of anti-RSVPreF3-specific antibody concentrations over the fold increase (pre to post-vaccination) of anti-RSV-A/-B neutralizing antibody titers will be tabulated using descriptive statistics and displayed graphically using scatter plots.

### Cell-mediated immune response

The kinetics of RSVPreF3-specific CD8+ T cells frequencies will be plotted as a function of time for participants with results available at all primary vaccination timepoints

Fold increase of the frequency of RSVPreF3-specific CD8+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 4-1BB, IL-2, TNF- $\alpha$ , IFN- $\gamma$ , IL-13, IL-17 at each post-primary vaccination timepoint over pre-vaccination (Day 1), at each post-revaccination over the corresponding pre-revaccination and at one month post-revaccination over 1 month post-previous dose in the RSV annual group.

### Safety (see section 5.4.4)

The prevalence of each solicited administration site event and solicited systemic event (any grade and grade 3) will be represented graphically over time for each group after each dose.

The following safety analyses have been added.

Summary tables of unsolicited adverse events and SAEs/pIMDs will be generated by SOC, **HLT** and PTs.

Safety analyses to be conducted by region in order to align with the immunogenicity analyses.

The number of each solicited events (any and Grade 3) that are ongoing beyond the 4-day follow-up period will be reported with the duration in days (mean, min, Q1, median, Q3, maximum) (see section 5.4.5).

The persistence modelling has been updated (see section 5.4.3.3).

## 8.1. Other changes in the SAP

Solicited events will be coded by MedDRA as per the following codes:

| Solicited event | Lower level term code | Corresponding Lower |
|-----------------|-----------------------|-------------------------|
| | | level term decode |
| Erythema | 10022061 | Injection site erythema |
| Fever | 10016558 | Fever |

The aim is to align the lower level term in the SAP with the coding done in CE domain in SDTM.

Clarification on how age at first dose in years will be computed (see section 10.1.3.1)

Clarification on how duration of events will be calculated (see section 10.1.3.6).

Clarification on counting rules for combining grade 3 solicited and unsolicited adverse events (see section 10.1.3.7)
212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

# 9. NON-STANDARD DATA DERIVATION RULES AND STATISTICAL METHODS

The following sections describe additional derivation rules and statistical methods which are not presented in section 10.1 (Business rules for standard data derivations and statistical methods).

# 9.1. Handling of missing data

#### 9.1.1. Dates

When partially completed dates (i.e. with missing day or month) are used in calculations, the following rules will be applied:

- Adverse event start dates with missing day:
  - If the month is not the same as the vaccine dose, then the imputed start date will be the 1<sup>st</sup> of the month
  - If the event starts in the same month as the vaccine dose, the flag indicating if the event occurred before or after vaccination (AE.AESTRTPT) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the vaccine dose given during that month. If 'before vaccination' is selected, the imputed date will be one day before the vaccine dose given during that month.
- Adverse event start dates with missing day and month:
  - If the year is not the same as the vaccine dose, then the imputed start date will be the 1<sup>st</sup> of January.
  - If the event starts in the same year as the vaccine dose, the flag indicating if the event occurred before or after vaccination (AE.AESTRTPT) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first vaccine dose given during that year. If 'before vaccination' is selected, the imputed date will be one day before the first vaccine dose given during that year.
- Adverse event end dates with missing day: the imputed end date will be the last day of the month (30 or 31) or the study conclusion date whichever comes first.
- Adverse event end dates with missing day and month: the imputed end date will be the last day of the year (31st of December) or the study conclusion date whichever comes first.

All incomplete concomitant medication/vaccination start/end date will follow the rules above.

## 10. ANNEXES

# 10.1. Business rules for standard data derivations and statistical methods

This section contains standard rules for data display and derivation for clinical and epidemiological studies.

## 10.1.1. Attributing events to vaccine doses

The dose relative to an event is the most recent study dose given to a participant prior to the start of a given event. For example, if the start date of an adverse event is between Dose 1 and Dose 2, the relative dose will be Dose 1.

If an event starts on the same day as a study dose, the relative dose will be derived from the additional information provided in the case report form (CRF) using the contents of the flag indicating if the event occurred before or after study dose. If 'after vaccination is selected, the relative dose for the event will be the one administered on the start day of the event. If 'before vaccination is selected, the relative dose for the event will be the dose prior to this one.

## 10.1.2. Handling of missing data

#### 10.1.2.1. Dates

When partially completed dates (i.e. dates missing a day and/or month) are used in calculations, the following standard rules will be applied:

- A missing day will be replaced by 15
- A missing day and month will be replaced by June 30<sup>th</sup>.

See also exceptions in section 9.1.

#### 10.1.2.2. Laboratory data

Refer to section 5.1.2 for more details

#### 10.1.2.3. Daily recording of solicited events

#### 10.1.2.3.1. Studies with paper diaries

For studies using paper diaries which have questions in the CRF indicating the presence or absence of solicited events, the following rules are applicable:

• Denominators for the summary of administration site (or systemic) solicited events will be calculated using the number of participants who respond "Yes" or "No" to the question concerning the occurrence of administration site (or systemic) events.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

- When a specific solicited event is marked as having not occurred following a specific study dose (i.e. SDTM CE.CEOCCUR=N for the specified post-dose period for the event in question), all daily measurements will be imputed as Grade 0.
- When a specific solicited event is marked as having occurred following a specific study dose (i.e. SDTM CE.CEOCCUR=Y for the specified post-dose period for the event in question), any missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the solicited event summary tables.
- When the occurrence of a specific solicited event is not present (i.e. SDTM CE.CEOCCUR is neither Y nor N for the specified post-dose period for the event in question) but the group of solicited events (administration site or systemic) is marked as having occurred (i.e. SDTM CE.CEOCCUR=Y), all missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the solicited event summary tables.

The following table shows how participants contribute to each category for a specific solicited event over the Day X to Day Y post-dose period:

| Solicited event category | Participants included in the calculation of the numerator |
|---|---|
| Any | All participants with at least one occurrence of the adverse event at grade 1, grade 2, or grade 3 between Day X and Day Y or with the adverse event marked as present and at least one missing daily recording between Day X and Day Y |
| At least grade 1 | All participants with at least one occurrence of the adverse event at grade 1, grade 2, or grade 3 between Day X and Day Y |
| At least grade 2 | All participants with at least one occurrence of the adverse event at grade 2 or grade 3 between Day X and Day Y |
| At least grade 3 | All participants with at least one occurrence of the adverse event at grade 3 between Day X and Day Y |

#### 10.1.2.4. Unsolicited adverse events

Unsolicited adverse event summaries are including serious adverse events unless specified otherwise.

Missing severity, relationship with study vaccine, and outcome of unsolicited adverse events will not be replaced and will appear as 'UNKNOWN' when displayed in a statistical output.

#### 10.1.3. Data derivation

#### 10.1.3.1. Age at first dose in years

When age at first dose is to be displayed in years, it will be calculated as the number of complete calendar years between the date of birth and the date of first dose. For example:

DOB = 
$$10SEP1983$$
, Date of first dose =  $09SEP2018 -> Age = 34$  years

DOB = 
$$10SEP1983$$
, Date of first dose =  $10SEP2018 -> Age = 35$  years

In this study, we will collect only the year of birth. The rules for handling missing day and/or month in the DOB are given in section 10.1.2.1.

Since only the year of birth will be collected in the eCRF, there might be some discrepancies between the age computed using standard derivation rules and the age category used in SBIR for the minimization.

Therefore, for the analysis by age, the age categories defined in Table 4 will be determined according to the information entered in SBIR (variable AGEGRP in SDTM SUPPDM), except for ">65 YOA" category which will be obtained using the derived age because this category is not used in SBIR for minimization

#### 10.1.3.2. Temperature

Temperatures will be presented in degrees Celsius (°C). Temperatures reported in degrees Fahrenheit (°F) will be converted as follows:

Temperature (Celsius) = 
$$((Temperature (Fahrenheit) - 32) \times 5)/9$$

#### 10.1.3.3. Numerical serology results

Numerical serology results will be derived from the content of IS.ISORRES in the SDTM dataset. For humoral assays with a specific cut-off, the following derivation rules apply:

| IS.ISORRES | Derived value |
|-----------------------------------------------------|---------------|
| "NEG", "-", or "(-)" | cut-off/2 |
| "POS", "+", or "(+)" | cut-off |
| "< value" and value is <= assay cut-off | cut-off/2 |
| "< value" and value is > assay cut-off | Value |
| "> value" and value is < assay cut-off | cut-off/2 |
| "> value" and value is >= assay cut-off | Value |
| "value" and value is < cut-off | cut-off/2 |
| "value" and value is >= cut-off and value is <=ULOQ | value |
| "value" and value is > ULOQ | ULOQ* |
| All other cases | Missing |

<sup>\*</sup>This rule will be used to compute descriptive statistics (GMTs, fold increase etc).

212496 (RSV OA=ADJ-004) Statistical Analysis Plan Amendment 1

## 10.1.3.4. Geometric mean titres (GMTs) and concentrations (GMCs)

GMT or GMC calculations are performed by taking the inverse logarithm of the mean of the log titre or concentration transformations. Non quantifiable antibody titres or concentrations will be converted as described in section 10.1.3.3 for the purpose of GMT/GMC calculation. Cut-off values are defined by the laboratory before the analysis.

#### 10.1.3.5. Onset day

The onset day for an event (e.g. AE, concomitant medication/vaccination) is the number of days between the last study dose and the start date of the event. This is 1 for an event occurring on the same day as a study dose (and reported as starting after study dose).

#### 10.1.3.6. Duration of events

The duration of an event with a start and end date will be the difference between the start and end date plus one day, i.e. an event that starts on 3 March 2018 and ends on 12 March 2018 has a duration of 10 days.

The duration of solicited events will be calculated as the sum of the individual days with the event reported at grade 1 or higher or reported as missing ("NOT DONE"), during the solicited event period. The duration of solicited events ongoing beyond the solicited period will be calculated as end date – start date + 1. The goal of this change was to align this text with the standard programs.

#### 10.1.3.7. Counting rules for combining solicited and unsolicited adverse events

For output combining solicited and unsolicited adverse events, all serious adverse events will be considered systemic events since the administration site flag is not included in the expedited adverse event CRF pages. Unsolicited adverse events with missing administration site flag will also be considered systemic.

Multiple events with the same preferred term which start on the same day are counted as only one occurrence.

In case a solicited event is worsening to Grade 3 after the solicited period, it should be reported only in the following table.

Summary of grade 3 adverse events (solicited and unsolicited) within 30 days following each dose and overall

## 10.1.3.8. Counting rules for occurrences of solicited events

When the occurrences of solicited events are summarized, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurs. Also, in the case of co-administered study interventions, an administration site event recorded for a participant following multiple study interventions will be counted as only one occurrence.

## 10.1.4. Display of decimals

### 10.1.4.1. Percentages

Percentages and their corresponding confidence limits will be displayed with one decimal except for 100% in which case no decimal will be displayed.

## 10.1.4.2. Demographic/baseline characteristics statistics

The mean, median, and standard deviation for continuous baseline characteristics will be presented with one decimal.

The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values.

The maximum and minimum of transformed body temperatures will be displayed with one decimal.

#### 10.1.4.3. Serological summary statistics

For each assay, geometric mean titers (GMT) or concentrations (GMC) and their confidence limits will be presented with one decimal, as well as GMT/GMC fold increase from pre-dose.

The mean, median, standard deviation and quartile values for frequency of RSVPreF3 specific-CD4+ and CD8+ T cells and for the fold increase (post over pre-vaccination) will be presented with one decimal. The minimum and maximum values will be presented with no decimal.

### 10.1.5. Statistical methodology

## 10.1.5.1. Exact confidence intervals around proportions

The exact confidence intervals around within-group proportions are derived using the method of Clopper and Pearson [Clopper, 1934].

# 11. ADDITIONAL ANALYSES DUE TO THE COVID-19 PANDEMIC

Depending on how the Covid-19 situation evolves, the SAP might be amended to reflect the analysis corresponding to Covid-19.

## 12. REFERENCES

Clopper CJ, Pearson E. The Use of Confidence or Fiducial Limits Illustrated in the case of the Binomial. *Biometrika*. 1934;26:404-13.

David M-P, Van Herck K, Hardt K, Tibaldi F, Dubin G, Descamps D, et al. Long-term persistence of anti-HPV-16 and-18 antibodies induced by vaccination with the AS04-adjuvanted cervical cancer vaccine: modeling of sustained antibody responses. GYNECOLOGIC ONCOLOGY. 2009;115(3):S1–6.

Fraser C, Tomassini JE, Xi L, Golm G, Watson M, Giuliano AR, et al. Modeling the long-term antibody response of a human papillomavirus (HPV) virus-like particle (VLP) type 16 prophylactic vaccine. Vaccine 2007 May 22;25(21):4324-33

Pan W Akaike's information criterion in generalized estimating equations Biometrics, 57 (1) (2001), pp. 120-125

Rubin, D. B., Stern, H. S. AND Vehovar, V. Handling "don't know" survey responses: the case of the Slovenian plebiscite. Journal of the American Statistical Association 90, 1995, 822–828

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

| gsk | Statistical Analysis Plan |
|---|---|
| Title: | A phase 3, randomized, open-label, multi-country study to evaluate the immunogenicity, safety, reactogenicity and persistence of a single dose of the RSVPreF3 OA investigational vaccine and different revaccination schedules in adults aged 60 years and above. |
| eTrack study number and<br>Abbreviated Title | 212496 (RSV OA=ADJ-004) |
| Scope: | All data pertaining to the above study except the Safety Review Team analyses for the first 50 participants aged 80 years and above |
| Date of Statistical Analysis<br>Plan | Final: 9 February 2021 |

APP 9000058193 Statistical Analysis Plan Template V5 (Effective date: 1July2020)

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| LIS | TOF | ABBREV | IATIONS | 6 |
| 1. | DOC | JMENT H | HISTORY | 7 |
| 2. | OBJE | CTIVES/ | ENDPOINTS | 7 |
| 3. | 3.1. | | GNdesign | |
| 4. | | | TS | |
| | 4.1. | | for climinating data from Applyoic Cata | |
| | 4.2. | 4.2.1. | for eliminating data from Analysis Sets Randomized Set | |
| | | 4.2.1. | Elimination from Exposed Set (ES) | |
| | | 4.2.3. | Elimination from Per-protocol analysis Set (PPS) | |
| | | | 4.2.3.1. Excluded participants | |
| 5. | STAT | ISTICAL | ANALYSES | 16 |
| | 5.1. | | considerations | |
| | | 5.1.1. | Demography | |
| | | 5.1.2. | Immunogenicity | |
| | <b>-</b> 0 | 5.1.3. | Reactogenicity/Safety | |
| | 5.2. | 5.2.1. | s of demography and baseline characteristics | |
| | | 5.2.1.<br>5.2.2. | Analysis planned in the protocol | |
| | 5.3. | | endpoint(s) | |
| | 0.0. | 5.3.1. | | |
| | | 0.0 | 5.3.1.1. Humoral immune response – up to Month | |
| | 5.4. | Second | ary endpoint(s) | |
| | 0.4. | 5.4.1. | Humoral immune response | |
| | | 5.4.2. | Cell-mediated immune response | |
| | | 5.4.3. | Additional considerations | |
| | | | 5.4.3.1. Assessment of long-term persistence of the immune response at Months 12, 24 and 36 | |
| | | | after dose 1 | |
| | | E 4 4 | 5.4.3.2. Sensitivity analyses | |
| | | 5.4.4. | Safety analysis | |
| | | 5.4.5. | Additional considerations | |
| | | 5.4.6. | Sensitivity Analyses | |
| 6. | ANAL | YSIS IN | TERPRETATION | 24 |
| 7 | INITE | ΣΙΜ ΔΝΙΔ | LVSES | 24 |

| | | | | | 212496 (RSV OA=ADJ-<br>Statistical Analysis | |
|---|---|---|---|---|---|---|
| | 7.1. | Sequen | ce of analy | /ses | • | |
| | 7.2. | | | rations for interim analyses | | |
| 8. | | | | TOCOL DEFINED STATIST | | |
| | ANAL | YSIS | | | | 25 |
| 9. | | | | <b>DERIVATION RULES AND</b> | | |
| | 9.1. | | | ng data | | |
| | | 9.1.1. | Dates | | | 26 |
| 10. | | | | | | 26 |
| | 10.1. | | s rules for | standard data derivations a | | 26 |
| | | | | g events to vaccine doses | | |
| | | 10.1.2. | | of missing data | | |
| | | 10.1.2. | _ | Dates | | |
| | | | | Laboratory data | | |
| | | | | Daily recording of solicited | | |
| | | | 101112101 | 10.1.2.3.1. Studies with pa | | |
| | | | 10.1.2.4. | Unsolicited adverse events | | |
| | | 10.1.3. | | vation | | |
| | | | | Age at first dose in years | | |
| | | | | Temperature | | |
| | | | | Numerical serology results. | | |
| | | | | Geometric mean titres (GM | | |
| | | | | concentrations (GMCs) | | 29 |
| | | | 10.1.3.5. | Onset day | | |
| | | | 10.1.3.6. | Duration of events | | 29 |
| | | | | Counting rules for combining | | |
| | | | | unsolicited adverse events. | | 30 |
| | | | 10.1.3.8. | Counting rules for occurren | | |
| | | | | events | | 30 |
| | | 10.1.4. | Display of | f decimals | | 30 |
| | | | 10.1.4.1. | Percentages | | 30 |
| | | | 10.1.4.2. | Demographic/baseline cha | racteristics | |
| | | | | statistics | | 30 |
| | | | 10.1.4.3. | Serological summary statis | tics | 30 |
| | | 10.1.5. | | I methodology | | 31 |
| | | | 10.1.5.1. | Exact confidence intervals | around | |
| | | | | proportions | | 31 |
| 11. | ADDI <sup>*</sup> | TIONAL | ANALYSE | S DUE TO THE COVID-19 F | PANDEMIC | 31 |
| 12. | REFE | RENCES | 3 | | | 31 |

# 212496l Statistical Analysis Plan $\,$ 09 Feb2021l TMF-11813731 | 1.0 $\,$

## **CONFIDENTIAL**

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

# **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | Study groups, intervention and blinding foreseen in the study | S |
| Table 2 | Group names and definition for footnote in the TFLs | g |
| Table 3 | Pooled group names and definition for footnote in the TFLs | 10 |
| Table 4 | Sub-group names and definitions for footnote in the TFLs | 10 |
| Table 5 | Populations for analyses | 11 |
| Table 6 | List of elimination codes | 12 |
| Table 7 | Intensity grading scale for solicited events | 23 |

# 212496l Statistical Analysis Plan $\;$ 09 Feb2021l TMF-11813731 | 1.0

## **CONFIDENTIAL**

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

# **LIST OF FIGURES**

| | | PAGE |
|----------|-----------------------|------|
| Figure 1 | Study design overview | 8 |

#### 212496 | Statistical Analysis Plan 09 Feb 2021 | TMF-11813731 | 1.0


212496 (RSV OA=ADJ-004) Statistical Analysis Plan

## LIST OF ABBREVIATIONS

**AE** Adverse event

**AESI** Adverse Events of Special Interest

**CD** Community Dwelling

**CI** Confidence Interval

**COVID-19** Coronavirus Disease 2019

**CRF** Case Report Form

CTRS Clinical Trial Registry Summary

Eli Type Internal database code for type of elimination code

**ELISA** Enzyme-linked immunosorbent assay

ELU/mL ELISA unit per milliliter

**ES** Exposed Set

**GMC** Geometric mean antibody concentration

**GMT** Geometric mean antibody titre

**GSK** GlaxoSmithKline

IU/mL International units per milliliter

LL Lower Limit of the confidence interval

LTCF Long Term Care Facility

**MedDRA** Medical Dictionary for Regulatory Activities

NA Not Applicable

**PD** Protocol Deviation

**PPS** Per-Protocol Set

**SAE** Serious adverse event

**SAP** Statistical Analysis Plan

SBIR GSK Biologicals Internet Randomization System

**SD** Standard Deviation

**SDTM** Study Data Tabulation Model

UL Upper Limit of the confidence interval

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

# 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|------------------|---------------|------------------------|
| 15 February 2021 | First version | Final: 28 October 2020 |

# 2. OBJECTIVES/ENDPOINTS

| Objectives Endpoints | |
|---|---|
| Primary | |
| To evaluate the humoral immune response following a 1-dose primary schedule of RSVPreF3 OA investigational vaccine up to 12 months post-Dose 1. Humoral immune response at pre-vaccination (Day 1), 30 post-Dose 1 (Day 31), and at 6 and 12 months post-Dose 1 (Months 6 and 12), in a subset of participants: Neutralizing antibody titers against RSV-A Neutralizing antibody titers against RSV-B. | |
| Sec | ondary |
| To further evaluate the humoral immune response following a 1-dose primary schedule of RSVPreF3 OA investigational vaccine up to 12 months post-Dose 1. | Humoral immune response at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), and at 6 and 12 months post-Dose 1 (Months 6 and 12), in a subset of participants: RSVPreF3-specific Immunoglobulin G (IgG) antibody concentrations. |
| To evaluate the humoral immune response following 1 dose of the RSVPreF3 OA investigational vaccine and following revaccination doses, up to study end. | Humoral immune response at Months 18, 24, 30 and 36 post- Dose 1, and at 1 month after each revaccination dose (Months 13 and 25), in a subset of participants: Neutralizing antibody titers against RSV-A and RSV-B RSVPreF3-specific IgG antibody concentrations. |
| To evaluate the cell-mediated immune (CMI) response following 1 dose of the RSVPreF3 OA investigational vaccine and following revaccination doses up to study end. | <ul> <li>CMI response at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), at Months 6, 12, 18, 24, 30 and 36 post-Dose 1, and at 1 month after each revaccination dose (Months 13 and 25), in a subset of participants:</li> <li>Frequency of RSVPreF3-specific CD4+ and/or CD8+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 4-1BB, IL-2, TNF-α, IFN-γ, IL-13, IL-17.</li> </ul> |
| To evaluate the safety and reactogenicity of each vaccination schedule of the RSVPreF3 OA investigational vaccine in all participants. | <ul> <li>Occurrence of each solicited administration-site and systemic event during a 4-day follow-up period (i.e., on the day of vaccination and 3 subsequent days) after each vaccination.</li> <li>Occurrence of any unsolicited AE during a 30-day follow up period (i.e., on the day of vaccination and 29 subsequent days) after each vaccination.</li> <li>Occurrence of all SAEs and pIMDs up to 6 months after each vaccination.</li> <li>Occurrence of fatal SAEs, related SAEs and related pIMDs from first vaccination (Day 1) up to study end (Month 36).</li> </ul> |
| | iary |
| To further characterize immune responses to the RSVPreF3 OA investigational vaccine. | Any further exploratory immunology in a subset of participants, such as, but not limited to: Antibodies against specific protein F epitopes. Potential new immunological markers for protection. Frequency of RSVPreF3-specific CD4+ and/or CD8+ T cells expressing one or any combination of immune marker(s) nt, SAE = serious adverse event, pIMD = potential immune-mediated |

CMI = cell-mediated immunity, AE = adverse event, SAE = serious adverse event, pIMD = potential immune-mediated disease.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

## 3. STUDY DESIGN

## 3.1. Overall design

## Figure 1 Study design overview



N = number of participants; D = Day; M = Month; AE = adverse event; HI = humoral immunity; CMI = cell-mediated immunity; pIMD = potential immune-mediated disease; SAE = serious adverse event.

- = blood sample for humoral immune responses (only applicable for the 345 participants of the RSV\_annual group; and for all participants of the RSV\_flexible revaccination and RSV\_1dose groups)
- = blood sample for CMI (only applicable for the ~345 participants of the RSV\_annual group, and ~115 participants each from the RSV\_flexible revaccination and RSV\_1dose groups).

Note: For group RSV\_annual, Revaccination Year 1 = Month 12; Revaccination Year 2 = Month 24.

- \* Visit and follow-up of solicited events, unsolicited AEs, SAEs and pIMDs only applicable for RSV annual group
- \*\* For the RSV\_annual group, the same ~345 participants will be part of both the HI and CMI subsets. The remaining ~645 participants will have no blood draws, and will only be followed up for safety and reactogenicity.
- \*\*\*For those participants in the RSV\_annual group without blood sample collections, visits at Months 6, 18, 30 and 36 may be through a phone contact. However, phone contact should be attempted only if site visit is not possible at Months 6, 18, 30 and 36.
- Type of study: self-contained.
- **Experimental design**: Phase 3, randomized, open-label, multi-country study with 3 parallel groups (see Figure 1).
- **Duration of the study**: ~ 36 months for each participant.
- **Primary completion date**: Month 12.
- Control: none.
- **Blinding**: open-label. Refer to the protocol for details.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

- **Data collection**: standardized electronic Case Report Form (eCRF). Solicited events and unsolicited AEs will be collected using a participant Diary card (paper Diary card).
- Safety monitoring: the study will be conducted with oversight by the project Safety Review Team (SRT). Please refer to protocol for the description of review of safety data by the SRT.
- Study groups: refer to Figure 1 and Table 1 for an overview of the study groups

Table 1 Study groups, intervention and blinding foreseen in the study

| Number of | | | Intervention | | | Blinding |
|---|---|---|---|---|---|---|
| Study Groups | participant<br>s | Age | Primary vaccination | Revaccination<br>Year 1 (Month<br>12) | Revaccination<br>Year 2 (Month<br>24) | Open |
| RSV_annual* | ~990 | ≥60 years | RSVPreF3 OA investigational vaccine | RSVPreF3 OA investigational vaccine | RSVPreF3 OA investigational vaccine | Х |
| RSV_flexible revaccination** | ~330 | ≥60 years | RSVPreF3 OA investigational vaccine | | | Х |
| RSV_1dose | ~330 | ≥60 years | RSVPreF3 OA investigational vaccine | (none) | (none) | Х |

<sup>\*</sup> RSV\_annual group will be split in 3 technical groups in SBIR in order to have a randomization ratio of 1:1:1:1: for treatment allocation and avoid predictability.

• Groups and sub-groups definition for analysis: Refer to the tables below for a description of the groups and subgroups labels that will be used in the Tables Figures and Listings (TFLs).

For some of the analyses up to 12 months post dose 1, the 3 study groups will be pooled, and from Month 13, the RSV\_flexible revaccination and RSV\_1dose groups will be pooled, at applicable timepoints. The following group names will be used in the TFLs:

Table 2 Group names and definition for footnote in the TFLs

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | RSV_annual | Participants receiving the first dose (Dose 1) of RSVPreF3 OA investigational vaccine at Day 1, followed by a revaccination dose at 12 months post-Dose 1 and at 24 months post-Dose 1 |
| 2 | RSV_flexible revaccination | Participants receiving the first dose (Dose 1) of RSVPreF3 OA investigational vaccine at Day 1 and a revaccination dose will be given whenever a revaccination would be needed |
| 3 | RSV_1dose | Participants receiving a single dose (Dose 1) of RSVPreF3 OA investigational vaccine at Day 1 |

<sup>\*\*</sup>Based on immunogenicity data from this study and efficacy results from the Phase 3 study RSV OA=ADJ-006, a revaccination might be decided for this group.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

Table 3 Pooled group names and definition for footnote in the TFLs

| Pooled Group label in tables | Groups to be pooled | Pooled definition for footnote | Comment |
|---|---|---|---|
| All | RSV_annual,<br>RSV_flexible<br>revaccination and<br>RSV_1dose | Participants receiving one dose of RSVPreF3 OA investigational vaccine in all three groups | Applicable on data reported up to Month 12 |
| Flexible+1dose | RSV_flexible<br>revaccination, and<br>RSV_1dose | Participants receiving one dose of RSVPreF3 OA investigational vaccine in the RSV_flexible revaccination, and RSV_1dose groups | Applicable on data reported from Month 13 |

Table 4 Sub-group names and definitions for footnote in the TFLs

| Sub-analysis | Subgroup order in tables | Subgroup label in tables | Subgroup definition for footnote |
|---|---|---|---|
| By age | 1 | ≥65YOA | ≥65 years old participants |
| | 2 | ≥70YOA | ≥70 years old participants |
| | 3 | ≥80YOA | ≥80 years old participants |
| | 4 | 60-69YOA | 60-69 years old participants |
| | 5 | 70-79YOA | 70-79 years old participants |
| By sex | 1 | Female | Female |
| | 2 | Male | Male |
| By region | 1 | North America | Participants from North America<br>(United States of America) |
| | 2 | Europe | Participants from Europe (Finland, Germany) |
| | 3 | Asia | Participants from Asia (Japan, Taiwan) |

YOA = Years of age

#### Allocation of participants to assay subsets

Allocation of participants to assay subsets will be performed using SBIR. The subsets are detailed below.

| | RSV_annual | RSV_flexible revaccination | RSV_1dose |
|---|---|---|---|
| HI subset | ~345* | All participants (~330) | All participants (~330) |
| CMI subset | ~345* | ~115 | ~115 |

<sup>\*</sup>For the RSV\_annual group, the same ~345 participants will be part of both the HI and CMI subsets. The remaining ~645 participants will have no blood draws, and will only be followed up for safety and reactogenicity.

- **HI subset:** ~345 participants from the RSV\_annual group, and all participants from the RSV\_flexible revaccination and RSV\_1dose groups. These participants will have blood samples collected for testing of humoral immunity at each visit applicable for their study group.
- **CMI subset**: ~345 participants from the RSV\_annual group, and ~115 participants each from the RSV\_flexible revaccination and RSV\_1dose groups. These participants will have additional blood samples collected for CMI testing at each visit applicable for their study group.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

## 4. ANALYSIS SETS

#### 4.1. Definition

Table 5 Populations for analyses

| Analysis set | Description |
|---|---|
| Enrolled set | Participants who agreed to participate in a clinical study after completion of the |
| | informed consent process. |
| Exposed set (ES) | All participants who received at least 1 dose of the study intervention. The |
| | allocation in a group is done in function of the administered intervention. |
| Per Protocol set (PPS) | All participants who received at least 1 dose of the study intervention to which they |
| , , | are randomized and have post-vaccination data, minus participants with protocol |
| | deviations that lead to exclusion. |

The primary analysis for immunogenicity will be performed on the Per Protocol set (PPS). If in any study group the percentage of vaccinated participants with serological results excluded from the PPS for immunogenicity is at least 10%, a second analysis will be performed on the Exposed Set (ES). The immunogenicity analysis will be performed overall, by sex, by age category (age at Dose  $1: \ge 65 \text{ YOA}, \ge 70 \text{ YOA}, \ge 80 \text{ YOA}, 60-69 \text{ YOA}$  and 70-79 YOA, and by region (North America, Europe, Asia).

# 4.2. Criteria for eliminating data from Analysis Sets

#### 4.2.1. Randomized Set

All participants who will be randomized to 1 of the 3 study groups at Day 1 will be included in the Randomized Set. Code 1010 (Vaccine number not allocated) will be used for identifying participants eliminated from the Randomized Set (Table 6)

# 4.2.2. Elimination from Exposed Set (ES)

Code 1030 (Study intervention not administered at all), 800 (Fraudulent data) and code 900 (invalid informed consent) will be used for identifying participants eliminated from the ES.

## 4.2.3. Elimination from Per-protocol analysis Set (PPS)

#### 4.2.3.1. Excluded participants

A participant will be excluded from the populations of analysis under the following conditions

- For codes 800, 900, 1010, 1030 and 1050: participants will be eliminated for all visits
- For codes 1040, 1070, 1080, 1090, 2010, 2040, 2050, 2080: participants will be eliminated from a specific visit (at which the condition is met) onwards.
- For codes 2090, 2100, 2120, 2130: participants will be eliminated at the specific visit at which the condition is met.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

# Table 6 List of elimination codes

| Code | Condition under which the code is used | Visit (timepoints) where the code is checked | Applicable for analysis set |
|---|---|---|---|
| 800 | Fraudulent data | All | ES and PPS |
| 900 | Invalid informed consent | All | ES and PPS |
| 1010 | Vaccine number not allocated | Day 1 | Randomized Set,<br>ES, PPS |
| 1030 | Study intervention not administered at all | All | ES and PPS |
| 1040 | Administration of concomitant vaccine(s) forbidden in the protocol • Any investigational or non-registered vaccine other than the study vaccine used during the study period beginning 30 days before the first dose of study vaccine, or planned use during the study period. • Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before each dose and ending 30 days after each dose of study vaccine administration, with the exception of inactivated, split virion and subunit influenza vaccines which can be administered up to 14 days before or from 14 days after each study vaccination. • Previous vaccination with an | All | PPS |
| 1050 | RSV vaccine Randomization failure | Day 1 | PPS |
| 1070 | Vaccine administration not according to protocol Incomplete vaccination course | Vaccination visits at Day 1, Month 12, and 24 Months 12 and 24 are applicable to the | PPS |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

| C 1 | Statistical Ar | | |
|---|---|---|---|
| Code | Condition under which the code | Visit (timepoints) | Applicable for |
| | is used | where the code is | analysis set |
| | | checked | |
| | Participant was vaccinated | RSV_annual group | |
| | with the correct vaccine but | only | |
| | containing a lower volume | | |
| | Participant was re-vaccinated while it was not planned | | |
| | - | | |
| | Route of the study intervention is not intramuscular | | |
| | Wrong reconstitution of<br>administered vaccine | | |
| 1080 | Vaccine administration after a | Day 1, Month 12, and | PPS |
| | Temperature deviation | 24 | |
| | • Vaccine administered despite a | Months 12 and 24 are | |
| | Good Manufacturing Practices | applicable to the | |
| | (GMP) no-go temperature | RSV_annual group | |
| | deviation | only | |
| 1090 | Vaccine administration after | Day 1, Month 12, and | PPS |
| | expiration | 24 | |
| | - | Months 12 and 24 are | |
| | | applicable to the | |
| | | RSV annual group | |
| | | only | |
| 2010 | Protocol deviation linked to | All | PPS |
| 2010 | inclusion/exclusion criteria | 1 111 | |
| 2040 | | A 11 | DDC |
| 2040 | Administration of any medication | All | PPS |
| | forbidden by the protocol | | |
| | Any investigational or non- | | |
| | registered medication used | | |
| | during the study period | | |
| | Administration of long-acting | | |
| | immune-modifying drugs at | | |
| | any time during the study | | |
| | period (e.g. <i>infliximab</i> ) | | |
| | Immunoglobulins and/or any has a medicate a desiriate and | | |
| | blood products administered during the study period | | |
| | Chronic administration (defined as more than 14) | | |
| | (defined as more than 14 consecutive days in total) of | | |
| | immunosuppressants or other | | |
| | minumosuppressants of other | | |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

| ~ - | Statistical Analy | | |
|---|---|---|---|
| Code | Condition under which the code is used | Visit (timepoints) where the code is checked | Applicable for analysis set |
| | immune-modifying drugs during the period starting 90 days prior to the study vaccine administration or planned administration during the study period. For corticosteroids, this will mean prednisone ≥20 mg/day, or equivalent. | | |
| 2050 | Intercurrent medical condition | All | PPS |
| | • Participants may be eliminated from the PPS for immunogenicity if, during the study, they incur a condition that has the capability of altering their immune response (intercurrent medical condition) or are confirmed to have an alteration of their initial immune status. | | |
| 2080 | Participants did not comply with dosing schedule | Month 12 and 24 | PPS |
| | • RSV_annual: number of days between dose 1 and revaccination dose at Month 12 is outside [350-380 days] | | |
| | • RSV_annual: number of days between dose 1 and revaccination dose at Month 24 is outside [715-745 days] | | |
| 2090 | Participants did not comply with blood sample schedule | Day 31, Month 6, 12, 13, 18, 24, 25, 30, 36 | PPS |
| | • Number of days between dose 1 and Day 31 blood sample is outside [30-42 days] | | |
| | • Number of days between dose 1 and Month 6 blood sample is outside [180-210 days] | | |
| | Number of days between dose 1 and Month 12 blood sample is outside [350-380 days] | | |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

| | Statistical Analysis | | |
|---|---|---|---|
| Code | Condition under which the code is used | Visit (timepoints) where the code is checked | Applicable for analysis set |
| | Number of days between Month 12 and Month 18 blood sample is outside [180-210 days] | | |
| | • Number of days between dose 1 and Month 24 blood sample is outside [715-745 days] | | |
| | Number of days between Month 24 and Month 30 blood sample is outside [180-210 days] | | |
| | Number of days between dose 1 and Month 36 blood sample is outside [1080-1110 days] | | |
| | For RSV_annual group only: | | |
| | • Number of days between revaccination at Month 12 and Month 13 blood sample is outside [30-42 days] | | |
| | Number of days between<br>revaccination at Month 24 and<br>Month 25 blood sample is<br>outside [30-42 days] | | |
| 2100 | Serological results not available post-vaccination | Day 31, Month 6, 12, 13, 18, 24, 25, 30, 36 | PPS |
| | No immunological result at visit x for all the following tests: RSV A/B Neutralizing antibody titer, RSVPreF3-specific IgG antibody concentration and RSVPreF3-specific CD4+/CD8+ T cells frequency | Month 13 and 25 are applicable to the RSV_annual group only | |
| 2120 | Obvious incoherence or abnormality or error in laboratory data | Day 1, 31, Month 6, 12, 13, 18, 24, 25, 30, 36 | PPS |
| | Unreliable released data as a result of confirmed sample mismatch or confirmed inappropriate sample handling at laboratory | | |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

## 5. STATISTICAL ANALYSES

Standard data derivation rules and stat methods are described in section 10.1 while the study specific data derivation rules and stat methods are described in section 9.

For the sake of analysis, data up to Month 12 will be analyzed by group (RSV\_annual, RSV\_flexible revaccination and RSV\_1dose), and also the 3 groups will be pooled. From Month 13, the analysis will be tabulated by group, and also for RSV\_annual versus the pooled RSV\_flexible revaccination and RSV\_1dose groups, at applicable time points.

If more than 5% of participants in the RSV\_annual group received only 1 dose or only 2 doses, an analysis by subgroup according to the number of dose(s) administered will be performed. The goal of this analysis is to describe the characteristics of participants in the RSV\_annual group who ultimately receive different numbers of revaccination doses in order to rule out the possibility of systematic differences between these subgroups.

#### 5.1. General considerations

## 5.1.1. Demography

For a given participant and a given demographic variable, missing measurements will not be replaced.

## 5.1.2. Immunogenicity

- Any missing or non-evaluable immunogenicity measurement will not be replaced. The descriptive analysis performed for each assay at each time point will exclude participants with a missing or non-evaluable measurement.
- The geometric mean titers/concentrations (GMTs/GMCs) will be computed by taking the anti-logarithm of the arithmetic mean of the log<sub>10</sub> transformed titers/concentrations.
- A seronegative participant will be defined as a participant whose antibody titer/concentration is below the cut-off value of the assay. A seropositive participant is a participant whose antibody titer/concentration is greater than or equal to the cut-off value of the assay.
- Antibody titers/concentrations below the assay cut-off will be given an arbitrary value of half the assay cut-off for the purpose of GMT/GMC calculation.
- Antibody titers/concentrations above the Upper Limit of Quantification (ULOQ) value will be given the ULOQ value for the purpose of GMT/GMC calculation.
- The mean geometric increase (MGI) is calculated by the geometric mean of ratios of antibody titer/concentrations of each post-primary vaccination time point over preprimary vaccination (Day 1).

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

## 5.1.3. Reactogenicity/Safety

- For a given participant and the analysis of solicited events within 4 days post-vaccination, missing or non-evaluable measurements will not be replaced. Therefore, the analysis of solicited events will include only vaccinated participants with documented solicited safety data (i.e., paper diary completed).
- For analysis of unsolicited AEs, SAEs, pIMDs and concomitant medications, all vaccinated participants will be considered. Participants who did not report an event or concomitant medication will be considered as participants without the event or the concomitant medication, respectively.

# 5.2. Analysis of demography and baseline characteristics

## 5.2.1. Analysis planned in the protocol

Descriptive summaries will be performed for each group (RSV\_annual, RSV\_flexible revaccination and RSV\_1dose) and overall. The same will be performed in each subset (humoral immune subset and CMI subset).

Demographic/baseline characteristics (age at vaccination in years, sex, race, ethnicity, type of residence (CD/LTCF) and smoking status) will be summarized using descriptive statistics:

- Frequency tables will be generated for categorical variables such as race.
- Mean, median, standard deviation and range will be provided for continuous data such as age.
- The distribution of participants will be tabulated as a whole and per group, for each age category and for each subset.

The number of doses of the study intervention administered will be tabulated by group.

Withdrawal status will be summarized by group using descriptive statistics:

- The number of participants enrolled into the study as well as the number of participants excluded from Per Protocol (PP) analyses will be tabulated.
- The numbers of withdrawn participants will be tabulated according to the reason for withdrawal.

Participant disposition in the ES and PPS will be reported as a whole and per group, and for each age category.

• The number and percentage of participants using concomitant medication (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) during the 4-day follow-up period (i.e., on the day of vaccination and 3 subsequent days) and during the 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) will be summarized by group after each vaccine dose and overall, and after the revaccination.

#### 212496 | Statistical Analysis Plan 09 Feb 2021 | TMF-11813731 | 1.0


212496 (RSV OA=ADJ-004) Statistical Analysis Plan

#### 5.2.2. Additional considerations

- The analysis of demographic characteristics by group will be performed on the ES and on the PPS.
- Demography and baseline characteristics will also be summarized by country.
- The smoking status and exposure history of participants will be tabulated according to the
  - number of years of smoking exposure for both current and former smokers.
  - number of years of smoking exposure, summarized separately for tobacco and electronic smoking devices

## 5.3. Primary endpoint(s)

## 5.3.1. Analysis planned in the protocol

The primary analysis for immunogenicity will be performed on the Per Protocol set (PPS). If in any study group the percentage of vaccinated participants with serological results excluded from the PPS for immunogenicity is at least 10%, a second analysis will be performed on the Exposed Set (ES).

## 5.3.1.1. Humoral immune response – up to Month 12

The analysis of the primary vaccination time points up to Month 12 will be performed for each group and for the 3 groups pooled. For each time point with blood sample collection for humoral immune response up to Month 12 and for each assay (RSV-A/-B neutralization assays), unless otherwise specified, the following analyses will be performed:

## Within groups evaluation:

- Percentage of participants with antibody titers/concentrations above a positivity cutoff and their exact 95% confidence interval (CI) will be tabulated.
- GMTs/GMCs and their 95% CI will be tabulated and represented graphically. Furthermore, to account for all the time points at which the blood samples are collected, a mixed model will be fitted, from which the GMTs/GMCs will be computed.
- Antibody titers/concentrations will be displayed using reverse cumulative curves.
- The MGI i.e. geometric mean of ratios of antibody titer/concentrations will be tabulated with 95% CI.
- Individual post-vaccination results (at Days 31 and at Months 6 and 12) versus prevaccination results (Day 1) will be plotted using scatter plots.
- Distribution of the fold increase of the antibody titers/concentrations (post- over preprimary vaccination titers) will be tabulated.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

## 5.4. Secondary endpoint(s)

## 5.4.1. Humoral immune response

The same analyses as described above for the primary endpoint will be performed for PreF3 IgG ELISA up to Month 12 and for each time point with blood sample collection for humoral immune response **from study Month 13 up to study end** and for each assay (preF3 IgG **ELISA and RSV-A/-B neutralization assays**). The analysis of the post-primary vaccination time points from study Month 13 up to study end will be performed for each group and for the pooled RSV\_flexible revaccination and RSV\_ldose groups.

Only the analyses requiring further clarification of the exact time points analyzed are summarized below:

## Within groups evaluation:

- The MGI i.e. geometric mean of ratios of antibody titer/concentrations will be tabulated with 95% CI:
  - For each post-primary vaccination time point (at Months 18, 24, 30 and 36 when applicable) over pre-primary vaccination (Day 1),
  - For each post-revaccination time point over corresponding pre-revaccination (Months 12/24) in the RSV annual group,
  - For 1 month post-revaccination at Month 12 (Month 13) over 1 month post-Dose 1 vaccination (Day 31) in RSV annual group.
  - For 1 month post-revaccination at Month 24 (Month 25) over 1 month post-revaccination at Month 12 (Month 13) in RSV annual group
- Individual post-primary vaccination results (at Months 18, 24, 30 and 36 when applicable) versus pre-vaccination results (Day 1) by group and individual post-revaccination results versus the corresponding pre-revaccination results (Months 12/24) in the RSV annual group will be provided using scatter plots.
- Distribution of the fold increase of the antibody titers/concentrations (post- over preprimary vaccination dose, post- over the corresponding pre-revaccination and 1 month post-revaccination over 1 month post-previous dose) will be tabulated when applicable.
- The ratio of fold increase (pre to post-vaccination) of anti-RSVPreF3-specific antibody concentrations over the fold increase (pre to post-vaccination) of anti-RSV-A/-B neutralizing antibody titers will be tabulated using descriptive statistics and displayed graphically using scatter plots.

In addition, the following evaluations will be performed:

• The kinetics of GMTs/GMCs will be plotted as a function of time for participants with results available at all post-primary vaccination time points.

The immunogenicity analysis will be performed overall, by sex, age category (age at Dose  $1: \ge 65 \text{ YOA}, \ge 70 \text{ YOA}, \ge 80 \text{ YOA}, 60-69 \text{ YOA}$  and 70-79 YOA, and region (North America, Europe, Asia).

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

## 5.4.2. Cell-mediated immune response

#### Within groups evaluation:

The following parameters will be summarized by group at each time point for which blood samples are collected, for the 3 groups pooled for time points up to study Month 12, for the pooled RSV\_flexible revaccination and RSV\_1 dose up to study end using descriptive statistics (N, geometric mean, min, Q1, median, Q3, max) in the CMI subset:

- Frequency of RSVPreF3-specific CD4+ and/or CD8+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13, IL-17.
- The kinetics of RSVPreF3-specific CD4+ T cells frequencies will be plotted as a function of time for participants with results available at all primary vaccination time points.
- Fold increase of the frequency of RSVPreF3-specific CD4+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13, IL-17 at each post-primary vaccination time point over prevaccination (Day 1) by group, at each post-revaccination over the corresponding prerevaccination and at one month post-revaccination over 1 month post-previous dose in the RSV\_annual group.

The immunogenicity analysis will be performed by sex, age category (age at Dose  $1: \ge 65$  YOA,  $\ge 70$  YOA,  $\ge 80$  YOA, 60-69 YOA and 70-79 YOA, and region (North America, Europe, Asia).

#### 5.4.3. Additional considerations

• **Descriptive statistics** of the cell-mediated immune response will be tabulated and displayed graphically using boxplots (min, Q1, median, Q3, max), by group and timepoint.

The RSVPreF3-specific CD4+ T cell frequencies will be obtained by subtracting the background value to the antigen-induced value, and by setting to 1 all values less than or equal to zero for geomean calculation and graphical representation. Frequencies will be expressed as the number of cells per million of CD4+ T cells.

More specifically, the frequencies of RSVPreF3-specific CD4+ T cells expressing at least 2 activation markers including at least one cytokine [ Freq<sup>2+</sup> ] will be computed as follows:

$$Freq_{Background}^{2+} = \frac{n_{background}^{2+}}{N_{Background}^{CD4}}$$
 and  $Freq_{Induction}^{2+} = \frac{n_{Induction}^{2+}}{N_{Induction}^{CD4}}$ ,

And

$$Freq_{Specific}^{2+} = Freq_{Induction}^{2+} - Freq_{Background}^{2+}$$

# 212496 | Statistical Analysis Plan 09 Feb 2021 | TMF-11813731 | 1.0


212496 (RSV OA=ADJ-004) Statistical Analysis Plan

where

 $n_{Background}^{2+}$  = number of CD4+ T cells expressing at least 2 activation markers including at least one cytokine after stimulation with medium only (background)

 $n_{Induction}^{2+}$  = number of CD4+ T cells expressing at least 2 activation markers including at least one cytokine after stimulation with a pool of peptides covering RSVPreF3 (induction)

 $N_{\it Back/Ind}^{\it CD4}$  = Total number of CD4 T cells involved in the assay (background or induction)

Same computations will be done for all CMI responses that will be analysed, i.e.:

- Frequency of RSVPreF3-specific CD4+ and/or CD8+T-cells expressing at least 2 activation markers including at least 1 cytokine\* among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13, and IL-17, as measured by ICS using PBMCs.
  - \* cytokines are IL-2, TNF-α, IFN-γ, IL-13, and IL-17

# 5.4.3.1. Assessment of long-term persistence of the immune response at Months 12, 24 and 36 after dose 1.

The exploratory analysis for modelling the long-term persistence of immune response (humoral and cellular) post dose 1 vaccination will constitute of the following;

- A piece-wise linear mixed model, power law model and modified power law model [David, 2009] for repeated measurements (all data available from Day 1, 31 and Month 6, 12, 18, 24, 30, 36 post dose 1 vaccination, for the 3 groups pooled for time points up to study Month 12, for the pooled RSV\_flexible revaccination and RSV 1dose from Month 13 up to study end) will be used to model over time
  - the frequency of RSVPreF3-specific CD4+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 4-1BB, IL-2, TNF-α, IFN-γ, IL-13, IL-17.
  - the neutralizing antibody titers against RSV-A, RSV-B and RSVPreF3-specific IgG antibody concentrations.
- The three models based on data up to M36 will be presented graphically. Models based on data up to M12 and on data up to M36 will be presented side by side.

#### 5.4.3.2. Sensitivity analyses

- In case the COVID-19 pandemic is still ongoing during the study conduct, the following sensitivity analyses might be considered.
  - During the assessment of long-term persistence of the immune response, the models described in section 5.4.3.1 might be fitted taking into account;
     Participants who received the first dose of study vaccine and with full follow-up (attending all study visits)

#### 212496 | Statistical Analysis Plan 09 Feb 2021 | TMF-11813731 | 1.0


212496 (RSV OA=ADJ-004) Statistical Analysis Plan

 Similarly, a mixed model will be fitted for the evaluation of GMT/GMC based on participants with full follow-up (attending all study visits).

The goal of this sensitivity analysis is to determine the extent to which results might be impacted by considering the different scenarios.

## 5.4.4. Safety analysis

#### Primary vaccination and revaccination dose:

The safety analysis will be performed on the ES. A descriptive analysis by group, for the 3 groups pooled up to Month 12, for the RSV\_flexible revaccination and RSV\_ldose groups pooled vs RSV\_annual group from study Month 13 up to study end will present a summary of:

- The number and percentage of participants with at least one administration site event (solicited and unsolicited), with at least one systemic event (solicited and unsolicited) and with any AE during the 4-day or 30-day follow-up period will be tabulated with exact 95% CI after each dose. The same computations will be done for Grade 3 AEs, and for Grade 3 non-serious AEs and for AEs resulting in medically attended visit.
- The number and percentage of participants reporting each individual solicited administration site event (any grade, Grade 3 and resulting in medically attended visit) and solicited systemic event (any grade, Grade 3 and resulting in medically attended visit) during the 4-day follow-up period (i.e., on the day of vaccination and 3 subsequent days) will be tabulated for each group after each dose.
- For fever, the number and percentage of participants reporting fever by half degree (°C) cumulative increments during the 4-day follow-up period (i.e., on the day of vaccination and 3 subsequent days) will be tabulated for each group after each dose.
- In addition, the prevalence of each solicited administration site event and solicited systemic event (any grade and grade 3) will be represented graphically over time for each group after each dose. The incidence of each solicited administration site event and solicited systemic event (any grade and grade 3) will be represented graphically for each group after each dose.
- The number and percentage of participants with any unsolicited AEs during the 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) with its exact 95% CI will be tabulated for each dose by group and by Medical Dictionary for Regulatory Activities (MedDRA) preferred term. Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs, for Grade 3 causally related unsolicited AEs and for unsolicited AEs resulting in a medically attended visit. The verbatim reports of unsolicited AEs will be reviewed by a qualified person and the signs and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. Every verbatim term will be matched with the appropriate Preferred Term.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

- The number and percentage of participants with at least one report of SAE classified by the MedDRA Preferred Terms and reported from Dose 1 up to 6 months post-Dose 1 and from revaccination dose up to 6 months post-revaccination will be tabulated with exact 95% CI.
- The number and percentage of participants with at least one report of causally related SAE classified by the MedDRA Preferred Terms and reported during the entire study period will be tabulated with exact 95% CI.
- The same tabulation will be presented for fatal SAEs.
- All SAEs will also be described in detail.
- All AEs/SAEs leading to study/intervention discontinuation from dose 1 up to study end will be tabulated.
- The number and percentage of participants with at least one report of pIMD classified by the MedDRA Preferred Terms and reported from Dose 1 up to 6 months post-Dose 1 and from revaccination dose up to 6 months post-revaccination will be tabulated with exact 95% CI.
- The number and percentage of participants with at least one causally related pIMD classified by the MedDRA Preferred Terms and reported during the entire study period will be tabulated with exact 95% CI.
- All pIMDs will also be described in detail.
- The analyses of unsolicited AEs will include SAEs (unless otherwise specified).

The analysis of safety will also be performed by age category (age at Dose  $1: \ge 65 \text{ YOA}$ ,  $\ge 70 \text{ YOA}$ ,  $\ge 80 \text{ YOA}$ , 60-69 YOA and 70-79 YOA).

#### 5.4.5. Additional considerations

- Compliance in completing solicited events information will be tabulated after each dose and overall.
- The number of days with solicited events reported during the 4-day follow-up period will be tabulated for each solicited event, after each dose using descriptive statistics (mean, min, Q1, median, Q3, maximum).
- The list of solicited administration site and systemic events, and definition of intensity are described in Section 10.3.3 and 10.3.9.1 of the protocol.

The measurement of erythema/swelling (in mm) and fever (in °C/F) will be categorized as follows:

Table 7 Intensity grading scale for solicited events

| Grading | Erythema/swelling | Fever |
|---------|-------------------|---------------------------------------|
| 0: | ≤ 20 mm | < 38.0°C (100.4°F) |
| 1: | > 20 - ≤ 50 mm | ≥ 38.0°C(100.4°F) - ≤ 38.5°C(101.3°F) |
| 2: | > 50 - ≤ 100 mm | > 38.5°C(101.3°F) - ≤ 39.0°C(102.2°F) |
| 3: | > 100 mm | > 39.0°C(102.2°F) |

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

#### **Combined Solicited events and Unsolicited AEs**

For clinicaltrials.gov and EudraCT posting purposes, a summary of combined solicited and unsolicited non-serious adverse events will be produced by System Organ Class and preferred terms and according to occurrence of each event.

Solicited events will be coded by MedDRA as per the following codes:

| Solicited event | Lower level term code | Corresponding Lower |
|-----------------|-----------------------|-------------------------|
| | | level term decode |
| Pain | 10022086 | Injection site pain |
| Erythema | 10015150 | Erythema |
| Swelling | 10053425 | Injection site swelling |
| Fever | 10016558 | Pyrexia |
| Headache | 10019211 | Headache |
| Fatigue | 10016256 | Fatigue |
| Myalgia | 10028411 | Myalgia |
| Arthralgia | 10003239 | Arthralgia |

#### 5.4.5.1. Concomitant Medication

Medications will be coded using the GSKDRUG dictionary.

## 5.4.6. Sensitivity Analyses

If more than 10% of participants miss the revaccination dose or don't have safety data reported after revaccination, the safety analysis described in section 5.4.4 will also be conducted on participants with full follow-up (attending all study visits).

The goal of this sensitivity analysis is to determine the extent to which results might be impacted by considering the different scenarios.

### 6. ANALYSIS INTERPRETATION

All analyses are descriptive.

## 7. INTERIM ANALYSES

## 7.1. Sequence of analyses

Analyses to evaluate objectives and endpoints will be performed stepwise:

• Month 6: A first analysis\* will be performed on all reactogenicity, safety and immunogenicity data available and as clean as possible, when data for at least primary and secondary endpoints up to Month 6 are available for all participants. This analysis will be considered as final for those endpoints.

\*Note: the analysis at Month 6 may be merged with the analysis at the subsequent timepoint.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

- Month 13: A second analysis will be performed on all reactogenicity, safety and immunogenicity data available and as clean as possible, when data for at least primary and secondary endpoints up to Month 12 are available for all participants, as well as data up to 1 month after the first revaccination (Month 13) in the RSV annual group. This analysis will be considered as final for those endpoints.
- Month 18: A third analysis will be performed on all safety and/or immunogenicity data available and as clean as possible, when data for secondary endpoints up to Month 18 are available for all participants. This analysis will be considered as final for those endpoints. Safety and immunogenicity analysis may be performed at different time depending on data availability.
- Month 25: A fourth analysis will be performed on all reactogenicity, safety and immunogenicity data available and as clean as possible, when data for at least primary and secondary endpoints up to Month 24 are available for all participants, as well as data up to 1 month after the second revaccination (Month 25) in the RSV annual group. This analysis will be considered as final for those endpoints.
- The final **End of Study** analysis will be performed when all reactogenicity, safety and immunogenicity data for at least primary and secondary endpoints up to study conclusion are available for all participants (Month 36).
- If the data for tertiary endpoints become available at a later stage, (an) additional analysis/analyses will be performed.

| Description | Analysis<br>ID | Disclosure Purpose<br>(CTRS=public posting, SR=study report,<br>internal) | Reference for TFL<br>TOC |
|---|---|---|---|
| End of study analysis | E1_01 | CTRS, SR | See column 5 in TFL TOC |
| Analysis up to Month 6 | E1_02 | CTRS, SR | See column 5 in TFL TOC |
| Analysis up to Month 13 | E1_03 | CTRS, SR | See column 5 in TFL TOC |
| Analysis up to Month 18 | E1_04 | Internal | See column 5 in TFL TOC |
| Analysis up to Month 25 | E1_05 | Internal | See column 5 in TFL TOC |

# 7.2. Statistical considerations for interim analyses

All analyses will be conducted on final data (as clean as possible) and therefore no statistical adjustment for interim analyses is required.

# 8. CHANGES TO THE PROTOCOL DEFINED STATISTICAL ANALYSIS

Not Applicable

# 9. NON-STANDARD DATA DERIVATION RULES AND STATISTICAL METHODS

The following sections describe additional derivation rules and statistical methods which are not presented in section 10.1 (Business rules for standard data derivations and statistical methods).

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

## 9.1. Handling of missing data

#### 9.1.1. Dates

When partially completed dates (i.e. with missing day or month) are used in calculations, the following rules will be applied:

- Adverse event start dates with missing day:
  - If the month is not the same as the vaccine dose, then the imputed start date will be the 1<sup>st</sup> of the month
  - If the event starts in the same month as the vaccine dose, the flag indicating if the event occurred before or after vaccination (AE.AESTRTPT) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the vaccine dose given during that month. If 'before vaccination' is selected, the imputed date will be one day before the vaccine dose given during that month.
- Adverse event start dates with missing day and month:
  - If the year is not the same as the vaccine dose, then the imputed start date will be the 1<sup>st</sup> of January.
  - If the event starts in the same year as the vaccine dose, the flag indicating if the event occurred before or after vaccination (AE.AESTRTPT) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first vaccine dose given during that year. If 'before vaccination' is selected, the imputed date will be one day before the first vaccine dose given during that year.
- Adverse event end dates with missing day: the imputed end date will be the last day of the month (30 or 31) or the study conclusion date whichever comes first.
- Adverse event end dates with missing day and month: the imputed end date will be the last day of the year (31st of December) or the study conclusion date whichever comes first.

All incomplete concomitant medication/vaccination start/end date will follow the rules above.

#### 10. ANNEXES

# 10.1. Business rules for standard data derivations and statistical methods

This section contains standard rules for data display and derivation for clinical and epidemiological studies.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

## 10.1.1. Attributing events to vaccine doses

The dose relative to an event is the most recent study dose given to a participant prior to the start of a given event. For example, if the start date of an adverse event is between Dose 1 and Dose 2, the relative dose will be Dose 1.

If an event starts on the same day as a study dose, the relative dose will be derived from the additional information provided in the case report form (CRF) using the contents of the flag indicating if the event occurred before or after study dose. If 'after vaccination is selected, the relative dose for the event will be the one administered on the start day of the event. If 'before vaccination is selected, the relative dose for the event will be the dose prior to this one.

## 10.1.2. Handling of missing data

#### 10.1.2.1. Dates

When partially completed dates (i.e. dates missing a day and/or month) are used in calculations, the following standard rules will be applied:

- A missing day will be replaced by 15
- A missing day and month will be replaced by June 30<sup>th</sup>.

See also exceptions in section 9.1.

#### 10.1.2.2. Laboratory data

Missing laboratory results (including immunological data) will not be replaced.

#### 10.1.2.3. Daily recording of solicited events

#### 10.1.2.3.1. Studies with paper diaries

For studies using paper diaries which have questions in the CRF indicating the presence or absence of solicited events, the following rules are applicable:

- Denominators for the summary of administration site (or systemic) solicited events will be calculated using the number of participants who respond "Yes" or "No" to the question concerning the occurrence of administration site (or systemic) events.
- When a specific solicited event is marked as having not occurred following a specific study dose (i.e. SDTM CE.CEOCCUR=N for the specified post-dose period for the event in question), all daily measurements will be imputed as Grade 0.
- When a specific solicited event is marked as having occurred following a specific study dose (i.e. SDTM CE.CEOCCUR=Y for the specified post-dose period for the event in question), any missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the solicited event summary tables.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

• When the occurrence of a specific solicited event is not present (i.e. SDTM CE.CEOCCUR is neither Y nor N for the specified post-dose period for the event in question) but the group of solicited events (administration site or systemic) is marked as having occurred (i.e. SDTM CE.CEOCCUR=Y), all missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the solicited event summary tables.

The following table shows how participants contribute to each category for a specific solicited event over the Day X to Day Y post-dose period:

| Solicited event category | Participants included in the calculation of the numerator |
|---|---|
| Any | All participants with at least one occurrence of the adverse event at grade 1, grade 2, or grade 3 between Day X and Day Y or with the adverse event marked as present and at least one missing daily recording between Day X and Day Y |
| At least grade 1 | All participants with at least one occurrence of the adverse event at grade 1, grade 2, or grade 3 between Day X and Day Y |
| At least grade 2 | All participants with at least one occurrence of the adverse event at grade 2 or grade 3 between Day X and Day Y |
| At least grade 3 | All participants with at least one occurrence of the adverse event at grade 3 between Day X and Day Y |

#### 10.1.2.4. Unsolicited adverse events

Unsolicited adverse event summaries are including serious adverse events unless specified otherwise.

Missing severity, relationship with study vaccine, and outcome of unsolicited adverse events will not be replaced and will appear as 'UNKNOWN' when displayed in a statistical output.

## 10.1.3. Data derivation

#### 10.1.3.1. Age at first dose in years

When age at first dose is to be displayed in years, it will be calculated as the number of complete calendar years between the date of birth and the date of first dose. For example:

DOB = 
$$10$$
SEP1983, Date of first dose =  $0$ 9SEP2018 -> Age = 34 years

DOB = 
$$10$$
SEP1983, Date of first dose =  $10$ SEP2018 -> Age = 35 years

In this study, we will collect only the year of birth. The rules for handling missing day and/or month in the DOB are given in section 10.1.2.1.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

#### 10.1.3.2. Temperature

Temperatures will be presented in degrees Celsius (°C). Temperatures reported in degrees Fahrenheit (°F) will be converted as follows:

Temperature (Celsius) =  $((Temperature (Fahrenheit) - 32) \times 5)/9$ 

#### 10.1.3.3. Numerical serology results

Numerical serology results will be derived from the content of IS.ISORRES in the SDTM dataset. For assays with a specific cut-off, the following derivation rules apply:

| IS.ISORRES | Derived value |
|-----------------------------------------------------|---------------|
| "NEG", "-", or "(-)" | cut-off/2 |
| "POS", "+", or "(+)" | cut-off |
| "< value" and value is <= assay cut-off | cut-off/2 |
| "< value" and value is > assay cut-off | Value |
| "> value" and value is < assay cut-off | cut-off/2 |
| "> value" and value is >= assay cut-off | Value |
| "value" and value is < cut-off | cut-off/2 |
| "value" and value is >= cut-off and value is <=ULOQ | value |
| "value" and value is > ULOQ | ULOQ* |
| All other cases | Missing |

<sup>\*</sup>This rule will be used to compute descriptive statistics (GMTs, fold increase,etc). All values might be displayed in scatter plots with individual results.

#### 10.1.3.4. Geometric mean titres (GMTs) and concentrations (GMCs)

GMT or GMC calculations are performed by taking the inverse logarithm of the mean of the log titre or concentration transformations. Non quantifiable antibody titres or concentrations will be converted as described in section 10.1.3.3 for the purpose of GMT/GMC calculation. Cut-off values are defined by the laboratory before the analysis.

## 10.1.3.5. Onset day

The onset day for an event (e.g. AE, concomitant medication/vaccination) is the number of days between the last study dose and the start date of the event. This is 1 for an event occurring on the same day as a study dose (and reported as starting after study dose).

#### 10.1.3.6. Duration of events

The duration of an event with a start and end date will be the difference between the start and end date plus one day, i.e. an event that starts on 3 March 2018 and ends on 12 March 2018 has a duration of 10 days.

The duration of solicited events will be calculated as the sum of the individual days with the adverse event reported at grade 1 or higher during the solicited event period.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

## 10.1.3.7. Counting rules for combining solicited and unsolicited adverse events

For output combining solicited and unsolicited adverse events, all serious adverse events will be considered systemic events since the administration site flag is not included in the expedited adverse event CRF pages. Unsolicited adverse events with missing administration site flag will also be considered systemic.

Multiple events with the same preferred term which start on the same day are counted as only one occurrence.

#### 10.1.3.8. Counting rules for occurrences of solicited events

When the occurrences of solicited events are summarized, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurs. Also, in the case of co-administered study interventions, an administration site event recorded for a participant following multiple study interventions will be counted as only one occurrence.

## 10.1.4. Display of decimals

### 10.1.4.1. Percentages

Percentages and their corresponding confidence limits will be displayed with one decimal except for 100% in which case no decimal will be displayed.

#### 10.1.4.2. Demographic/baseline characteristics statistics

The mean, median, and standard deviation for continuous baseline characteristics will be presented with one decimal.

The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values.

The maximum and minimum of transformed body temperatures will be displayed with one decimal.

#### 10.1.4.3. Serological summary statistics

For each assay, geometric mean titers (GMT) or concentrations (GMC) and their confidence limits will be presented with one decimal, as well as GMT/GMC fold increase from pre-dose.

The mean, median, standard deviation and quartile values for frequency of RSVPreF3 specific-CD4+ and CD8+ T cells and for the fold increase (post over pre-vaccination) will be presented with one decimal. The minimum and maximum values will be presented with no decimal.

212496 (RSV OA=ADJ-004) Statistical Analysis Plan

## 10.1.5. Statistical methodology

## 10.1.5.1. Exact confidence intervals around proportions

The exact confidence intervals around within-group proportions are derived using the method of Clopper and Pearson [Clopper, 1934].

# 11. ADDITIONAL ANALYSES DUE TO THE COVID-19 PANDEMIC

Depending on how the Covid-19 situation evolves, the SAP might be amended to reflect the analysis corresponding to Covid-19.

#### 12. REFERENCES

Clopper CJ, Pearson E. The Use of Confidence or Fiducial Limits Illustrated in the case of the Binomial. *Biometrika*. 1934;26:404-13.

David MP, Van Herck K, Hardt K, Tibaldi F, Dubin G, Descamps D et al. Long-term persistence of anti-HPV-16 and -18 antibodies induced by vaccination with the AS04-adjuvanted cervical cancer vaccine: modeling of sustained antibody responses. Gynecol Oncol 2009; 115 (Suppl 3):S1-6.